CLINICAL TRIAL: NCT01641809
Title: A Phase IIb, Dose Ranging Study of Oral GSK1265744 in Combination With Nucleoside Reverse Transcriptase Inhibitors for Induction of Human Immunodeficiency Virus -1 (HIV-1) Virologic Suppression Followed by an Evaluation of Maintenance of Virologic Suppression When Oral GSK1265744 is Combined With Oral Rilpivirine in HIV-1 Infected, Antiretroviral Therapy Naive Adult Subjects
Brief Title: Dose Ranging Study of GSK1265744 Plus Nucleoside Reverse Transcriptase Inhibitors for Induction of Human Immunodeficiency Virus-1 (HIV-1) Virologic Suppression Followed by Virologic Suppression Maintenance by GSK1265744 Plus Rilpivirine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116482
Record Dates: First submitted 2012-06-28; First posted 2012-07-17 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: HIV -1; GSK1265744; maintenance phase; dose selection
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — cabotegravir; efavirenz; Rilpivirine; abacavir; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 GSK1265744 10 mg (Experimental): In the Induction Phase subjects will receive oral tablets of GSK1265744 10 mg + matching placebo + investigator-selected background NRTIs (either abacavir/lamivudine or tenofovir/emtricitabine) once daily from Day 1 to Week 24. Subjects continuing in the Maintenance Phase will receive oral tablets of GSK1265744 10 mg + matching placebo + Rilpivirine 25 mg once daily from Week 24 to Week 96.
  Interventions: Drug: GSK1265744 10 mg; Drug: Rilpivirine 25 mg; Drug: Placebo; Drug: Abacavir/Lamivudine (ABC/3TC) or Tenofovir/Emtricitabine (TDF/FTC)
- Arm 2 GSK1265744 30 mg (Experimental): In the Induction Phase subjects will receive oral tablets of GSK1265744 30 mg + matching placebo + investigator-selected background NRTIs (either abacavir/lamivudine or tenofovir/emtricitabine) once daily from Day 1 to Week 24. Subjects continuing in the Maintenance Phase will receive oral tablets of GSK1265744 30 mg + matching placebo + Rilpivirine 25 mg once daily from Week 24 to Week 96.
  Interventions: Drug: GSK1265744 30 mg; Drug: Rilpivirine 25 mg; Drug: Placebo; Drug: Abacavir/Lamivudine (ABC/3TC) or Tenofovir/Emtricitabine (TDF/FTC)
- Arm 3 GSK1265744 60 mg (Experimental): In the Induction Phase subjects will receive oral tablets of GSK1265744 60 mg + investigator-selected background NRTIs (either abacavir/lamivudine or tenofovir/emtricitabine) once daily from Day 1 to Week 24. Subjects continuing in the Maintenance Phase will receive oral tablets of GSK1265744 60 mg + Rilpivirine 25 mg once daily from Week 24 to Week 96.
  Interventions: Drug: GSK1265744 60 mg; Drug: Rilpivirine 25 mg; Drug: Abacavir/Lamivudine (ABC/3TC) or Tenofovir/Emtricitabine (TDF/FTC)
- Arm 4 Efavirenz 600 mg (Active Comparator): In the Induction Phase and Maintenance Phase subjects will receive oral tablets of Efavirenz 600 mg + investigator-selected background NRTIs (either abacavir/lamivudine or tenofovir/emtricitabine).
  Interventions: Drug: Efavirenz 600 mg; Drug: Abacavir/Lamivudine (ABC/3TC) or Tenofovir/Emtricitabine (TDF/FTC)

INTERVENTIONS:
Drug: GSK1265744 10 mg — GSK1265744 10 mg will be administered orally once daily in combination with investigator-selected background NRTIs in the Induction Phase of the study and in combination with Rilpivirine 25 mg in the Maintenance Phase of the study.
  Arms: Arm 1 GSK1265744 10 mg
Drug: GSK1265744 30 mg — GSK1265744 30 mg will be administered orally once daily in combination with investigator-selected background NRTIs in the Induction Phase of the study and in combination with Rilpivirine 25 mg in the Maintenance Phase of the study.
  Arms: Arm 2 GSK1265744 30 mg
Drug: GSK1265744 60 mg — GSK1265744 60 mg will be administered orally once daily in combination with investigator-selected background NRTIs in the Induction Phase of the study and in combination with Rilpivirine 25 mg in the Maintenance Phase of the study.
  Arms: Arm 3 GSK1265744 60 mg
Drug: Efavirenz 600 mg — Efavirenz 600 mg will be administered orally once daily in combination with investigator-selected background NRTIs in the Induction Phase and Maintenance Phase of the study.
  Arms: Arm 4 Efavirenz 600 mg
Drug: Rilpivirine 25 mg — Rilpivirine 25 mg will be administered orally once daily in combination with GSK1265744 10 mg, 30 mg and 60 mg in the Maintenance Phase of the study.
  Arms: Arm 1 GSK1265744 10 mg; Arm 2 GSK1265744 30 mg; Arm 3 GSK1265744 60 mg
Drug: Placebo — Placebo matching to GSK1265744 will be administered along with GSK1265744 10 mg and 30 mg in the Induction phase and Maintenance phase of the study.
  Arms: Arm 1 GSK1265744 10 mg; Arm 2 GSK1265744 30 mg
Drug: Abacavir/Lamivudine (ABC/3TC) or Tenofovir/Emtricitabine (TDF/FTC) — The background dual NRTI therapy for all arms in the Induction Phase and Efavirenz 600 mg arm in the Maintenance Phase will be either abacavir 600 mg + lamivudine 300 mg (ABC/3TC) or tenofovir 300 mg + emtricitabine 200 mg (TDF/FTC) as selected by the Investigator.

SUMMARY:
The study is designed to select a dose of GSK1265744 primarily on the basis of antiviral activity and tolerability in HIV-1 infected, antiretroviral naive subjects.

This study consists of two parts:

Induction Phase: Approximately 200 subjects will be randomized (50 subjects in each of the 4 treatment arms). The Induction Phase consists of a 24 week dose-ranging evaluation of GSK1265744 at blinded doses of 10 mg, 30 mg and 60 mg once-daily and a control arm of open-label efavirenz (EFV) 600 mg once daily. The background dual nucleoside reverse transcriptase inhibitor (NRTI) antiretroviral therapy (ART) for all arms will be either abacavir/lamivudine (ABC/3TC) or tenofovir/emtricitabine (TDF/FTC) as selected by the Investigator. Subjects randomized to a GSK1265744 containing arm, who successfully complete 24 weeks on study and demonstrate virologic suppression (defined as having a plasma HIV-1 ribonucleic acid [RNA] <50 copies per milliliter [c/mL] before Week 24, with no signs of virologic rebound) will become eligible for the Maintenance Phase of this study.

Maintenance Phase: The background NRTIs will be discontinued and the subjects will continue their randomized dose of GSK1265744 in combination with rilpivirine (RPV) 25 mg once-daily for an additional 72 weeks. The Maintenance phase will evaluate the ability of this two drug ART regimen to maintain virologic suppression through Week 48, Week 72 and Week 96. Subjects randomized to the EFV arm will continue on their randomized regimen through Week 96.

After completion of the maintenance phase, subjects could enroll in the Open-Label Phase to continue GSK1265744 + RPV treatment as long as they continue to derive clinical benefit and until it is locally approved and commercially available.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected male or female subjects >= 18 years of age
* Screening plasma HIV-1 RNA >=1000 c/mL
* CD4+ cell count >=200 cells/millimeter (mm)^3
* ART-naive defined as having =<10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection
* Female subjects of child bearing potential are eligible to enter if they are not pregnant and willing to use protocol-specified methods of contraception to prevent pregnancy during the study

Exclusion Criteria:

* Any evidence at screening of an active Centers for Disease and Prevention Control (CDC) Category C disease
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* History of ongoing or clinically relevant hepatitis within the previous 6 months, and subjects with moderate to severe hepatic impairment will be excluded
* Women who are breastfeeding
* Subject, who in the investigator's judgment, poses a significant suicide risk
* Any clinically significant finding on screening or baseline electrocardiograph (ECG)
* The presence of any specific laboratory abnormalities at Screening
* History of cardiac disease
* Clinically relevant pancreatitis
* Subjects who are unlikely to complete the dosing schedule due to a pre-existing physical or mental condition
* Any condition which impairs the absorption, distribution, metabolism or excretion of the investigational product
* Any evidence of primary resistance based upon the presence of a major resistance associated mutation in the Screening HIV genotype, or any historical genotype
* Treatment with any protocol-specified excluded medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2013-10-10 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (41):
- United States (38):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Annandale, Virginia
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec

REFERENCES:
- [Derived] Mills A, Richmond GJ, Newman C, Osiyemi O, Cade J, Brinson C, De Vente J, Margolis DA, Sutton KC, Wilches V, Hatch S, Roberts J, McCoig C, Garris C, Vandermeulen K, Spreen WR. Long-acting cabotegravir and rilpivirine for HIV-1 suppression: switch to 2-monthly dosing after 5 years of daily oral therapy. AIDS. 2022 Feb 1;36(2):195-203. doi: 10.1097/QAD.0000000000003085. PMID 34652287
- [Derived] Patel P, Xue Z, King KS, Parham L, Ford S, Lou Y, Bakshi KK, Sutton K, Margolis D, Hughes AR, Spreen WR. Evaluation of the effect of UGT1A1 polymorphisms on the pharmacokinetics of oral and long-acting injectable cabotegravir. J Antimicrob Chemother. 2020 Aug 1;75(8):2240-2248. doi: 10.1093/jac/dkaa147. PMID 32361755
- [Derived] Margolis DA, Brinson CC, Smith GHR, de Vente J, Hagins DP, Eron JJ, Griffith SK, Clair MHS, Stevens MC, Williams PE, Ford SL, Stancil BS, Bomar MM, Hudson KJ, Smith KY, Spreen WR; LAI116482 Study Team. Cabotegravir plus rilpivirine, once a day, after induction with cabotegravir plus nucleoside reverse transcriptase inhibitors in antiretroviral-naive adults with HIV-1 infection (LATTE): a randomised, phase 2b, dose-ranging trial. Lancet Infect Dis. 2015 Oct;15(10):1145-1155. doi: 10.1016/S1473-3099(15)00152-8. Epub 2015 Jul 19. PMID 26201299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, two part study in human immunodeficiency virus-1 (HIV-1) infected antiretroviral therapy (ART) naïve adult participants conducted across 48 sites in the United States (US) and Canada.
Pre-assignment Details: A total of 324 participants were screened, of which 80 failed screening and 244 participants were randomized to one of the four treatment arms in a ratio of 1:1:1:1. Of the 244 randomized participants, only 243 received atleast one dose of study treatment and comprised the Intent-to-Treat-Exposed (ITT-E) Population.
Groups:
- GSK1265744 10 mg: Participants were administered one tablet of GSK1265744 10 milligrams (mg) and one tablet of placebo once daily along with investigator selected, fixed dose dual nucleoside reverse transcriptase inhibitor (NRTI) therapy (either abacavir/lamivudine ABC/3TC 600 mg/300 mg or tenofovir/emtricitabine TDF/FTC 300 mg/200 mg from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received one tablet of GSK1265744 10 mg and one tablet of placebo in combination with one tablet of rilpivirine (RPV) 25 mg once daily from Week 24 to Week 96. Participants continuing in the open-label phase of the study received one tablet of GSK1265744 30 mg along with RPV 25 mg once daily. All doses were administered orally with a meal.
- GSK1265744 30 mg: Participants were administered one tablet of GSK1265744 30 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received one tablet of GSK1265744 30 mg and one tablet of placebo in combination with one tablet of RPV 25 mg once daily from Week 24 to Week 96. Participants continuing in the open-label phase of the study received one tablet of GSK1265744 30 mg along with RPV 25 mg once daily. All doses were administered orally with a meal.
- GSK1265744 60 mg: Participants were administered two tablets of GSK1265744 30 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received two tablets of GSK1265744 30 mg in combination with one tablet of RPV 25 mg once daily from Week 24 to Week 96. Participants continuing in the open-label phase of the study received one tablet of GSK1265744 30 mg along with RPV 25 mg once daily. All doses were administered orally with a meal.
- Efavirenz 600 mg: Participants were administered one tablet of efavirenz 600 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants continued to receive one tablet of efavirenz 600 mg in combination with ABC/3TC or TDF/FTC once daily. Participants in this arm did not enter open-label phase and were considered to have completed the study after Week 96.
Period: Induction Phase (Day 1 to Week 24)
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Started | 60 | 60 | 61 | 62
Completed | 52 | 53 | 55 | 47
Not Completed | 8 | 7 | 6 | 15
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0 | 3
Not completed — Protocol Violation | 2 | 1 | 1 | 0
Not completed — Lack of Efficacy | 4 | 1 | 2 | 3
Not completed — Adverse Event | 0 | 1 | 3 | 7
Period: Maintenance Phase (Week 24 to Week 96)
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Started | 52 | 53 | 55 | 47
Completed | 46 | 48 | 52 | 41
Not Completed | 6 | 5 | 3 | 6
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 2
Not completed — Lack of Efficacy | 1 | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 2
Period: Open-label (Week 96 to Week 324)
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Started | 46 | 47 (1 participant completed study as per protocol at Week 96 and opted to not enter open-label phase) | 51 (1 participant completed study as per protocol at Week 96 and opted to not enter open-label phase) | 0 (Participants completed study at Week 96 and did not enter open-label phase)
Completed | 30 | 35 | 43 | 0
Not Completed | 16 | 12 | 8 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 5 | 4 | 5 | 0
Not completed — Site closed | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg | Total
Number analyzed (Participants) | 60 | 60 | 61 | 62 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (9.91) | 34.4 (10.24) | 36.2 (10.15) | 35.6 (12.30) | 35.1 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 1 | 10
  Male | 57 | 58 | 57 | 61 | 233
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American (Af Am)/African Heritage (Her) | 21 | 17 | 18 | 20 | 76
  American Indian or Alaskan Native (Nat) | 0 | 0 | 2 | 2 | 4
  Asian-Central/South Asian Her | 1 | 1 | 1 | 0 | 3
  Asian-Japanese/East Asian/South East Asian Her | 0 | 1 | 2 | 0 | 3
  White | 37 | 39 | 36 | 39 | 151
  Af Am/Af Her and Asian and White | 0 | 0 | 1 | 0 | 1
  Af Am/Af Her & Nat Hawaiian/other Pacific islander | 0 | 0 | 1 | 0 | 1
  Af Am/Af Her & White | 0 | 2 | 0 | 0 | 2
  American Indian or Alaskan Native & White | 1 | 0 | 0 | 0 | 1
  Asian & White | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) <50 Copies/Milliliter (mL) at Week 48 Using the Missing, Switch, Discontinuation Equals Failure (MSDF) Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 was determined using the MSDF algorithm based on the current US Food and Drug Administration (FDA) definition of Snapshot algorithm. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to visit window) as well as participants who switch their concomitant antiretroviral therapy prior to the visit of interest as non-responders. Virological response within an analysis window was determined by the last available HIV-1 RNA measurement in that window while the participant was on-treatment. MSDF response rate was calculated as number of responders in the analysis window divided by the number of participants in the analysis population. ITT-E Population comprised of all randomized participants who received at least one dose of investigational product.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants | 80 [70 to 90] | 80 [70 to 90] | 87 [78 to 95] | 71 [60 to 82]

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <400 Copies/mL Until Week 96 Using the MSDF Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The percentage of participants with HIV-1 RNA <400 copies/mL over time was determined using the MSDF algorithm based on the current US FDA definition of the Snapshot algorithm. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to visit window) as well as participants who switch their concomitant antiretroviral therapy prior to the visit of interest as non-responders. Virological response within an analysis window was determined by the last available HIV-1 RNA measurement in that window while the participant was on-treatment. MSDF response rate was calculated as number of responders in the analysis window divided by the number of participants in the analysis population.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants
  Baseline | 0 | 0 | 0 | 0
  Week 2 | 87 | 80 | 84 | 68
  Week 4 | 93 | 93 | 93 | 68
  Week 8 | 93 | 92 | 92 | 79
  Week 12 | 90 | 85 | 89 | 73
  Week 16 | 93 | 87 | 93 | 81
  Week 24 | 93 | 87 | 92 | 79
  Week 26 | 80 | 80 | 87 | 71
  Week 28 | 85 | 83 | 85 | 73
  Week 32 | 87 | 85 | 89 | 73
  Week 36 | 87 | 85 | 90 | 73
  Week 40 | 87 | 85 | 90 | 73
  Week 48 | 83 | 85 | 89 | 73
  Week 60 | 80 | 77 | 87 | 71
  Week 72 | 77 | 75 | 85 | 68
  Week 84 | 77 | 77 | 85 | 68
  Week 96 | 75 | 77 | 85 | 65

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <400 Copies/mL Until Week 96 Using the Observed Case Analysis
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with HIV-1 RNA <400 copies/mL over time was determined using the observed case analysis, which did not impute for any missing assessments. Observed case response rate was calculated as the number of participants with a positive response at the time point where the participant is on randomized therapy divided by the number of participants in the analysis population with an assessment in the scheduled visit window during the randomized period.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles)
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants
  Baseline; n=60, 60, 61, 62 | 0 | 0 | 0 | 0
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 91 | 86 | 86 | 71
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | 97 | 98 | 97 | 74
  Week 8; n=59, 56, 57, 55: number analyzed (Participants) | 59 | 56 | 57 | 55
  Week 8; n=59, 56, 57, 55 | 95 | 98 | 98 | 91
  Week 12; n=58, 52, 57, 51: number analyzed (Participants) | 58 | 52 | 57 | 51
  Week 12; n=58, 52, 57, 51 | 97 | 100 | 98 | 92
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 98 | 100 | 100 | 96
  Week 20; n=56, 54, 56, 47: number analyzed (Participants) | 56 | 54 | 56 | 47
  Week 20; n=56, 54, 56, 47 | 100 | 100 | 100 | 100
  Week 24; n=56, 53, 56, 48: number analyzed (Participants) | 56 | 53 | 56 | 48
  Week 24; n=56, 53, 56, 48 | 100 | 100 | 100 | 100
  Week 26; n=48, 50, 53, 44: number analyzed (Participants) | 48 | 50 | 53 | 44
  Week 26; n=48, 50, 53, 44 | 100 | 100 | 100 | 100
  Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  Week 28; n=51, 52, 52, 45 | 100 | 100 | 100 | 100
  Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 32; n=52, 53, 55, 45 | 100 | 100 | 98 | 100
  Week 36; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 36; n=52, 53, 55, 45 | 100 | 100 | 100 | 100
  Week 40; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 40; n=52, 53, 55, 45 | 100 | 100 | 100 | 100
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 98 | 98 | 100 | 100
  Week 60; n=48, 48, 53, 44: number analyzed (Participants) | 48 | 48 | 53 | 44
  Week 60; n=48, 48, 53, 44 | 96 | 100 | 100 | 98
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 98 | 96 | 100 | 100
  Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Week 84; n=46, 48, 52, 42 | 100 | 98 | 100 | 100
  Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Week 96; n=45, 48, 52, 40 | 96 | 100 | 100 | 100

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL Over Time by Visit Using the MSDF Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with HIV-1 RNA <50 copies/mL over time was determined using the MSDF algorithm based on the current US FDA definition of the Snapshot algorithm. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to visit window) as well as participants who switch their concomitant antiretroviral therapy prior to the visit of interest as non-responders. Virological response within an analysis window was determined by the last available HIV-1 RNA measurement in that window while the participant was on-treatment. MSDF response rate was calculated as number of responders in the analysis window divided by the number of participants in the analysis population.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300 and 312
Population: ITT-E Population. Participants randomized to Efavirenz 600 mg arm were considered to have completed their participation in the study after Week 96; hence were no longer followed as part of this study.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants
  Baseline | 0 | 0 | 0 | 0
  Week 2 | 48 | 50 | 51 | 13
  Week 4 | 80 | 78 | 70 | 24
  Week 8 | 90 | 83 | 87 | 48
  Week 12 | 88 | 75 | 82 | 61
  Week 16 | 90 | 83 | 87 | 74
  Week 24 | 87 | 85 | 87 | 74
  Week 26 | 78 | 75 | 85 | 66
  Week 28 | 85 | 78 | 85 | 69
  Week 32 | 83 | 80 | 87 | 69
  Week 36 | 85 | 82 | 85 | 71
  Week 40 | 83 | 82 | 85 | 68
  Week 48 | 80 | 80 | 87 | 71
  Week 60 | 78 | 73 | 85 | 68
  Week 72 | 72 | 73 | 85 | 68
  Week 84 | 72 | 75 | 85 | 68
  Week 96 | 68 | 75 | 84 | 63
  Week 108 | 68 | 72 | 80 | 0
  Week 120 | 65 | 73 | 80 | 0
  Week 132 | 62 | 70 | 80 | 0
  Week 144 | 58 | 67 | 77 | 0
  Week 156 | 58 | 63 | 80 | 0
  Week 168 | 57 | 65 | 75 | 0
  Week 180 | 58 | 67 | 75 | 0
  Week 192 | 57 | 65 | 74 | 0
  Week 204 | 55 | 62 | 75 | 0
  Week 216 | 55 | 63 | 77 | 0
  Week 228 | 53 | 63 | 75 | 0
  Week 240 | 50 | 62 | 74 | 0
  Week 252 | 52 | 62 | 75 | 0
  Week 264 | 53 | 62 | 75 | 0
  Week 276 | 52 | 62 | 70 | 0
  Week 288 | 50 | 62 | 74 | 0
  Week 300 | 52 | 60 | 70 | 0
  Week 312 | 52 | 52 | 70 | 0

5. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL Over Time by Visit Using Observed Case Analysis
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with HIV-1 RNA <50 copies/mL over time was determined using the observed case analysis, which did not impute for any missing assessments. Observed case response rate was calculated as the number of participants with a positive response at the time point where the participant is on therapy divided by the number of participants in the analysis population with an assessment in the scheduled visit window during the randomized period or open-label phase.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312 and 324
Population: ITT-E Population. Participants randomized to Efavirenz 600 mg arm were considered to have completed their participation in the study after Week 96; hence were no longer followed as part of this study. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles)
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants
  Baseline; n=60, 60, 61, 62 | 0 | 0 | 0 | 0
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 51 | 54 | 53 | 14
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | 83 | 82 | 73 | 26
  Week 8; n=59, 56, 57, 55: number analyzed (Participants) | 59 | 56 | 57 | 55
  Week 8; n=59, 56, 57, 55 | 92 | 89 | 93 | 55
  Week 12; n=58, 52, 57, 51: number analyzed (Participants) | 58 | 52 | 57 | 51
  Week 12; n=58, 52, 57, 51 | 95 | 88 | 91 | 76
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 95 | 94 | 93 | 87
  Week 20; n=56, 54, 56, 47: number analyzed (Participants) | 56 | 54 | 56 | 47
  Week 20; n=56, 54, 56, 47 | 91 | 98 | 98 | 91
  Week 24; n=56, 53, 56, 48: number analyzed (Participants) | 56 | 53 | 56 | 48
  Week 24; n=56, 53, 56, 48 | 93 | 98 | 95 | 96
  Week 26; n=48, 50, 53, 44: number analyzed (Participants) | 48 | 50 | 53 | 44
  Week 26; n=48, 50, 53, 44 | 98 | 94 | 98 | 93
  Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  Week 28; n=51, 52, 52, 45 | 100 | 94 | 100 | 96
  Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 32; n=52, 53, 55, 45 | 96 | 94 | 96 | 96
  Week 36; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 36; n=52, 53, 55, 45 | 98 | 96 | 95 | 98
  Week 40; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 40; n=52, 53, 55, 45 | 96 | 96 | 95 | 93
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 92 | 92 | 98 | 98
  Week 60; n=48, 48, 53, 44: number analyzed (Participants) | 48 | 48 | 53 | 44
  Week 60; n=48, 48, 53, 44 | 94 | 96 | 98 | 95
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 91 | 92 | 100 | 100
  Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Week 84; n=46, 48, 52, 42 | 91 | 94 | 100 | 100
  Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Week 96; n=45, 48, 52, 40 | 89 | 98 | 98 | 98
  Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  Week 108; n=43, 46, 49, 0 | 95 | 96 | 100 |
  Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  Week 120; n=41, 46, 49, 0 | 95 | 100 | 98 |
  Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  Week 132; n=40, 46, 49, 0 | 95 | 96 | 100 |
  Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  Week 144; n=37, 45, 47, 0 | 92 | 93 | 98 |
  Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  Week 156; n=37, 42, 49, 0 | 95 | 95 | 98 |
  Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  Week 168; n=35, 43, 47, 0 | 94 | 95 | 98 |
  Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  Week 180; n=36, 41, 47, 0 | 97 | 100 | 98 |
  Week 192; n=36, 40, 47, 0: number analyzed (Participants) | 36 | 40 | 47 | 0
  Week 192; n=36, 40, 47, 0 | 94 | 100 | 96 |
  Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  Week 204; n=34, 39, 47, 0 | 97 | 97 | 98 |
  Week 216; n=33, 39, 47, 0: number analyzed (Participants) | 33 | 39 | 47 | 0
  Week 216; n=33, 39, 47, 0 | 100 | 100 | 98 |
  Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Week 228; n=32, 39, 47, 0 | 100 | 100 | 98 |
  Week 240; n=31, 39, 45, 0: number analyzed (Participants) | 31 | 39 | 45 | 0
  Week 240; n=31, 39, 45, 0 | 97 | 97 | 100 |
  Week 252; n=31, 38, 47, 0: number analyzed (Participants) | 31 | 38 | 47 | 0
  Week 252; n=31, 38, 47, 0 | 100 | 97 | 98 |
  Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  Week 264; n=32, 38, 47, 0 | 100 | 100 | 98 |
  Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  Week 276; n=31, 38, 45, 0 | 100 | 100 | 96 |
  Week 288; n=30, 38, 45, 0: number analyzed (Participants) | 30 | 38 | 45 | 0
  Week 288; n=30, 38, 45, 0 | 100 | 100 | 100 |
  Week 300; n=31, 37, 44, 0: number analyzed (Participants) | 31 | 37 | 44 | 0
  Week 300; n=31, 37, 44, 0 | 97 | 100 | 95 |
  Week 312; n=31, 33, 43, 0: number analyzed (Participants) | 31 | 33 | 43 | 0
  Week 312; n=31, 33, 43, 0 | 100 | 97 | 100 |
  Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  Week 324; n=3, 4, 3, 0 | 100 | 100 | 100 |

6. Secondary Outcome: Absolute Values for Plasma Logarithm to the Base 10 (log10) HIV-1 RNA Over Time by Visit
Description: Plasma samples for quantitative analysis of HIV-1 RNA were collected at indicated time points. Baseline value is the last pre-treatment value observed.
Time Frame: as for outcome 5
Population: ITT-E Population. Participants randomized to Efavirenz 600 mg arm were considered to have completed their participation in the study after Week 96; hence were no longer followed as part of this study. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Log10 copies per milliliter
  Baseline; n=60, 60, 61, 62 | 4.424 (0.5834) | 4.270 (0.6359) | 4.428 (0.6418) | 4.290 (0.6683)
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 1.883 (0.4551) | 1.984 (0.5786) | 1.939 (0.5071) | 2.415 (0.5717)
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | 1.706 (0.3245) | 1.731 (0.4141) | 1.725 (0.2750) | 2.201 (0.5780)
  Week 8; n=59, 56, 57, 55: number analyzed (Participants) | 59 | 56 | 57 | 55
  Week 8; n=59, 56, 57, 55 | 1.695 (0.4114) | 1.666 (0.3676) | 1.666 (0.3926) | 1.950 (0.5636)
  Week 12; n=58, 52, 57, 51: number analyzed (Participants) | 58 | 52 | 57 | 51
  Week 12; n=58, 52, 57, 51 | 1.643 (0.2506) | 1.618 (0.0786) | 1.641 (0.2033) | 1.758 (0.4082)
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 1.619 (0.1418) | 1.602 (0.0354) | 1.616 (0.0956) | 1.697 (0.3277)
  Week 20; n=56, 54, 56, 47: number analyzed (Participants) | 56 | 54 | 56 | 47
  Week 20; n=56, 54, 56, 47 | 1.623 (0.1175) | 1.596 (0.0346) | 1.599 (0.0591) | 1.649 (0.1962)
  Week 24; n=56, 53, 56, 48: number analyzed (Participants) | 56 | 53 | 56 | 48
  Week 24; n=56, 53, 56, 48 | 1.615 (0.1010) | 1.597 (0.0360) | 1.603 (0.0532) | 1.610 (0.0902)
  Week 26; n=48, 50, 53, 44: number analyzed (Participants) | 48 | 50 | 53 | 44
  Week 26; n=48, 50, 53, 44 | 1.595 (0.0270) | 1.602 (0.0434) | 1.594 (0.0194) | 1.610 (0.0742)
  Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  Week 28; n=51, 52, 52, 45 | 1.591 (0.0000) | 1.607 (0.0565) | 1.591 (0.0000) | 1.600 (0.0451)
  Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 32; n=52, 53, 55, 45 | 1.609 (0.0955) | 1.620 (0.1277) | 1.618 (0.1742) | 1.614 (0.1022)
  Week 36; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 36; n=52, 53, 55, 45 | 1.604 (0.0782) | 1.610 (0.1070) | 1.606 (0.0722) | 1.607 (0.1068)
  Week 40; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 40; n=52, 53, 55, 45 | 1.612 (0.1206) | 1.618 (0.1214) | 1.608 (0.0752) | 1.607 (0.0650)
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 1.686 (0.4077) | 1.654 (0.3673) | 1.598 (0.0508) | 1.596 (0.0247)
  Week 60; n=48, 48, 53, 44: number analyzed (Participants) | 48 | 48 | 53 | 44
  Week 60; n=48, 48, 53, 44 | 1.648 (0.2643) | 1.598 (0.0300) | 1.594 (0.0205) | 1.657 (0.3948)
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 1.625 (0.1584) | 1.697 (0.4705) | 1.591 (0.0000) | 1.592 (0.0065)
  Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Week 84; n=46, 48, 52, 42 | 1.645 (0.1838) | 1.643 (0.2896) | 1.592 (0.0059) | 1.591 (0.0017)
  Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Week 96; n=45, 48, 52, 40 | 1.681 (0.2783) | 1.603 (0.0861) | 1.596 (0.0227) | 1.598 (0.0467)
  Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  Week 108; n=43, 46, 49, 0 | 1.634 (0.1979) | 1.609 (0.0885) | 1.591 (0.0000) |
  Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  Week 120; n=41, 46, 49, 0 | 1.638 (0.2216) | 1.591 (0.0000) | 1.618 (0.1884) |
  Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  Week 132; n=40, 46, 49, 0 | 1.646 (0.2491) | 1.631 (0.2097) | 1.591 (0.0000) |
  Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  Week 144; n=37, 45, 47, 0 | 1.682 (0.4027) | 1.698 (0.5940) | 1.630 (0.2656) |
  Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  Week 156; n=37, 42, 49, 0 | 1.634 (0.1850) | 1.603 (0.0520) | 1.619 (0.1833) |
  Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  Week 168; n=35, 43, 47, 0 | 1.665 (0.3351) | 1.642 (0.2908) | 1.603 (0.0810) |
  Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  Week 180; n=36, 41, 47, 0 | 1.613 (0.1324) | 1.591 (0.0000) | 1.600 (0.0584) |
  Week 192; n=36, 40, 47, 0: number analyzed (Participants) | 36 | 40 | 47 | 0
  Week 192; n=36, 40, 47, 0 | 1.689 (0.4119) | 1.591 (0.0000) | 1.699 (0.6971) |
  Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  Week 204; n=34, 39, 47, 0 | 1.628 (0.2162) | 1.595 (0.0252) | 1.634 (0.2936) |
  Week 216; n=33, 39, 47, 0: number analyzed (Participants) | 33 | 39 | 47 | 0
  Week 216; n=33, 39, 47, 0 | 1.591 (0.0000) | 1.592 (0.0052) | 1.634 (0.2948) |
  Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Week 228; n=32, 39, 47, 0 | 1.591 (0.0000) | 1.591 (0.0000) | 1.625 (0.2351) |
  Week 240; n=31, 39, 45, 0: number analyzed (Participants) | 31 | 39 | 45 | 0
  Week 240; n=31, 39, 45, 0 | 1.596 (0.0268) | 1.601 (0.0465) | 1.591 (0.0000) |
  Week 252; n=31, 38, 47, 0: number analyzed (Participants) | 31 | 38 | 47 | 0
  Week 252; n=31, 38, 47, 0 | 1.591 (0.0000) | 1.599 (0.0461) | 1.593 (0.0157) |
  Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  Week 264; n=32, 38, 47, 0 | 1.591 (0.0000) | 1.591 (0.0000) | 1.617 (0.1788) |
  Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  Week 276; n=31, 38, 45, 0 | 1.591 (0.0000) | 1.591 (0.0000) | 1.618 (0.1398) |
  Week 288; n=30, 38, 45, 0: number analyzed (Participants) | 30 | 38 | 45 | 0
  Week 288; n=30, 38, 45, 0 | 1.591 (0.000) | 1.592 (0.0052) | 1.591 (0.0000) |
  Week 300; n=31, 37, 44, 0: number analyzed (Participants) | 31 | 37 | 44 | 0
  Week 300; n=31, 37, 44, 0 | 1.601 (0.0551) | 1.591 (0.0000) | 1.625 (0.1753) |
  Week 312; n=31, 33, 43, 0: number analyzed (Participants) | 31 | 33 | 43 | 0
  Week 312; n=31, 33, 43, 0 | 1.597 (0.0214) | 1.600 (0.0494) | 1.591 (0.0000) |
  Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  Week 324; n=3, 4, 3, 0 | 1.591 (0.0000) | 1.591 (0.0000) | 1.591 (0.0000) |

7. Secondary Outcome: Change From Baseline in Plasma log10 HIV-1 RNA Over Time by Visit
Description: Plasma samples for quantitative analysis of HIV-1 RNA were collected at indicated time points. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312 and 324
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Log10 copies per milliliter
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | -2.534 (0.4175) | -2.306 (0.5937) | -2.504 (0.4311) | -1.875 (0.4273)
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | -2.731 (0.4158) | -2.550 (0.6300) | -2.718 (0.4981) | -2.092 (0.4866)
  Week 8; n=59, 56, 57, 55: number analyzed (Participants) | 59 | 56 | 57 | 55
  Week 8; n=59, 56, 57, 55 | -2.733 (0.6374) | -2.611 (0.6938) | -2.741 (0.7034) | -2.344 (0.6765)
  Week 12; n=58, 52, 57, 51: number analyzed (Participants) | 58 | 52 | 57 | 51
  Week 12; n=58, 52, 57, 51 | -2.793 (0.5574) | -2.634 (0.6308) | -2.790 (0.6515) | -2.533 (0.6580)
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | -2.823 (0.5118) | -2.659 (0.6363) | -2.815 (0.6170) | -2.602 (0.6698)
  Week 20; n=56, 54, 56, 47: number analyzed (Participants) | 56 | 54 | 56 | 47
  Week 20; n=56, 54, 56, 47 | -2.823 (0.5329) | -2.665 (0.6418) | -2.834 (0.6250) | -2.666 (0.6512)
  Week 24; n=56, 53, 56, 48: number analyzed (Participants) | 56 | 53 | 56 | 48
  Week 24; n=56, 53, 56, 48 | -2.831 (0.5465) | -2.659 (0.6488) | -2.830 (0.6304) | -2.694 (0.6843)
  Week 26; n=48, 50, 53, 44: number analyzed (Participants) | 48 | 50 | 53 | 44
  Week 26; n=48, 50, 53, 44 | -2.788 (0.5023) | -2.662 (0.6670) | -2.792 (0.6014) | -2.733 (0.6879)
  Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  Week 28; n=51, 52, 52, 45 | -2.784 (0.4944) | -2.663 (0.6356) | -2.791 (0.5831) | -2.714 (0.6873)
  Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 32; n=52, 53, 55, 45 | -2.763 (0.5164) | -2.636 (0.6598) | -2.781 (0.6146) | -2.672 (0.6812)
  Week 36; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 36; n=52, 53, 55, 45 | -2.768 (0.5000) | -2.646 (0.6786) | -2.792 (0.5803) | -2.679 (0.6776)
  Week 40; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 40; n=52, 53, 55, 45 | -2.760 (0.5143) | -2.638 (0.6581) | -2.790 (0.5736) | -2.679 (0.6817)
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | -2.682 (0.6637) | -2.602 (0.7855) | -2.799 (0.5946) | -2.676 (0.6773)
  Week 60; n=48, 48, 53, 44: number analyzed (Participants) | 48 | 48 | 53 | 44
  Week 60; n=48, 48, 53, 44 | -2.729 (0.6405) | -2.613 (0.6068) | -2.787 (0.5920) | -2.615 (0.8875)
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | -2.745 (0.5229) | -2.514 (0.7487) | -2.783 (0.6009) | -2.738 (0.6415)
  Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Week 84; n=46, 48, 52, 42 | -2.722 (0.5650) | -2.568 (0.7144) | -2.782 (0.5994) | -2.739 (0.6431)
  Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Week 96; n=45, 48, 52, 40 | -2.670 (0.5277) | -2.608 (0.6342) | -2.778 (0.5943) | -2.731 (0.6586)
  Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  Week 108; n=43, 46, 49, 0 | -2.723 (0.5396) | -2.632 (0.6265) | -2.743 (0.5851) |
  Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  Week 120; n=41, 46, 49, 0 | -2.712 (0.5477) | -2.650 (0.6137) | -2.717 (0.6180) |
  Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  Week 132; n=40, 46, 49, 0 | -2.705 (0.5504) | -2.610 (0.6718) | -2.743 (0.5851) |
  Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  Week 144; n=37, 45, 47, 0 | -2.690 (0.6615) | -2.555 (0.9008) | -2.703 (0.6903) |
  Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  Week 156; n=37, 42, 49, 0 | -2.737 (0.5476) | -2.645 (0.6129) | -2.716 (0.6309) |
  Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  Week 168; n=35, 43, 47, 0 | -2.680 (0.6170) | -2.592 (0.7138) | -2.700 (0.5907) |
  Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  Week 180; n=36, 41, 47, 0 | -2.747 (0.4984) | -2.628 (0.6251) | -2.767 (0.5672) |
  Week 192; n=36, 40, 47, 0: number analyzed (Participants) | 36 | 40 | 47 | 0
  Week 192; n=36, 40, 47, 0 | -2.671 (0.6656) | -2.641 (0.6272) | -2.667 (0.8708) |
  Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  Week 204; n=34, 39, 47, 0 | -2.750 (0.5359) | -2.632 (0.6353) | -2.718 (0.7294) |
  Week 216; n=33, 39, 47, 0: number analyzed (Participants) | 33 | 39 | 47 | 0
  Week 216; n=33, 39, 47, 0 | -2.787 (0.4956) | -2.636 (0.6337) | -2.718 (0.6660) |
  Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Week 228; n=32, 39, 47, 0 | -2.770 (0.4940) | -2.636 (0.6346) | -2.726 (0.6757) |
  Week 240; n=31, 39, 45, 0: number analyzed (Participants) | 31 | 39 | 45 | 0
  Week 240; n=31, 39, 45, 0 | -2.798 (0.4923) | -2.627 (0.6181) | -2.736 (0.5861) |
  Week 252; n=31, 38, 47, 0: number analyzed (Participants) | 31 | 38 | 47 | 0
  Week 252; n=31, 38, 47, 0 | -2.787 (0.5092) | -2.601 (0.6209) | -2.758 (0.5875) |
  Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  Week 264; n=32, 38, 47, 0 | -2.780 (0.5022) | -2.659 (0.6264) | -2.734 (0.6213) |
  Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  Week 276; n=31, 38, 45, 0 | -2.786 (0.5095) | -2.659 (0.6264) | -2.764 (0.6002) |
  Week 288; n=30, 38, 45, 0: number analyzed (Participants) | 30 | 38 | 45 | 0
  Week 288; n=30, 38, 45, 0 | -2.768 (0.5083) | -2.659 (0.6246) | -2.775 (0.5984) |
  Week 300; n=31, 37, 44, 0: number analyzed (Participants) | 31 | 37 | 44 | 0
  Week 300; n=31, 37, 44, 0 | -2.776 (0.5062) | -2.664 (0.6344) | -2.730 (0.6786) |
  Week 312; n=31, 33, 43, 0: number analyzed (Participants) | 31 | 33 | 43 | 0
  Week 312; n=31, 33, 43, 0 | -2.780 (0.5085) | -2.569 (0.6037) | -2.789 (0.5825) |
  Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  Week 324; n=3, 4, 3, 0 | -2.488 (0.1409) | -2.215 (0.4624) | -2.438 (0.5904) |

8. Secondary Outcome: Number of Participants With Post-Baseline HIV-1 Associated Conditions Progression of Disease
Description: HIV-1 associated conditions were assessed according to the 1993 Centers for Disease Control and Prevention (CDC) Revised Classification System for HIV Infection in Adults. The clinical categories of HIV infection as per CDC system are class A=Asymptomatic HIV infection or lymphadenopathy or acute HIV infection; class B=symptomatic non-acquired immunodeficiency syndrome (AIDS) conditions and class C=AIDS indicator conditions. Number of participants experiencing disease progression is presented, where disease progression is defined as the progression from Baseline HIV disease status as follows: CDC class A at Baseline to CDC class C event; CDC Class B at Baseline to CDC Class C event; CDC Class C at Baseline to new CDC Class C event; and CDC class A, B or C at Baseline to death.
Time Frame: Up to Week 324
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  CDC Class A to CDC Class C | 1 | 1 | 0 | 0
  CDC Class B to CDC Class C | 0 | 0 | 0 | 0
  CDC Class C to new CDC Class C | 0 | 0 | 0 | 0
  CDC Class A, B or C to Death | 0 | 1 | 1 | 0

9. Secondary Outcome: Absolute Values for Cluster of Differentiation 4+ (CD4+) Cell Count During Double-blind Randomized Treatment Until Week 96
Description: CD4+ cell counts were assessed by flow cytometry. Baseline value is the last pre-treatment value observed.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Cells per cubic millimeter
  Baseline; n=60, 60, 61, 62 | 445.5 (155.60) | 444.9 (190.98) | 459.0 (170.64) | 456.5 (196.11)
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 544.0 (197.54) | 525.1 (181.29) | 549.3 (206.68) | 487.0 (222.84)
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | 580.5 (230.40) | 522.0 (205.80) | 545.8 (196.79) | 509.9 (198.21)
  Week 8; n=58, 56, 57, 55: number analyzed (Participants) | 58 | 56 | 57 | 55
  Week 8; n=58, 56, 57, 55 | 576.6 (196.55) | 555.2 (210.92) | 544.3 (176.01) | 531.4 (175.95)
  Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Week 12; n=58, 53, 57, 51 | 588.4 (208.15) | 599.0 (226.06) | 596.6 (181.00) | 564.3 (222.99)
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 608.3 (200.34) | 595.8 (197.47) | 599.7 (166.77) | 594.4 (212.63)
  Week 20; n=56, 54, 56, 49: number analyzed (Participants) | 56 | 54 | 56 | 49
  Week 20; n=56, 54, 56, 49 | 607.3 (204.87) | 607.4 (199.27) | 636.6 (225.04) | 607.7 (186.36)
  Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Week 24; n=56, 53, 56, 47 | 614.6 (194.13) | 626.5 (210.63) | 658.0 (253.19) | 599.5 (219.52)
  Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Week 26; n=48, 50, 53, 45 | 632.8 (210.93) | 629.5 (207.34) | 645.8 (188.61) | 625.7 (196.46)
  Week 28; n=49, 52, 52, 45: number analyzed (Participants) | 49 | 52 | 52 | 45
  Week 28; n=49, 52, 52, 45 | 652.2 (225.32) | 635.9 (217.52) | 653.3 (261.11) | 635.7 (224.72)
  Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 32; n=52, 53, 55, 45 | 638.1 (192.54) | 650.8 (209.66) | 665.2 (246.84) | 663.8 (257.25)
  Week 36; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 36; n=52, 53, 55, 45 | 638.7 (198.05) | 658.6 (226.51) | 720.3 (257.85) | 651.5 (212.15)
  Week 40; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 40; n=52, 53, 55, 45 | 650.2 (218.40) | 658.5 (204.08) | 667.6 (187.30) | 687.9 (241.35)
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 677.3 (219.75) | 687.2 (227.06) | 713.8 (215.70) | 732.6 (273.19)
  Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  Week 60; n=48, 47, 53, 44 | 668.1 (222.61) | 720.9 (268.74) | 719.8 (219.04) | 733.9 (238.90)
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 683.2 (242.75) | 651.3 (217.19) | 710.9 (259.89) | 722.5 (263.47)
  Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Week 84; n=46, 48, 52, 42 | 718.3 (212.59) | 736.9 (271.85) | 735.0 (236.25) | 744.7 (250.90)
  Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  Week 96; n=46, 46, 52, 41 | 726.2 (272.28) | 722.9 (246.22) | 743.1 (242.23) | 747.8 (263.27)

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count Over Time by Visit
Description: CD4+ cell counts were assessed by flow cytometry. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: as for outcome 7
Population: ITT-E Population.Participants randomized to Efavirenz 600 mg arm were considered to have completed their participation in the study after Week 96; hence were no longer followed as part of this study. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Cells per cubic millimeter
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 92.6 (112.44) | 79.5 (118.15) | 91.7 (127.92) | 24.8 (138.47)
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | 136.4 (157.36) | 76.9 (107.01) | 88.2 (110.01) | 46.0 (106.35)
  Week 8; n=58, 56, 57, 55: number analyzed (Participants) | 58 | 56 | 57 | 55
  Week 8; n=58, 56, 57, 55 | 129.9 (123.47) | 117.8 (132.19) | 90.5 (148.25) | 65.6 (120.25)
  Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Week 12; n=58, 53, 57, 51 | 140.5 (142.86) | 140.8 (165.02) | 145.2 (142.24) | 103.4 (125.39)
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 159.3 (115.36) | 142.2 (145.64) | 148.3 (131.81) | 135.5 (153.48)
  Week 20; n=56, 54, 56, 49: number analyzed (Participants) | 56 | 54 | 56 | 49
  Week 20; n=56, 54, 56, 49 | 165.2 (146.90) | 153.8 (150.40) | 182.6 (142.18) | 149.0 (117.44)
  Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Week 24; n=56, 53, 56, 47 | 172.5 (112.04) | 180.9 (161.43) | 204.0 (166.78) | 143.4 (145.18)
  Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Week 26; n=48, 50, 53, 45 | 186.4 (153.99) | 177.7 (146.84) | 194.7 (149.66) | 166.4 (145.11)
  Week 28; n=49, 52, 52, 45: number analyzed (Participants) | 49 | 52 | 52 | 45
  Week 28; n=49, 52, 52, 45 | 205.0 (164.91) | 188.1 (132.08) | 193.3 (154.43) | 178.2 (150.25)
  Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 32; n=52, 53, 55, 45 | 191.4 (151.79) | 205.2 (145.53) | 209.9 (157.56) | 197.4 (170.48)
  Week 36; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 36; n=52, 53, 55, 45 | 192.0 (165.97) | 213.0 (144.89) | 265.0 (169.42) | 185.2 (152.91)
  Week 40; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Week 40; n=52, 53, 55, 45 | 203.6 (171.74) | 212.8 (180.38) | 212.3 (114.67) | 221.5 (188.99)
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 235.1 (179.89) | 241.6 (182.90) | 259.0 (154.21) | 262.5 (201.33)
  Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  Week 60; n=48, 47, 53, 44 | 217.7 (152.92) | 269.4 (188.34) | 266.1 (156.03) | 263.8 (181.15)
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 232.0 (191.05) | 201.4 (206.54) | 254.0 (189.26) | 257.1 (216.41)
  Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Week 84; n=46, 48, 52, 42 | 261.5 (171.65) | 287.0 (207.10) | 278.1 (166.11) | 279.4 (191.30)
  Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  Week 96; n=46, 46, 52, 41 | 269.4 (204.32) | 267.5 (196.27) | 286.2 (181.50) | 281.7 (232.90)
  Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  Week 108; n=43, 46, 49, 0 | 296.2 (215.21) | 304.3 (195.30) | 288.4 (184.61) |
  Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  Week 120; n=41, 46, 49, 0 | 266.1 (173.09) | 279.3 (181.10) | 307.2 (225.39) |
  Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  Week 132; n=40, 46, 49, 0 | 297.1 (167.59) | 305.2 (184.98) | 313.2 (168.30) |
  Week 144; n=37, 45, 46, 0: number analyzed (Participants) | 37 | 45 | 46 | 0
  Week 144; n=37, 45, 46, 0 | 330.7 (225.42) | 308.9 (224.63) | 322.4 (224.57) |
  Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  Week 156; n=37, 42, 49, 0 | 334.5 (213.79) | 319.2 (182.15) | 320.4 (187.58) |
  Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  Week 168; n=35, 43, 47, 0 | 338.1 (252.13) | 332.4 (222.37) | 361.3 (198.98) |
  Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  Week 180; n=36, 41, 47, 0 | 338.0 (218.72) | 348.6 (203.73) | 384.2 (192.86) |
  Week 192; n=35, 40, 47, 0: number analyzed (Participants) | 35 | 40 | 47 | 0
  Week 192; n=35, 40, 47, 0 | 300.8 (168.24) | 351.0 (205.56) | 342.3 (204.83) |
  Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  Week 204; n=34, 39, 47, 0 | 369.5 (196.17) | 332.9 (179.28) | 340.0 (191.82) |
  Week 216; n=33, 39, 47, 0: number analyzed (Participants) | 33 | 39 | 47 | 0
  Week 216; n=33, 39, 47, 0 | 397.0 (202.03) | 373.4 (188.28) | 357.8 (199.87) |
  Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Week 228; n=32, 39, 47, 0 | 331.8 (168.64) | 366.5 (231.25) | 383.7 (253.17) |
  Week 240; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Week 240; n=32, 39, 47, 0 | 356.5 (195.99) | 395.9 (205.55) | 408.4 (201.05) |
  Week 252; n=31, 38, 47, 0: number analyzed (Participants) | 31 | 38 | 47 | 0
  Week 252; n=31, 38, 47, 0 | 400.3 (183.36) | 343.7 (196.09) | 383.1 (217.20) |
  Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  Week 264; n=32, 38, 47, 0 | 344.4 (160.38) | 365.0 (210.00) | 391.8 (222.00) |
  Week 276; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  Week 276; n=31, 38, 46, 0 | 398.3 (250.45) | 350.3 (210.98) | 362.2 (243.30) |
  Week 288; n=30, 38, 45, 0: number analyzed (Participants) | 30 | 38 | 45 | 0
  Week 288; n=30, 38, 45, 0 | 411.0 (161.93) | 383.5 (279.75) | 337.1 (187.13) |
  Week 300; n=30, 37, 44, 0: number analyzed (Participants) | 30 | 37 | 44 | 0
  Week 300; n=30, 37, 44, 0 | 437.7 (196.33) | 404.4 (239.11) | 353.5 (200.23) |
  Week 312; n=30, 34, 43, 0: number analyzed (Participants) | 30 | 34 | 43 | 0
  Week 312; n=30, 34, 43, 0 | 335.0 (176.73) | 433.0 (264.63) | 407.0 (178.06) |
  Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  Week 324; n=3, 4, 3, 0 | 402.0 (197.55) | 276.0 (278.28) | 272.0 (277.44) |

11. Secondary Outcome: Number of Participants With Treatment Emergent Phenotypic Resistance
Description: Plasma samples were collected for drug resistance testing. Phenotypic resistance data for the following drugs under integrase inhibitor (INI), non-nucleoside reverse transcriptase inhibitor (NNRTI), NRTI and proteasome inhibitor drug classes is presented for participants with confirmed virologic failure: GSK1265744, Raltegravir [RAL], Delavirdine [DLV], Efavirenz [EFV], Etravirine [ETR], Nevirapine (NVP), RPV, 3TC, ABC, FTC, TDF, Zidovudine [ZDV], Stavudine [d4T], Didanosine [ddI], Atazanavir/ritonavir [ATV/r], Darunavir (DRV)/r, Fosamprenavir/r [FPV/r], Indinavir/r [IDV/r], Lopinavir/r [LPV/r], Nelfinavir [NFV], Ritonavir [RTV], Saquinavir/r [SQV/r], Tipranavir/r [TPV/r]. On-treatment Phenotypic Resistance population comprised of all participants in the ITT-E Population with available on-treatment phenotypic resistance data, excluding participants who are not protocol-defined virologic failures.
Time Frame: Up to Week 324
Population: On-treatment Phenotypic Resistance Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 6 | 2 | 2 | 5
Participants
  INI, GSK1265744; Resistant; n=5, 1, 2, 2: number analyzed (Participants) | 5 | 1 | 2 | 2
  INI, GSK1265744; Resistant; n=5, 1, 2, 2 | 2 | 0 | 1 | 0
  INI, GSK1265744; Sensitive; n=5, 1, 2, 2: number analyzed (Participants) | 5 | 1 | 2 | 2
  INI, GSK1265744; Sensitive; n=5, 1, 2, 2 | 3 | 1 | 1 | 2
  INI, RAL; Resistant; n=5, 1, 2, 2: number analyzed (Participants) | 5 | 1 | 2 | 2
  INI, RAL; Resistant; n=5, 1, 2, 2 | 3 | 0 | 1 | 0
  INI, RAL; Sensitive; n=5, 1, 2, 2: number analyzed (Participants) | 5 | 1 | 2 | 2
  INI, RAL; Sensitive; n=5, 1, 2, 2 | 2 | 1 | 1 | 2
  NNRTI, DLV; Resistant; n=6, 2, 2, 5 | 3 | 0 | 0 | 0
  NNRTI, DLV; Sensitive; n=6, 2, 2, 5 | 3 | 2 | 2 | 5
  NNRTI, EFV; Resistant; n=6, 2, 2, 5 | 3 | 0 | 0 | 0
  NNRTI, EFV; Sensitive; n=6, 2, 2, 5 | 3 | 2 | 2 | 5
  NNRTI, ETR; Resistant; n=6, 2, 2, 5 | 3 | 0 | 0 | 0
  NNRTI, ETR; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NNRTI, ETR; Sensitive; n=6, 2, 2, 5 | 3 | 2 | 2 | 5
  NNRTI, NVP; Resistant; n=6, 2, 2, 5 | 3 | 0 | 0 | 0
  NNRTI, NVP; Sensitive; n=6, 2, 2, 5 | 3 | 2 | 2 | 5
  NNRTI, RPV; Resistant; n=6, 2, 2, 5 | 3 | 0 | 0 | 0
  NNRTI, RPV; Sensitive; n=6, 2, 2, 5 | 3 | 2 | 2 | 5
  NRTI, 3TC; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, 3TC; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  NRTI, ABC; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, ABC; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, ABC; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  NRTI, FTC; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, FTC; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  NRTI, TDF; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, TDF; Partially sensitive; n=6, 2, 2, 5 | 1 | 0 | 0 | 0
  NRTI, TDF; Sensitive; n=6, 2, 2, 5 | 5 | 2 | 2 | 5
  NRTI, ZDV; Resistant; n=6, 2, 2, 5 | 2 | 0 | 0 | 0
  NRTI, ZDV; Sensitive; n=6, 2, 2, 5 | 4 | 2 | 2 | 5
  NRTI, d4T; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, d4T; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  NRTI, ddI; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, ddI; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  NRTI, ddI; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, ATV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, ATV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, DRV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, DRV/r; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, DRV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, FPV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, FPV/r; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, FPV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, IDV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, IDV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, LPV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, LPV/r; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, LPV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, NFV; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, NFV; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, RTV; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, RTV; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, SQV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, SQV/r; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, SQV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5
  PI, TPV/r; Resistant; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, TPV/r; Partially sensitive; n=6, 2, 2, 5 | 0 | 0 | 0 | 0
  PI, TPV/r; Sensitive; n=6, 2, 2, 5 | 6 | 2 | 2 | 5

12. Secondary Outcome: Number of Participants With Treatment Emergent Genotypic Mutations Associated With Development of Resistance
Description: Plasma samples were collected for drug resistance testing. The treatment emergent INI mutations associated with development of resistance to RAL, ELV, dolutegravir (DTG) or GSK1265744 and major resistance mutations to other classes (NRTI, NNRTI, PI) as defined by International AIDS society (IAS)-United States of America (USA) are presented. On-treatment Genotypic Resistance population comprised of all participants in the ITT-E Population with available on-treatment genotypic resistance data, excluding participants who are not protocol-defined virologic failures.
Time Frame: Up to Week 324
Population: On-treatment Genotypic resistance Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 6 | 2 | 2 | 5
Participants
  Any INI mutation | 3 | 0 | 1 | 0
  Any mutation to other classes | 4 | 0 | 1 | 0

13. Secondary Outcome: Number of Participants With Adherence to Study Treatment
Description: Number of participants with >=90% adherence to study treatment based on pill count is summarized.
Time Frame: Baseline (Day 1), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300 and 312
Population: ITT-E Population. Only participants who were dispensed and returned drug on scheduled visits were included in the analysis (represented by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 57 | 55 | 56 | 52
Participants
  Baseline; n=57, 55, 56, 52 | 53 | 51 | 55 | 48
  Week 4; n=54, 52, 53, 50: number analyzed (Participants) | 54 | 52 | 53 | 50
  Week 4; n=54, 52, 53, 50 | 46 | 49 | 52 | 44
  Week 8; n=53, 50, 56, 48: number analyzed (Participants) | 53 | 50 | 56 | 48
  Week 8; n=53, 50, 56, 48 | 49 | 45 | 53 | 47
  Week 12; n=55, 48, 53, 48: number analyzed (Participants) | 55 | 48 | 53 | 48
  Week 12; n=55, 48, 53, 48 | 44 | 40 | 46 | 43
  Week 16; n=53, 51, 53, 44: number analyzed (Participants) | 53 | 51 | 53 | 44
  Week 16; n=53, 51, 53, 44 | 44 | 45 | 50 | 42
  Week 20; n=51, 49, 55, 44: number analyzed (Participants) | 51 | 49 | 55 | 44
  Week 20; n=51, 49, 55, 44 | 45 | 40 | 51 | 41
  Week 24; n=51, 46, 51, 43: number analyzed (Participants) | 51 | 46 | 51 | 43
  Week 24; n=51, 46, 51, 43 | 47 | 41 | 48 | 39
  Week 28; n=49, 48, 53, 41: number analyzed (Participants) | 49 | 48 | 53 | 41
  Week 28; n=49, 48, 53, 41 | 45 | 46 | 48 | 35
  Week 32; n=47, 48, 55, 41: number analyzed (Participants) | 47 | 48 | 55 | 41
  Week 32; n=47, 48, 55, 41 | 46 | 42 | 52 | 37
  Week 36; n=46, 48, 50, 41: number analyzed (Participants) | 46 | 48 | 50 | 41
  Week 36; n=46, 48, 50, 41 | 40 | 43 | 48 | 36
  Week 40; n=38, 35, 45, 39: number analyzed (Participants) | 38 | 35 | 45 | 39
  Week 40; n=38, 35, 45, 39 | 33 | 30 | 41 | 34
  Week 48; n=33, 37, 45, 35: number analyzed (Participants) | 33 | 37 | 45 | 35
  Week 48; n=33, 37, 45, 35 | 32 | 33 | 41 | 33
  Week 60; n=38, 38, 40, 37: number analyzed (Participants) | 38 | 38 | 40 | 37
  Week 60; n=38, 38, 40, 37 | 37 | 35 | 37 | 35
  Week 72; n=35, 37, 44, 32: number analyzed (Participants) | 35 | 37 | 44 | 32
  Week 72; n=35, 37, 44, 32 | 32 | 35 | 41 | 27
  Week 84; n=36, 39, 42, 33: number analyzed (Participants) | 36 | 39 | 42 | 33
  Week 84; n=36, 39, 42, 33 | 34 | 36 | 39 | 29
  Week 96; n=31, 36, 33, 0: number analyzed (Participants) | 31 | 36 | 33 | 0
  Week 96; n=31, 36, 33, 0 | 25 | 32 | 30 |
  Week 108; n=23, 23, 29, 0: number analyzed (Participants) | 23 | 23 | 29 | 0
  Week 108; n=23, 23, 29, 0 | 21 | 20 | 27 |
  Week 120; n=30, 38, 41, 0: number analyzed (Participants) | 30 | 38 | 41 | 0
  Week 120; n=30, 38, 41, 0 | 28 | 36 | 39 |
  Week 132; n=29, 32, 40, 0: number analyzed (Participants) | 29 | 32 | 40 | 0
  Week 132; n=29, 32, 40, 0 | 28 | 30 | 35 |
  Week 144; n=33, 34, 43, 0: number analyzed (Participants) | 33 | 34 | 43 | 0
  Week 144; n=33, 34, 43, 0 | 32 | 29 | 41 |
  Week 156; n=31, 28, 39, 0: number analyzed (Participants) | 31 | 28 | 39 | 0
  Week 156; n=31, 28, 39, 0 | 30 | 25 | 35 |
  Week 168; n=29, 33, 41, 0: number analyzed (Participants) | 29 | 33 | 41 | 0
  Week 168; n=29, 33, 41, 0 | 29 | 24 | 35 |
  Week 180; n=26, 29, 39, 0: number analyzed (Participants) | 26 | 29 | 39 | 0
  Week 180; n=26, 29, 39, 0 | 24 | 24 | 34 |
  Week 192; n=30, 30, 39, 0: number analyzed (Participants) | 30 | 30 | 39 | 0
  Week 192; n=30, 30, 39, 0 | 28 | 27 | 35 |
  Week 204; n=29, 32, 38, 0: number analyzed (Participants) | 29 | 32 | 38 | 0
  Week 204; n=29, 32, 38, 0 | 27 | 26 | 33 |
  Week 216; n=29, 30, 37, 0: number analyzed (Participants) | 29 | 30 | 37 | 0
  Week 216; n=29, 30, 37, 0 | 29 | 27 | 31 |
  Week 228; n=27, 34, 40, 0: number analyzed (Participants) | 27 | 34 | 40 | 0
  Week 228; n=27, 34, 40, 0 | 25 | 28 | 35 |
  Week 240; n=28, 26, 41, 0: number analyzed (Participants) | 28 | 26 | 41 | 0
  Week 240; n=28, 26, 41, 0 | 28 | 22 | 35 |
  Week 252; n=23, 26, 33, 0: number analyzed (Participants) | 23 | 26 | 33 | 0
  Week 252; n=23, 26, 33, 0 | 18 | 21 | 29 |
  Week 264; n=15, 18, 24, 0: number analyzed (Participants) | 15 | 18 | 24 | 0
  Week 264; n=15, 18, 24, 0 | 12 | 16 | 21 |
  Week 276; n=14, 14, 21, 0: number analyzed (Participants) | 14 | 14 | 21 | 0
  Week 276; n=14, 14, 21, 0 | 13 | 13 | 18 |
  Week 288; n=12, 14, 18, 0: number analyzed (Participants) | 12 | 14 | 18 | 0
  Week 288; n=12, 14, 18, 0 | 12 | 10 | 17 |
  Week 300; n=12, 13, 20, 0: number analyzed (Participants) | 12 | 13 | 20 | 0
  Week 300; n=12, 13, 20, 0 | 11 | 7 | 18 |
  Week 312; n=1, 1, 0, 0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Week 312; n=1, 1, 0, 0 | 1 | 1 |  |

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 16 and Week 24 Using MSDF Algorithm-Induction Phase
Description: as for outcome 4
Time Frame: Week 16 and Week 24
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants
  Week 16 | 90 [82 to 98] | 83 [74 to 93] | 87 [78 to 95] | 74 [63 to 85]
  Week 24 | 87 [78 to 95] | 85 [76 to 94] | 87 [78 to 95] | 74 [63 to 85]

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL From Week 24 Through Week 96 by Visit Using MSDF Algorithm-Maintenance Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The end point was determined using MSDF algorithm based on the current US FDA definition of Snapshot algorithm. This algorithm treats all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to visit window) as well as participants who switch their concomitant antiretroviral therapy prior to the visit of interest as non-responders. Virological response within an analysis window was determined by the last available HIV-1 RNA measurement in that window while the participant was on-treatment. MSDF response rate was calculated as number of responders in the analysis window divided by the number of participants in the analysis population. ITT-Maintenance Exposed (ME) Population comprised of all participants randomized to GSK1265744 and who received at least one dose of investigational product during maintenance phase of the study.
Time Frame: Weeks 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: ITT-ME Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 52 | 53 | 55 | 47
Percentage of participants
  Week 24 | 96 | 94 | 96 | 96
  Week 26 | 90 | 85 | 95 | 87
  Week 28 | 98 | 89 | 95 | 91
  Week 32 | 96 | 91 | 96 | 91
  Week 36 | 98 | 92 | 95 | 94
  Week 40 | 96 | 92 | 95 | 89
  Week 48 | 92 | 91 | 96 | 94
  Week 60 | 90 | 83 | 95 | 89
  Week 72 | 83 | 83 | 95 | 89
  Week 84 | 83 | 85 | 95 | 89
  Week 96 | 79 | 85 | 93 | 83

16. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Maintenance Phase
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes mentioned before; all events of possible drug-induced liver injury with hyperbilirubinemia. Maintenance Safety Population comprised of all participants randomized to GSK1265744 and who were exposed to investigational products during the maintenance phase of the study with the exception of any participants with documented evidence of not having consumed any amount of investigational product.
Time Frame: Week 24 to Week 96
Population: Maintenance Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 52 | 53 | 55 | 47
Participants
  Any AE | 40 | 50 | 50 | 35
  Any SAE | 5 | 5 | 5 | 2

17. Secondary Outcome: Number of Participants With Maximum Treatment-emergent Clinical Chemistry Toxicities-Maintenance Phase
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: alanine aminotranferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), carbon dioxide(CO2)/bicarbonate, cholesterol, creatine kinase (CK), creatinine, glucose, low density lipoprotein (LDL) cholesterol, lipase, inorganic phosphorus, potassium, sodium, total bilirubin and triglycerides. A toxicity is considered treatment emergent if it developed or increased in intensity from Baseline while on-treatment. Laboratory toxicities were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=Mild, Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening.
Time Frame: Week 24 to Week 96
Population: Maintenance Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 52 | 53 | 55 | 47
Participants
  ALT; Grade 1 | 9 | 12 | 17 | 6
  ALT; Grade 2 | 6 | 6 | 5 | 3
  ALT; Grade 3 | 0 | 1 | 0 | 0
  ALT; Grade 4 | 1 | 1 | 0 | 1
  Albumin; Grade 1 | 0 | 1 | 0 | 0
  Albumin; Grade 2 | 0 | 0 | 0 | 0
  Albumin; Grade 3 | 0 | 0 | 0 | 0
  Albumin; Grade 4 | 0 | 0 | 0 | 0
  ALP; Grade 1 | 2 | 1 | 4 | 4
  ALP; Grade 2 | 0 | 1 | 0 | 0
  ALP; Grade 3 | 0 | 0 | 0 | 0
  ALP; Grade 4 | 0 | 0 | 0 | 0
  AST; Grade 1 | 5 | 13 | 13 | 5
  AST; Grade 2 | 5 | 8 | 5 | 2
  AST; Grade 3 | 2 | 0 | 2 | 3
  AST; Grade 4 | 2 | 1 | 0 | 2
  CO2/bicarbonate; Grade 1 | 6 | 14 | 9 | 8
  CO2/bicarbonate; Grade 2 | 1 | 0 | 0 | 1
  CO2/bicarbonate; Grade 3 | 0 | 0 | 0 | 0
  CO2/bicarbonate; Grade 4 | 0 | 0 | 0 | 0
  Cholesterol; Grade 1 | 17 | 17 | 19 | 9
  Cholesterol; Grade 2 | 6 | 12 | 15 | 10
  Cholesterol; Grade 3 | 3 | 0 | 3 | 4
  Cholesterol; Grade 4 | 0 | 0 | 0 | 0
  CK; Grade 1 | 8 | 9 | 11 | 5
  CK; Grade 2 | 2 | 4 | 4 | 0
  CK; Grade 3 | 3 | 2 | 4 | 3
  CK; Grade 4 | 6 | 6 | 5 | 5
  Creatinine; Grade 1 | 1 | 1 | 2 | 1
  Creatinine; Grade 2 | 1 | 0 | 0 | 0
  Creatinine; Grade 3 | 0 | 0 | 0 | 0
  Creatinine; Grade 4 | 0 | 0 | 0 | 0
  Glucose; Grade 1 | 17 | 17 | 20 | 11
  Glucose; Grade 2 | 14 | 10 | 11 | 5
  Glucose; Grade 3 | 0 | 0 | 2 | 0
  Glucose; Grade 4 | 0 | 0 | 0 | 0
  LDL cholesterol; Grade 1 | 14 | 16 | 13 | 8
  LDL cholesterol; Grade 2 | 6 | 11 | 14 | 6
  LDL cholesterol; Grade 3 | 4 | 2 | 7 | 4
  LDL cholesterol; Grade 4 | 0 | 0 | 0 | 0
  Lipase; Grade 1 | 9 | 9 | 8 | 9
  Lipase; Grade 2 | 9 | 8 | 11 | 7
  Lipase; Grade 3 | 5 | 1 | 6 | 0
  Lipase; Grade 4 | 2 | 0 | 2 | 0
  Inorganic phosphorus; Grade 1 | 5 | 3 | 9 | 7
  Inorganic phosphorus; Grade 2 | 10 | 11 | 5 | 9
  Inorganic phosphorus; Grade 3 | 2 | 1 | 5 | 2
  Inorganic phosphorus; Grade 4 | 0 | 0 | 0 | 0
  Potassium; Grade 1 | 12 | 7 | 8 | 4
  Potassium; Grade 2 | 0 | 0 | 0 | 1
  Potassium; Grade 3 | 0 | 0 | 0 | 0
  Potassium; Grade 4 | 0 | 0 | 0 | 0
  Sodium; Grade 1 | 14 | 12 | 16 | 7
  Sodium; Grade 2 | 2 | 1 | 0 | 1
  Sodium; Grade 3 | 0 | 0 | 0 | 0
  Sodium; Grade 4 | 0 | 0 | 0 | 0
  Total bilirubin; Grade 1 | 7 | 1 | 8 | 0
  Total bilirubin; Grade 2 | 2 | 3 | 4 | 0
  Total bilirubin; Grade 3 | 0 | 1 | 0 | 0
  Total bilirubin; Grade 4 | 0 | 0 | 0 | 0
  Triglycerides; Grade 1 | 0 | 0 | 0 | 0
  Triglycerides; Grade 2 | 1 | 4 | 3 | 1
  Triglycerides; Grade 3 | 1 | 0 | 3 | 1
  Triglycerides; Grade 4 | 0 | 0 | 1 | 0

18. Secondary Outcome: Number of Participants With Maximum Treatment-emergent Hematology Toxicities-Maintenance Phase
Description: Blood samples were collected for the analysis of following hematology parameters: Activated Partial Thromboplastin Time (APTT), hemoglobin, international normalized ratio (INR), platelet count, prothrombin time (PT), total neutrophils and white blood cell (WBC) count. A toxicity is considered treatment emergent if it developed or increased in intensity from Baseline while on-treatment. Laboratory toxicities were graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=Mild, Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening.
Time Frame: Week 24 to Week 96
Population: Maintenance Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 52 | 53 | 55 | 47
Participants
  APTT; Grade 1 | 5 | 5 | 5 | 5
  APTT; Grade 2 | 0 | 1 | 0 | 0
  APTT; Grade 3 | 0 | 0 | 0 | 0
  APTT; Grade 4 | 1 | 1 | 1 | 1
  Hemoglobin; Grade 1 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 2 | 1 | 0 | 0 | 0
  Hemoglobin; Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 4 | 0 | 0 | 0 | 0
  INR; Grade 1 | 2 | 4 | 0 | 3
  INR; Grade 2 | 0 | 1 | 1 | 1
  INR; Grade 3 | 1 | 0 | 0 | 0
  INR; Grade 4 | 0 | 1 | 0 | 0
  Platelet count; Grade 1 | 4 | 0 | 4 | 1
  Platelet count; Grade 2 | 0 | 0 | 1 | 0
  Platelet count; Grade 3 | 0 | 0 | 1 | 0
  Platelet count; Grade 4 | 0 | 0 | 1 | 0
  PT; Grade 1 | 1 | 3 | 0 | 3
  PT; Grade 2 | 0 | 0 | 0 | 1
  PT; Grade 3 | 0 | 1 | 1 | 0
  PT; Grade 4 | 0 | 1 | 0 | 0
  Total neutrophils; Grade 1 | 7 | 9 | 10 | 2
  Total neutrophils; Grade 2 | 5 | 2 | 3 | 3
  Total neutrophils; Grade 3 | 1 | 0 | 1 | 1
  Total neutrophils; Grade 4 | 1 | 1 | 3 | 1
  WBC count; Grade 1 | 2 | 5 | 2 | 3
  WBC count; Grade 2 | 1 | 1 | 1 | 0
  WBC count; Grade 3 | 0 | 0 | 1 | 0
  WBC count; Grade 4 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With AEs and SAEs Over Time
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes mentioned before; all events of possible drug-induced liver injury with hyperbilirubinemia. Safety Population comprised of all randomized participants who were exposed to investigational products with the exception of any participants with documented evidence of not having consumed any amount of investigational product.
Time Frame: Up to Week 324
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  Any AE | 57 | 57 | 60 | 60
  Any SAE | 13 | 12 | 11 | 4

20. Secondary Outcome: Number of Participants With Maximum Treatment-emergent Clinical Chemistry Toxicities Over Time
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: ALT, albumin, ALP, AST, CO2/bicarbonate, cholesterol, CK, creatinine, glucose, LDL cholesterol, lipase, inorganic phosphorus, potassium, sodium, total bilirubin and triglycerides. Laboratory toxicities were graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=Mild, Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening.
Time Frame: Up to Week 324
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  ALT; Grade 1 | 9 | 12 | 19 | 8
  ALT; Grade 2 | 6 | 6 | 5 | 4
  ALT; Grade 3 | 0 | 1 | 0 | 0
  ALT; Grade 4 | 1 | 1 | 2 | 1
  Albumin; Grade 1 | 0 | 1 | 0 | 0
  Albumin; Grade 2 | 0 | 0 | 0 | 0
  Albumin; Grade 3 | 0 | 0 | 0 | 0
  Albumin; Grade 4 | 0 | 0 | 0 | 0
  ALP; Grade 1 | 2 | 1 | 4 | 5
  ALP; Grade 2 | 0 | 1 | 0 | 0
  ALP; Grade 3 | 0 | 0 | 0 | 0
  ALP; Grade 4 | 0 | 0 | 0 | 0
  AST; Grade 1 | 7 | 13 | 15 | 7
  AST; Grade 2 | 6 | 8 | 5 | 2
  AST; Grade 3 | 2 | 0 | 4 | 3
  AST; Grade 4 | 2 | 1 | 0 | 2
  CO2/bicarbonate; Grade 1 | 6 | 14 | 9 | 8
  CO2/bicarbonate; Grade 2 | 1 | 0 | 0 | 1
  CO2/bicarbonate; Grade 3 | 0 | 0 | 0 | 0
  CO2/bicarbonate; Grade 4 | 0 | 0 | 0 | 0
  Cholesterol; Grade 1 | 17 | 17 | 19 | 9
  Cholesterol; Grade 2 | 7 | 12 | 15 | 10
  Cholesterol; Grade 3 | 3 | 0 | 3 | 6
  Cholesterol; Grade 4 | 0 | 0 | 0 | 0
  CK; Grade 1 | 9 | 10 | 12 | 5
  CK; Grade 2 | 2 | 4 | 4 | 0
  CK; Grade 3 | 3 | 2 | 4 | 4
  CK; Grade 4 | 7 | 6 | 5 | 5
  Creatinine; Grade 1 | 1 | 1 | 2 | 1
  Creatinine; Grade 2 | 1 | 0 | 0 | 1
  Creatinine; Grade 3 | 0 | 0 | 0 | 0
  Creatinine; Grade 4 | 0 | 0 | 0 | 0
  Glucose; Grade 1 | 19 | 18 | 21 | 12
  Glucose; Grade 2 | 14 | 10 | 11 | 6
  Glucose; Grade 3 | 0 | 0 | 2 | 0
  Glucose; Grade 4 | 0 | 0 | 0 | 1
  LDL cholesterol; Grade 1 | 14 | 17 | 13 | 8
  LDL cholesterol; Grade 2 | 7 | 11 | 14 | 7
  LDL cholesterol; Grade 3 | 4 | 2 | 7 | 4
  LDL cholesterol; Grade 4 | 0 | 0 | 0 | 0
  Lipase; Grade 1 | 11 | 9 | 9 | 10
  Lipase; Grade 2 | 9 | 8 | 11 | 7
  Lipase; Grade 3 | 5 | 2 | 6 | 1
  Lipase; Grade 4 | 2 | 0 | 2 | 0
  Inorganic phosphorus; Grade 1 | 5 | 3 | 10 | 8
  Inorganic phosphorus; Grade 2 | 11 | 11 | 6 | 9
  Inorganic phosphorus; Grade 3 | 2 | 1 | 5 | 2
  Inorganic phosphorus; Grade 4 | 0 | 0 | 0 | 0
  Potassium; Grade 1 | 14 | 7 | 8 | 4
  Potassium; Grade 2 | 0 | 0 | 0 | 1
  Potassium; Grade 3 | 0 | 0 | 0 | 0
  Potassium; Grade 4 | 0 | 0 | 0 | 0
  Sodium; Grade 1 | 14 | 12 | 16 | 11
  Sodium; Grade 2 | 2 | 1 | 0 | 1
  Sodium; Grade 3 | 0 | 0 | 0 | 0
  Sodium; Grade 4 | 0 | 0 | 0 | 0
  Total bilirubin; Grade 1 | 7 | 1 | 8 | 0
  Total bilirubin; Grade 2 | 2 | 3 | 4 | 0
  Total bilirubin; Grade 3 | 0 | 1 | 0 | 0
  Total bilirubin; Grade 4 | 0 | 0 | 0 | 0
  Triglycerides; Grade 1 | 0 | 0 | 0 | 0
  Triglycerides; Grade 2 | 1 | 4 | 3 | 1
  Triglycerides; Grade 3 | 1 | 0 | 3 | 1
  Triglycerides; Grade 4 | 0 | 0 | 1 | 1

21. Secondary Outcome: Number of Participants With Maximum Treatment-emergent Hematology Toxicities Over Time
Description: Blood samples were collected for the analysis of following hematology parameters: APTT, hemoglobin, INR, platelet count, PT, total neutrophils and WBC count. Laboratory toxicities were graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=Mild, Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening.
Time Frame: Up to Week 324
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  APTT; Grade 1 | 5 | 5 | 5 | 5
  APTT; Grade 2 | 0 | 1 | 0 | 0
  APTT; Grade 3 | 0 | 0 | 0 | 0
  APTT; Grade 4 | 1 | 1 | 1 | 1
  Hemoglobin; Grade 1 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 2 | 1 | 0 | 0 | 0
  Hemoglobin; Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 4 | 0 | 0 | 0 | 0
  INR; Grade 1 | 2 | 4 | 0 | 3
  INR; Grade 2 | 0 | 1 | 1 | 1
  INR; Grade 3 | 1 | 0 | 0 | 0
  INR; Grade 4 | 0 | 1 | 0 | 0
  Platelet count; Grade 1 | 4 | 0 | 4 | 1
  Platelet count; Grade 2 | 0 | 0 | 1 | 0
  Platelet count; Grade 3 | 0 | 0 | 1 | 0
  Platelet count; Grade 4 | 0 | 0 | 1 | 0
  PT; Grade 1 | 1 | 3 | 0 | 3
  PT; Grade 2 | 0 | 0 | 0 | 1
  PT; Grade 3 | 0 | 1 | 1 | 0
  PT; Grade 4 | 0 | 1 | 0 | 0
  Total neutrophils; Grade 1 | 7 | 9 | 10 | 2
  Total neutrophils; Grade 2 | 5 | 2 | 3 | 3
  Total neutrophils; Grade 3 | 1 | 0 | 1 | 1
  Total neutrophils; Grade 4 | 1 | 1 | 3 | 1
  WBC count; Grade 1 | 2 | 5 | 2 | 3
  WBC count; Grade 2 | 1 | 1 | 1 | 0
  WBC count; Grade 3 | 0 | 0 | 1 | 0
  WBC count; Grade 4 | 0 | 0 | 0 | 0

22. Secondary Outcome: Absolute Values for ALT, AST, CK During Double-blind Randomized Treatment Until Week 96
Description: Blood samples were collected for the analysis of ALT, AST and CK. Baseline value is the last pre-treatment value observed.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Mean (Standard Deviation); unit: International Units per Liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
International Units per Liter
  ALT; Baseline; n=60, 60, 61, 62 | 23.9 (12.38) | 28.1 (17.65) | 28.5 (20.60) | 30.5 (29.21)
  ALT; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  ALT; Week 2; n=58, 56, 58, 58 | 24.0 (13.29) | 26.3 (17.81) | 27.2 (14.49) | 30.0 (26.73)
  ALT; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  ALT; Week 4; n=58, 57, 59, 57 | 23.1 (14.31) | 25.6 (17.29) | 30.3 (24.25) | 31.4 (27.43)
  ALT; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  ALT; Week 8; n=58, 55, 57, 54 | 25.4 (16.06) | 29.3 (23.15) | 35.9 (63.11) | 25.0 (13.21)
  ALT; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  ALT; Week 12; n=58, 53, 57, 51 | 25.0 (15.37) | 31.4 (28.65) | 26.6 (16.27) | 25.7 (17.44)
  ALT; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  ALT; Week 16; n=57, 54, 57, 52 | 26.0 (25.88) | 28.5 (27.79) | 26.9 (18.68) | 30.4 (22.55)
  ALT; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  ALT; Week 20; n=56, 54, 55, 49 | 22.3 (11.62) | 24.9 (15.72) | 30.3 (24.34) | 27.0 (15.71)
  ALT; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  ALT; Week 24; n=56, 53, 56, 47 | 20.9 (9.86) | 27.5 (23.90) | 28.6 (19.62) | 25.7 (13.31)
  ALT; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  ALT; Week 26; n=48, 50, 53, 45 | 24.2 (16.54) | 26.6 (26.63) | 23.5 (10.77) | 28.3 (25.23)
  ALT; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  ALT; Week 28; n=51, 52, 52, 45 | 20.4 (11.47) | 26.5 (26.66) | 24.8 (14.94) | 24.2 (13.67)
  ALT; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  ALT; Week 32; n=52, 53, 55, 45 | 19.5 (9.83) | 26.9 (27.66) | 23.2 (14.67) | 23.1 (10.19)
  ALT; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  ALT; Week 36; n=52, 52, 55, 45 | 23.4 (26.79) | 24.7 (17.44) | 24.2 (15.60) | 23.5 (10.53)
  ALT; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  ALT; Week 40; n=52, 53, 55, 44 | 22.7 (18.13) | 24.6 (15.43) | 25.8 (23.50) | 23.4 (10.92)
  ALT; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  ALT; Week 48; n=51, 53, 54, 44 | 18.4 (8.32) | 24.8 (15.91) | 24.8 (19.60) | 22.6 (10.92)
  ALT; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  ALT; Week 60; n=48, 47, 53, 44 | 21.4 (17.70) | 25.9 (16.69) | 28.1 (26.70) | 24.9 (13.59)
  ALT; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  ALT; Week 72; n=47, 47, 52, 42 | 19.9 (9.98) | 30.7 (28.68) | 26.3 (20.29) | 22.7 (9.62)
  ALT; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  ALT; Week 84; n=46, 48, 52, 42 | 20.1 (11.56) | 29.9 (20.77) | 25.3 (19.53) | 27.1 (32.55)
  ALT; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  ALT; Week 96; n=45, 48, 52, 40 | 22.0 (18.20) | 48.7 (153.96) | 25.5 (21.23) | 24.3 (22.84)
  AST; Baseline; n=60, 60, 61, 62 | 25.0 (7.36) | 27.5 (11.15) | 28.1 (12.01) | 31.5 (28.43)
  AST; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  AST; Week 2; n=58, 56, 58, 58 | 25.6 (8.36) | 26.6 (11.38) | 26.8 (8.60) | 32.8 (51.17)
  AST; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  AST; Week 4; n=58, 57, 59, 57 | 24.0 (7.95) | 25.0 (11.37) | 28.3 (16.29) | 29.0 (15.61)
  AST; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  AST; Week 8; n=58, 55, 57, 54 | 28.7 (31.34) | 29.5 (23.47) | 32.8 (37.43) | 24.4 (5.73)
  AST; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  AST; Week 12; n=58, 53, 57, 51 | 26.3 (13.40) | 29.0 (24.56) | 25.5 (8.05) | 24.4 (9.49)
  AST; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  AST; Week 16; n=57, 54, 57, 52 | 24.2 (12.70) | 29.2 (24.00) | 26.5 (9.42) | 36.7 (71.83)
  AST; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  AST; Week 20; n=56, 54, 55, 49 | 26.0 (20.71) | 24.2 (10.38) | 31.7 (26.31) | 28.7 (28.75)
  AST; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  AST; Week 24; n=56, 53, 56, 47 | 23.3 (8.93) | 27.2 (17.43) | 28.6 (14.12) | 26.1 (9.61)
  AST; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  AST; Week 26; n=48, 50, 53, 45 | 28.4 (28.28) | 26.9 (18.86) | 24.5 (6.64) | 25.8 (12.21)
  AST; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  AST; Week 28; n=51, 52, 52, 45 | 22.6 (8.77) | 26.7 (16.58) | 25.5 (11.24) | 23.7 (7.89)
  AST; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  AST; Week 32; n=52, 53, 55, 45 | 21.9 (7.74) | 26.5 (19.14) | 25.6 (9.19) | 25.4 (12.33)
  AST; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  AST; Week 36; n=52, 52, 55, 45 | 29.2 (39.15) | 25.4 (12.50) | 26.4 (11.38) | 26.3 (13.66)
  AST; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  AST; Week 40; n=52, 53, 55, 44 | 24.7 (14.04) | 24.5 (10.35) | 26.5 (14.21) | 23.0 (6.17)
  AST; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  AST; Week 48; n=51, 53, 54, 44 | 21.4 (8.02) | 24.3 (12.32) | 24.2 (9.26) | 23.7 (8.45)
  AST; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  AST; Week 60; n=48, 47, 53, 44 | 23.4 (10.41) | 25.3 (12.77) | 30.4 (21.00) | 24.9 (8.31)
  AST; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  AST; Week 72; n=47, 47, 52, 42 | 21.8 (7.67) | 31.0 (22.80) | 26.4 (10.52) | 22.9 (6.28)
  AST; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  AST; Week 84; n=46, 48, 52, 42 | 22.3 (8.10) | 29.2 (16.93) | 25.2 (9.11) | 29.9 (37.33)
  AST; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  AST; Week 96; n=45, 48, 52, 40 | 23.6 (22.38) | 47.7 (150.51) | 25.9 (12.90) | 27.7 (35.71)
  CK; Baseline; n=60, 60, 61, 62 | 197.3 (178.83) | 295.9 (604.02) | 181.2 (217.99) | 349.8 (1521.09)
  CK; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  CK; Week 2; n=58, 56, 58, 58 | 237.9 (271.07) | 276.1 (468.74) | 184.8 (143.83) | 512.1 (2788.37)
  CK; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  CK; Week 4; n=58, 57, 59, 57 | 196.7 (159.74) | 221.8 (426.95) | 180.5 (174.80) | 236.2 (563.36)
  CK; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  CK; Week 8; n=58, 55, 57, 54 | 413.3 (1523.18) | 427.2 (1518.27) | 451.7 (1788.60) | 152.9 (94.19)
  CK; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  CK; Week 12; n=58, 53, 57, 51 | 316.1 (570.21) | 314.7 (1116.09) | 211.8 (174.07) | 161.2 (163.26)
  CK; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  CK; Week 16; n=57, 54, 57, 52 | 195.1 (180.51) | 427.3 (1339.99) | 213.3 (190.94) | 646.5 (3471.23)
  CK; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  CK; Week 20; n=56, 54, 55, 49 | 342.7 (953.66) | 202.1 (309.41) | 485.3 (1835.11) | 528.2 (2643.29)
  CK; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  CK; Week 24; n=56, 53, 56, 47 | 226.0 (230.13) | 306.3 (690.18) | 243.0 (228.95) | 247.4 (498.72)
  CK; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  CK; Week 26; n=48, 50, 53, 45 | 344.1 (606.10) | 267.7 (516.53) | 242.5 (275.72) | 163.5 (156.79)
  CK; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  CK; Week 28; n=51, 52, 52, 45 | 213.4 (182.12) | 276.8 (581.44) | 290.4 (457.59) | 154.7 (168.77)
  CK; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  CK; Week 32; n=52, 53, 55, 45 | 205.6 (171.74) | 248.8 (525.79) | 311.3 (437.31) | 254.7 (778.33)
  CK; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  CK; Week 36; n=52, 52, 55, 45 | 528.4 (1984.77) | 242.9 (353.65) | 255.2 (275.74) | 303.1 (615.91)
  CK; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  CK; Week 40; n=52, 53, 55, 44 | 259.5 (381.33) | 225.4 (342.50) | 292.6 (360.32) | 150.2 (96.11)
  CK; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  CK; Week 48; n=51, 53, 54, 44 | 203.5 (136.48) | 219.3 (527.75) | 219.8 (195.62) | 146.3 (88.07)
  CK; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  CK; Week 60; n=48, 47, 53, 44 | 315.7 (730.27) | 215.5 (340.37) | 399.6 (923.74) | 168.0 (154.36)
  CK; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  CK; Week 72; n=47, 47, 52, 42 | 182.5 (148.31) | 354.0 (911.76) | 247.7 (348.72) | 120.5 (59.89)
  CK; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  CK; Week 84; n=46, 48, 52, 42 | 204.3 (160.30) | 329.2 (724.97) | 195.0 (164.14) | 258.6 (650.38)
  CK; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  CK; Week 96; n=45, 48, 52, 40 | 542.7 (2451.57) | 272.8 (589.15) | 199.7 (194.46) | 281.1 (903.71)

23. Secondary Outcome: Absolute Values for Creatinine and Total Bilirubin During Double-blind Randomized Treatment Until Week 96
Description: Blood samples were collected for the analysis of creatinine and total bilirubin (T. bilirubin). Baseline value is the last pre-treatment value observed.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Micromoles per liter
  Creatinine; Baseline; n=60, 60, 61, 62 | 80.4 (13.69) | 80.5 (13.55) | 79.9 (14.11) | 83.1 (13.41)
  Creatinine; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  Creatinine; Week 2; n=58, 56, 58, 58 | 83.8 (14.33) | 83.3 (14.10) | 84.6 (15.27) | 83.8 (15.29)
  Creatinine; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Creatinine; Week 4; n=58, 57, 59, 57 | 82.9 (15.45) | 83.0 (14.55) | 84.2 (14.28) | 83.1 (14.22)
  Creatinine; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  Creatinine; Week 8; n=58, 55, 57, 54 | 82.9 (13.79) | 82.2 (13.03) | 83.5 (14.41) | 82.4 (13.94)
  Creatinine; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Creatinine; Week 12; n=58, 53, 57, 51 | 83.8 (13.33) | 82.7 (14.96) | 84.1 (14.64) | 81.1 (12.83)
  Creatinine; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Creatinine; Week 16; n=57, 54, 57, 52 | 83.4 (17.07) | 82.3 (14.56) | 82.4 (14.16) | 79.6 (11.83)
  Creatinine; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  Creatinine; Week 20; n=56, 54, 55, 49 | 83.2 (12.95) | 82.0 (14.42) | 86.1 (14.34) | 79.5 (11.72)
  Creatinine; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Creatinine; Week 24; n=56, 53, 56, 47 | 83.2 (13.07) | 83.3 (15.56) | 85.2 (13.93) | 80.0 (20.74)
  Creatinine; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Creatinine; Week 26; n=48, 50, 53, 45 | 83.4 (13.45) | 82.6 (14.15) | 87.0 (13.82) | 78.6 (9.61)
  Creatinine; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  Creatinine; Week 28; n=51, 52, 52, 45 | 83.0 (13.32) | 83.8 (14.84) | 85.6 (13.96) | 78.5 (10.34)
  Creatinine; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Creatinine; Week 32; n=52, 53, 55, 45 | 83.8 (14.11) | 82.6 (13.48) | 85.7 (14.34) | 78.1 (9.90)
  Creatinine; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  Creatinine; Week 36; n=52, 52, 55, 45 | 83.5 (12.68) | 84.6 (13.22) | 86.7 (16.21) | 78.4 (10.87)
  Creatinine; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  Creatinine; Week 40; n=52, 53, 55, 44 | 83.3 (12.60) | 83.2 (13.04) | 85.4 (14.38) | 79.2 (15.99)
  Creatinine; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Creatinine; Week 48; n=51, 53, 54, 44 | 83.4 (13.48) | 83.1 (14.55) | 85.0 (14.54) | 79.0 (12.52)
  Creatinine; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  Creatinine; Week 60; n=48, 47, 53, 44 | 83.9 (13.85) | 83.0 (14.31) | 85.2 (14.57) | 77.9 (11.13)
  Creatinine; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  Creatinine; Week 72; n=47, 47, 52, 42 | 84.5 (12.46) | 86.1 (14.95) | 87.3 (14.95) | 77.7 (11.44)
  Creatinine; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Creatinine; Week 84; n=46, 48, 52, 42 | 85.0 (15.06) | 84.8 (17.41) | 87.3 (13.15) | 79.7 (11.20)
  Creatinine; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Creatinine; Week 96; n=45, 48, 52, 40 | 82.0 (11.46) | 86.4 (17.24) | 88.5 (14.75) | 81.0 (10.10)
  T. Bilirubin; Baseline; n=60, 60, 61, 62 | 9.2 (4.65) | 9.4 (4.59) | 10.5 (5.48) | 9.7 (4.42)
  T. Bilirubin; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  T. Bilirubin; Week 2; n=58, 56, 58, 58 | 9.2 (4.48) | 9.1 (4.50) | 10.0 (5.92) | 6.8 (1.71)
  T. Bilirubin; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  T. Bilirubin; Week 4; n=58, 57, 59, 57 | 9.4 (4.40) | 9.3 (4.47) | 9.8 (6.05) | 6.4 (1.61)
  T. Bilirubin; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  T. Bilirubin; Week 8; n=58, 55, 57, 54 | 9.3 (4.50) | 9.0 (3.33) | 10.1 (5.55) | 6.3 (1.46)
  T. Bilirubin; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  T. Bilirubin; Week 12; n=58, 53, 57, 51 | 9.5 (5.16) | 8.9 (3.79) | 10.2 (5.47) | 7.0 (2.57)
  T. Bilirubin; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  T. Bilirubin; Week 16; n=57, 54, 57, 52 | 9.6 (5.04) | 8.5 (3.90) | 10.4 (4.88) | 7.0 (2.61)
  T. Bilirubin; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  T. Bilirubin; Week 20; n=56, 54, 55, 49 | 9.0 (4.09) | 9.0 (4.91) | 10.4 (5.49) | 6.8 (1.67)
  T. Bilirubin; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  T. Bilirubin; Week 24; n=56, 53, 56, 47 | 9.6 (5.18) | 9.8 (5.09) | 10.0 (4.52) | 6.6 (1.60)
  T. Bilirubin; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  T. Bilirubin; Week 26; n=48, 50, 53, 45 | 10.6 (4.97) | 9.9 (5.83) | 12.0 (5.11) | 6.8 (2.19)
  T. Bilirubin; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  T. Bilirubin; Week 28; n=51, 52, 52, 45 | 10.3 (4.87) | 10.2 (5.90) | 11.4 (4.77) | 6.4 (1.51)
  T. Bilirubin; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  T. Bilirubin; Week 32; n=52, 53, 55, 45 | 9.8 (4.91) | 9.8 (4.80) | 11.7 (6.70) | 6.6 (1.74)
  T. Bilirubin; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  T. Bilirubin; Week 36; n=52, 52, 55, 45 | 10.3 (5.25) | 10.1 (5.47) | 12.2 (6.08) | 6.5 (1.71)
  T. Bilirubin; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  T. Bilirubin; Week 40; n=52, 53, 55, 44 | 10.8 (5.81) | 11.2 (7.04) | 12.3 (6.67) | 6.3 (1.53)
  T. Bilirubin; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  T. Bilirubin; Week 48; n=51, 53, 54, 44 | 10.0 (4.96) | 9.6 (3.86) | 10.4 (4.91) | 6.6 (1.65)
  T. Bilirubin; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  T. Bilirubin; Week 60; n=48, 47, 53, 44 | 11.2 (4.28) | 9.8 (3.75) | 11.6 (6.28) | 7.0 (2.13)
  T. Bilirubin; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  T. Bilirubin; Week 72; n=47, 47, 52, 42 | 10.8 (6.63) | 10.0 (4.89) | 11.4 (5.87) | 6.5 (1.40)
  T. Bilirubin; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  T. Bilirubin; Week 84; n=46, 48, 52, 42 | 11.7 (6.77) | 9.9 (4.35) | 12.0 (5.64) | 6.6 (2.27)
  T. Bilirubin; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  T. Bilirubin; Week 96; n=45, 48, 52, 40 | 10.3 (5.29) | 9.9 (4.58) | 12.5 (5.61) | 6.8 (1.80)

24. Secondary Outcome: Absolute Values for Estimated Creatinine Clearance During Double-blind Randomized Treatment Until Week 96
Description: Blood samples were collected for the analysis of estimated creatinine clearance. Estimated creatinine clearance was calculated using Cockcroft-Gault formula. Baseline value is the last pre-treatment value observed.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 16, 20, 24, 26, 40, 48, 60 and 96
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Milliliters per minute
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Milliliters per minute
  Baseline; n=60, 60, 61, 62 | 131.0 (28.18) | 135.2 (41.33) | 128.3 (33.51) | 125.6 (35.30)
  Week 2; n=1, 1, 0, 3: number analyzed (Participants) | 1 | 1 | 0 | 3
  Week 2; n=1, 1, 0, 3 | 96.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | 106.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  | 99.0 (31.00)
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | 129.3 (31.29) | 132.5 (42.28) | 122.4 (33.00) | 127.0 (35.64)
  Week 8; n=2, 1, 1, 1: number analyzed (Participants) | 2 | 1 | 1 | 1
  Week 8; n=2, 1, 1, 1 | 125.0 (35.36) | 124.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | 143.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | 101.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  Week 16; n=55, 53, 56, 49: number analyzed (Participants) | 55 | 53 | 56 | 49
  Week 16; n=55, 53, 56, 49 | 132.4 (50.97) | 139.4 (42.30) | 123.9 (31.85) | 132.3 (39.97)
  Week 20; n=2, 0, 0, 1: number analyzed (Participants) | 2 | 0 | 0 | 1
  Week 20; n=2, 0, 0, 1 | 137.0 (11.31) |  |  | 122.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  Week 24; n=52, 53, 55, 46: number analyzed (Participants) | 52 | 53 | 55 | 46
  Week 24; n=52, 53, 55, 46 | 127.9 (30.90) | 132.8 (39.93) | 120.7 (27.41) | 135.1 (38.98)
  Week 26; n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 26; n=0, 1, 0, 0 |  | 147.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |
  Week 40; n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 40; n=0, 1, 0, 0 |  | 180.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |
  Week 48; n=51, 50, 54, 44: number analyzed (Participants) | 51 | 50 | 54 | 44
  Week 48; n=51, 50, 54, 44 | 127.0 (30.01) | 139.2 (42.07) | 122.3 (29.21) | 131.0 (44.41)
  Week 60; n=0, 0, 0, 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 60; n=0, 0, 0, 1 |  |  |  | 144.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Week 96; n=45, 48, 52, 40 | 130.8 (40.80) | 137.7 (45.07) | 116.6 (27.05) | 134.8 (43.35)

25. Secondary Outcome: Absolute Values for Hemoglobin During Double-blind Randomized Treatment Until Week 96
Description: Blood samples were collected for the analysis of hemoglobin level. Baseline value is the last pre-treatment value observed.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Grams per liter
  Baseline; n=60, 60, 61, 62 | 141.9 (12.46) | 143.2 (10.66) | 146.6 (13.41) | 145.4 (12.39)
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 142.0 (13.84) | 142.8 (11.68) | 145.9 (12.05) | 146.4 (13.49)
  Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  Week 4; n=57, 57, 59, 57 | 141.9 (13.39) | 143.5 (11.69) | 147.3 (12.13) | 146.6 (13.06)
  Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  Week 8; n=58, 56, 56, 55 | 144.9 (13.10) | 147.7 (11.88) | 148.6 (12.10) | 148.1 (12.32)
  Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Week 12; n=58, 53, 57, 51 | 144.3 (12.19) | 147.4 (10.60) | 149.1 (11.25) | 149.2 (13.14)
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 143.5 (11.77) | 146.5 (10.71) | 148.7 (11.08) | 147.6 (12.05)
  Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  Week 20; n=56, 54, 55, 49 | 144.3 (13.33) | 146.9 (11.23) | 149.8 (11.11) | 147.2 (12.18)
  Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Week 24; n=56, 53, 56, 47 | 144.8 (12.66) | 147.8 (10.69) | 150.4 (11.65) | 148.5 (11.31)
  Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Week 26; n=48, 50, 53, 45 | 144.4 (13.30) | 145.8 (11.63) | 149.8 (11.47) | 148.2 (12.32)
  Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  Week 28; n=50, 52, 52, 45 | 143.7 (13.20) | 146.8 (10.89) | 149.3 (10.15) | 145.9 (13.17)
  Week 32; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  Week 32; n=51, 53, 55, 45 | 144.6 (9.53) | 146.1 (10.44) | 150.5 (11.19) | 145.9 (11.41)
  Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  Week 36; n=52, 53, 55, 44 | 142.3 (11.07) | 145.9 (11.24) | 149.8 (11.26) | 145.0 (10.73)
  Week 40; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  Week 40; n=51, 53, 55, 45 | 142.2 (11.06) | 145.2 (11.03) | 149.2 (11.71) | 145.1 (9.98)
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 142.9 (9.15) | 145.7 (10.59) | 146.5 (12.48) | 145.4 (12.24)
  Week 60; n=48, 47, 52, 44: number analyzed (Participants) | 48 | 47 | 52 | 44
  Week 60; n=48, 47, 52, 44 | 144.5 (9.91) | 148.3 (10.96) | 149.8 (10.82) | 147.6 (12.73)
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 143.9 (10.24) | 148.1 (10.15) | 149.6 (11.46) | 147.7 (11.22)
  Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  Week 84; n=46, 48, 51, 42 | 145.6 (11.00) | 147.7 (10.04) | 150.3 (10.38) | 147.0 (11.77)
  Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  Week 96; n=46, 46, 52, 41 | 144.9 (12.41) | 147.1 (11.06) | 150.8 (10.37) | 147.0 (11.03)

26. Secondary Outcome: Absolute Values for Platelet Count, Total Neutrophils and WBC Count During Double-blind Randomized Treatment Until Week 96
Description: Blood samples were collected for the analysis of platelet count, total neutrophils (T. neutrophils) and WBC count. Baseline value is the last pre-treatment value observed.
Time Frame: Baseline (Day 1), Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 48, 60, 72, 84 and 96
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Giga cells per liter
  T. neutrophils; Baseline; n=60, 60, 61, 62 | 2.643 (1.1237) | 2.891 (1.4383) | 2.487 (1.0240) | 2.441 (1.1548)
  T. neutrophils; Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  T. neutrophils; Week 2; n=57, 56, 59, 59 | 2.723 (1.1402) | 2.776 (1.0729) | 2.598 (1.1295) | 3.207 (1.6307)
  T. neutrophils; Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  T. neutrophils; Week 4; n=57, 57, 59, 57 | 2.685 (1.2477) | 2.771 (1.2587) | 2.649 (1.0692) | 2.848 (1.8642)
  T. neutrophils; Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  T. neutrophils; Week 8; n=58, 56, 56, 55 | 2.899 (1.2111) | 2.802 (1.1296) | 2.738 (1.1533) | 2.746 (0.9969)
  T. neutrophils; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  T. neutrophils; Week 12; n=58, 53, 57, 51 | 2.812 (1.1377) | 2.933 (1.5977) | 2.822 (1.3294) | 2.979 (1.7673)
  T. neutrophils; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  T. neutrophils; Week 16; n=57, 54, 57, 52 | 3.078 (1.5948) | 2.716 (1.1022) | 2.665 (1.0287) | 2.858 (1.1909)
  T. neutrophils; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  T. neutrophils; Week 20; n=56, 54, 55, 49 | 2.958 (1.2918) | 2.904 (1.1794) | 2.989 (1.6589) | 3.187 (1.6424)
  T. neutrophils; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  T. neutrophils; Week 24; n=56, 53, 56, 47 | 3.151 (1.2378) | 2.996 (1.5425) | 2.884 (1.0047) | 3.142 (1.6483)
  T. neutrophils; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  T. neutrophils; Week 26; n=48, 50, 53, 45 | 2.885 (1.0874) | 2.958 (1.2097) | 2.830 (1.0354) | 2.886 (1.3159)
  T. neutrophils; Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  T. neutrophils; Week 28; n=50, 52, 52, 45 | 3.183 (1.0674) | 3.005 (1.0029) | 2.989 (1.4078) | 2.916 (1.0731)
  T. neutrophils; Week 32; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  T. neutrophils; Week 32; n=51, 53, 55, 45 | 2.797 (0.9490) | 3.036 (1.1931) | 3.167 (1.3992) | 3.174 (1.7150)
  T. neutrophils; Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  T. neutrophils; Week 36; n=52, 53, 55, 44 | 3.162 (1.1538) | 2.916 (1.2331) | 3.010 (1.0698) | 2.914 (1.2530)
  T. neutrophils; Week 40; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  T. neutrophils; Week 40; n=51, 53, 55, 45 | 3.155 (1.3417) | 3.065 (1.2945) | 3.050 (1.0745) | 3.187 (1.6006)
  T. neutrophils; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  T. neutrophils; Week 48; n=51, 53, 54, 44 | 3.138 (1.3751) | 3.132 (1.1976) | 3.004 (1.1720) | 3.134 (1.6646)
  T. neutrophils; Week 60; n=48, 47, 52, 44: number analyzed (Participants) | 48 | 47 | 52 | 44
  T. neutrophils; Week 60; n=48, 47, 52, 44 | 3.164 (1.3804) | 3.333 (1.5642) | 3.200 (1.2159) | 3.269 (1.3866)
  T. neutrophils; Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  T. neutrophils; Week 72; n=47, 48, 52, 42 | 3.197 (1.2931) | 3.131 (1.2337) | 3.163 (1.0874) | 3.361 (1.8047)
  T. neutrophils; Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  T. neutrophils; Week 84; n=46, 48, 51, 42 | 3.245 (1.4593) | 3.385 (1.3591) | 3.512 (1.3176) | 3.259 (1.6532)
  T. neutrophils; Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  T. neutrophils; Week 96; n=46, 46, 52, 41 | 3.466 (1.1229) | 3.540 (1.7870) | 3.494 (1.2790) | 3.297 (1.4509)
  Platelet count; Baseline; n=60, 60, 61, 62 | 212.5 (53.22) | 202.3 (51.74) | 190.0 (55.71) | 200.1 (52.36)
  Platelet count; Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Platelet count; Week 2; n=57, 56, 59, 59 | 225.0 (54.84) | 222.0 (48.82) | 204.8 (50.51) | 216.2 (52.60)
  Platelet count; Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  Platelet count; Week 4; n=57, 57, 59, 57 | 225.2 (52.94) | 222.4 (52.61) | 204.6 (57.51) | 216.0 (55.41)
  Platelet count; Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  Platelet count; Week 8; n=58, 56, 56, 55 | 224.5 (50.94) | 228.4 (57.01) | 211.5 (56.80) | 209.8 (48.62)
  Platelet count; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Platelet count; Week 12; n=58, 53, 57, 51 | 227.2 (49.64) | 216.4 (52.46) | 209.2 (51.62) | 213.7 (50.65)
  Platelet count; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Platelet count; Week 16; n=57, 54, 57, 52 | 230.0 (59.33) | 212.4 (54.22) | 209.5 (50.32) | 211.4 (50.56)
  Platelet count; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  Platelet count; Week 20; n=56, 54, 55, 49 | 231.3 (55.14) | 215.5 (47.03) | 205.4 (48.40) | 214.9 (51.41)
  Platelet count; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Platelet count; Week 24; n=56, 53, 56, 47 | 226.1 (52.17) | 219.7 (50.75) | 210.9 (56.34) | 220.9 (67.67)
  Platelet count; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Platelet count; Week 26; n=48, 50, 53, 45 | 224.9 (56.06) | 215.5 (53.10) | 199.4 (60.65) | 214.4 (53.90)
  Platelet count; Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  Platelet count; Week 28; n=50, 52, 52, 45 | 223.3 (50.28) | 217.0 (56.54) | 209.8 (56.65) | 215.4 (57.81)
  Platelet count; Week 32; n=51, 52, 55, 45: number analyzed (Participants) | 51 | 52 | 55 | 45
  Platelet count; Week 32; n=51, 52, 55, 45 | 220.5 (55.37) | 214.0 (46.66) | 207.8 (53.33) | 212.6 (52.27)
  Platelet count; Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  Platelet count; Week 36; n=52, 53, 55, 44 | 220.0 (47.58) | 212.1 (51.61) | 204.2 (54.34) | 209.8 (52.54)
  Platelet count; Week 40; n=51, 53, 54, 45: number analyzed (Participants) | 51 | 53 | 54 | 45
  Platelet count; Week 40; n=51, 53, 54, 45 | 224.9 (52.93) | 210.1 (55.87) | 199.3 (52.37) | 217.7 (54.40)
  Platelet count; Week 48; n=51, 52, 53, 44: number analyzed (Participants) | 51 | 52 | 53 | 44
  Platelet count; Week 48; n=51, 52, 53, 44 | 225.6 (60.05) | 221.2 (56.12) | 209.9 (56.81) | 220.3 (52.52)
  Platelet count; Week 60; n=48, 47, 51, 44: number analyzed (Participants) | 48 | 47 | 51 | 44
  Platelet count; Week 60; n=48, 47, 51, 44 | 232.5 (57.00) | 219.8 (55.01) | 212.2 (53.68) | 230.5 (56.39)
  Platelet count; Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Platelet count; Week 72; n=47, 48, 52, 42 | 234.0 (52.53) | 224.4 (50.06) | 212.2 (52.59) | 225.9 (52.62)
  Platelet count; Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  Platelet count; Week 84; n=46, 48, 51, 42 | 224.8 (52.36) | 218.8 (49.15) | 210.1 (51.72) | 216.5 (53.09)
  Platelet count; Week 96; n=46, 45, 51, 41: number analyzed (Participants) | 46 | 45 | 51 | 41
  Platelet count; Week 96; n=46, 45, 51, 41 | 237.1 (58.94) | 221.8 (57.95) | 210.6 (57.34) | 214.0 (51.10)
  WBC count; Baseline; n=60, 60, 61, 62 | 5.06 (1.552) | 5.19 (1.632) | 4.72 (1.332) | 4.70 (1.388)
  WBC count; Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  WBC count; Week 2; n=57, 56, 59, 59 | 5.32 (1.602) | 5.30 (1.448) | 5.02 (1.355) | 5.45 (1.856)
  WBC count; Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  WBC count; Week 4; n=57, 57, 59, 57 | 5.24 (1.802) | 5.17 (1.604) | 5.02 (1.342) | 5.02 (1.993)
  WBC count; Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  WBC count; Week 8; n=58, 56, 56, 55 | 5.44 (1.751) | 5.30 (1.556) | 5.04 (1.230) | 5.02 (1.195)
  WBC count; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  WBC count; Week 12; n=58, 53, 57, 51 | 5.41 (1.560) | 5.50 (1.794) | 5.34 (1.524) | 5.27 (1.899)
  WBC count; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  WBC count; Week 16; n=57, 54, 57, 52 | 5.56 (1.895) | 5.20 (1.337) | 4.97 (1.108) | 5.13 (1.480)
  WBC count; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  WBC count; Week 20; n=56, 54, 55, 49 | 5.46 (1.486) | 5.41 (1.354) | 5.39 (1.877) | 5.50 (1.763)
  WBC count; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  WBC count; Week 24; n=56, 53, 56, 47 | 5.57 (1.558) | 5.53 (1.993) | 5.28 (1.367) | 5.34 (1.854)
  WBC count; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  WBC count; Week 26; n=48, 50, 53, 45 | 5.30 (1.294) | 5.50 (1.642) | 5.29 (1.315) | 5.08 (1.381)
  WBC count; Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  WBC count; Week 28; n=50, 52, 52, 45 | 5.71 (1.426) | 5.53 (1.493) | 5.38 (1.542) | 5.14 (1.254)
  WBC count; Week 32; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  WBC count; Week 32; n=51, 53, 55, 45 | 5.30 (1.399) | 5.63 (1.456) | 5.57 (1.720) | 5.48 (1.939)
  WBC count; Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  WBC count; Week 36; n=52, 53, 55, 44 | 5.64 (1.461) | 5.48 (1.756) | 5.56 (1.303) | 5.17 (1.312)
  WBC count; Week 40; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  WBC count; Week 40; n=51, 53, 55, 45 | 5.63 (1.607) | 5.61 (1.687) | 5.45 (1.255) | 5.51 (1.808)
  WBC count; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  WBC count; Week 48; n=51, 53, 54, 44 | 5.51 (1.663) | 5.72 (1.695) | 5.41 (1.314) | 5.53 (1.818)
  WBC count; Week 60; n=48, 47, 52, 44: number analyzed (Participants) | 48 | 47 | 52 | 44
  WBC count; Week 60; n=48, 47, 52, 44 | 5.73 (1.749) | 5.93 (1.677) | 5.63 (1.491) | 5.75 (1.608)
  WBC count; Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  WBC count; Week 72; n=47, 48, 52, 42 | 5.80 (1.671) | 5.71 (1.550) | 5.73 (1.297) | 5.84 (2.104)
  WBC count; Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  WBC count; Week 84; n=46, 48, 51, 42 | 5.91 (1.845) | 6.11 (1.718) | 6.05 (1.469) | 5.78 (1.658)
  WBC count; Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  WBC count; Week 96; n=46, 46, 52, 41 | 6.14 (1.622) | 6.15 (1.933) | 6.01 (1.489) | 5.75 (1.556)

27. Secondary Outcome: Change From Baseline in ALT, AST and CK Over Time by Visit
Description: Blood samples were collected for the analysis of ALT, AST and CK. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: as for outcome 7
Population: Safety Population. Participants randomized to Efavirenz 600 mg arm were considered to have completed their participation in the study after Week 96; hence were no longer followed as part of this study. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Mean (Standard Deviation); unit: International Units per Liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
International Units per Liter
  ALT; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  ALT; Week 2; n=58, 56, 58, 58 | 0.1 (7.47) | -2.1 (12.74) | -1.5 (14.75) | -1.3 (23.63)
  ALT; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  ALT; Week 4; n=58, 57, 59, 57 | -0.7 (8.94) | -2.6 (12.13) | 1.7 (22.01) | 0.1 (29.43)
  ALT; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  ALT; Week 8; n=58, 55, 57, 54 | 2.2 (10.71) | 0.5 (18.49) | 8.0 (56.59) | -6.3 (29.64)
  ALT; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  ALT; Week 12; n=58, 53, 57, 51 | 1.2 (8.91) | 2.7 (24.70) | -0.6 (13.40) | -6.3 (33.57)
  ALT; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  ALT; Week 16; n=57, 54, 57, 52 | 2.1 (19.92) | 0.1 (27.07) | -0.3 (13.36) | -1.6 (38.90)
  ALT; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  ALT; Week 20; n=56, 54, 55, 49 | -0.7 (8.58) | -3.6 (14.07) | 3.0 (18.56) | -4.8 (34.09)
  ALT; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  ALT; Week 24; n=56, 53, 56, 47 | -2.1 (7.93) | -1.2 (20.79) | 1.4 (19.49) | -6.0 (33.13)
  ALT; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  ALT; Week 26; n=48, 50, 53, 45 | 1.1 (16.32) | -2.6 (24.31) | -1.7 (13.07) | -3.7 (41.02)
  ALT; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  ALT; Week 28; n=51, 52, 52, 45 | -2.3 (7.87) | -2.3 (25.40) | -2.9 (17.79) | -8.1 (33.92)
  ALT; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  ALT; Week 32; n=52, 53, 55, 45 | -3.1 (8.55) | -1.7 (25.75) | -4.0 (13.90) | -8.6 (34.85)
  ALT; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  ALT; Week 36; n=52, 52, 55, 45 | 0.8 (23.68) | -4.2 (17.84) | -3.0 (15.31) | -8.2 (32.34)
  ALT; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  ALT; Week 40; n=52, 53, 55, 44 | 0.1 (15.48) | -4.1 (15.85) | -1.4 (15.96) | -8.0 (32.36)
  ALT; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  ALT; Week 48; n=51, 53, 54, 44 | -4.1 (9.03) | -3.8 (17.77) | -2.4 (14.60) | -8.6 (34.80)
  ALT; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  ALT; Week 60; n=48, 47, 53, 44 | -1.0 (15.72) | -2.6 (17.74) | 0.5 (18.13) | -6.3 (36.82)
  ALT; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  ALT; Week 72; n=47, 47, 52, 42 | -2.8 (9.92) | 2.7 (30.95) | -0.9 (15.27) | -8.5 (36.32)
  ALT; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  ALT; Week 84; n=46, 48, 52, 42 | -2.4 (10.87) | 1.9 (22.60) | -2.0 (16.90) | -4.0 (49.06)
  ALT; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  ALT; Week 96; n=45, 48, 52, 40 | -0.4 (18.47) | 20.6 (154.71) | -1.7 (17.12) | -7.6 (20.22)
  ALT; Week 108; n=43, 46, 48, 0: number analyzed (Participants) | 43 | 46 | 48 | 0
  ALT; Week 108; n=43, 46, 48, 0 | 0.5 (11.41) | -2.7 (20.04) | -0.7 (20.63) |
  ALT; Week 120; n=40, 45, 48, 0: number analyzed (Participants) | 40 | 45 | 48 | 0
  ALT; Week 120; n=40, 45, 48, 0 | 4.4 (23.14) | -2.6 (18.42) | -3.7 (15.82) |
  ALT; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  ALT; Week 132; n=40, 46, 49, 0 | 4.3 (23.58) | -3.0 (20.18) | -3.8 (17.80) |
  ALT; Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  ALT; Week 144; n=37, 45, 47, 0 | 0.1 (13.01) | -3.4 (17.81) | -1.8 (15.40) |
  ALT; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  ALT; Week 156; n=37, 42, 49, 0 | -0.5 (13.86) | -1.8 (19.51) | -2.2 (27.94) |
  ALT; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  ALT; Week 168; n=35, 43, 47, 0 | 2.3 (11.40) | -1.1 (19.14) | -3.6 (24.29) |
  ALT; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  ALT; Week 180; n=36, 41, 47, 0 | 1.7 (12.96) | -2.8 (15.68) | -1.2 (31.69) |
  ALT; Week 192; n=36, 39, 47, 0: number analyzed (Participants) | 36 | 39 | 47 | 0
  ALT; Week 192; n=36, 39, 47, 0 | 4.9 (17.56) | -3.3 (16.07) | 1.3 (35.53) |
  ALT; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  ALT; Week 204; n=34, 39, 47, 0 | 1.9 (11.42) | -1.7 (16.25) | -3.4 (24.00) |
  ALT; Week 216; n=33, 39, 46, 0: number analyzed (Participants) | 33 | 39 | 46 | 0
  ALT; Week 216; n=33, 39, 46, 0 | 1.7 (11.28) | -3.0 (13.37) | -2.7 (26.90) |
  ALT; Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  ALT; Week 228; n=32, 39, 47, 0 | 36.8 (162.51) | -1.1 (13.68) | 0.5 (17.72) |
  ALT; Week 240; n=30, 39, 46, 0: number analyzed (Participants) | 30 | 39 | 46 | 0
  ALT; Week 240; n=30, 39, 46, 0 | 5.3 (38.37) | -0.1 (16.56) | -0.7 (18.20) |
  ALT; Week 252; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  ALT; Week 252; n=31, 38, 46, 0 | 2.0 (18.06) | 2.8 (22.54) | -1.6 (20.95) |
  ALT; Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  ALT; Week 264; n=32, 38, 47, 0 | 3.3 (19.88) | 0.7 (23.29) | 2.0 (29.60) |
  ALT; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  ALT; Week 276; n=31, 38, 45, 0 | 3.3 (19.97) | 2.9 (31.30) | 1.1 (23.92) |
  ALT; Week 288; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  ALT; Week 288; n=31, 38, 45, 0 | 6.6 (24.89) | 1.2 (27.16) | 1.9 (26.19) |
  ALT; Week 300; n=30, 37, 44, 0: number analyzed (Participants) | 30 | 37 | 44 | 0
  ALT; Week 300; n=30, 37, 44, 0 | 4.8 (25.46) | -1.4 (19.21) | -1.8 (24.06) |
  ALT; Week 312; n=31, 34, 43, 0: number analyzed (Participants) | 31 | 34 | 43 | 0
  ALT; Week 312; n=31, 34, 43, 0 | 5.5 (25.29) | 7.6 (42.61) | 0.0 (22.51) |
  ALT; Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  ALT; Week 324; n=3, 4, 3, 0 | 17.7 (40.15) | 1.3 (8.73) | 1.0 (4.36) |
  AST; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  AST; Week 2; n=58, 56, 58, 58 | 0.7 (6.11) | -1.3 (11.20) | -1.6 (8.85) | 0.9 (58.63)
  AST; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  AST; Week 4; n=58, 57, 59, 57 | -1.0 (5.96) | -2.8 (8.97) | 0.1 (14.56) | -2.9 (31.52)
  AST; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  AST; Week 8; n=58, 55, 57, 54 | 4.2 (30.51) | 1.5 (22.15) | 5.3 (36.86) | -7.3 (29.65)
  AST; Week 12; n=58, 53, 57, 50: number analyzed (Participants) | 58 | 53 | 57 | 50
  AST; Week 12; n=58, 53, 57, 50 | 1.3 (10.43) | 1.6 (21.65) | -1.7 (8.91) | -7.9 (32.18)
  AST; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  AST; Week 16; n=57, 54, 57, 52 | -0.7 (10.43) | 1.9 (23.46) | -0.6 (8.03) | 4.4 (79.53)
  AST; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  AST; Week 20; n=56, 54, 55, 49 | 1.3 (18.94) | -3.1 (10.44) | 4.6 (23.87) | -3.6 (41.56)
  AST; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  AST; Week 24; n=56, 53, 56, 47 | -1.4 (7.81) | -0.3 (15.64) | 1.5 (15.03) | -2.1 (13.59)
  AST; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  AST; Week 26; n=48, 50, 53, 45 | 3.3 (28.47) | -0.9 (16.10) | -1.7 (8.21) | -2.6 (17.81)
  AST; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  AST; Week 28; n=51, 52, 52, 45 | -2.0 (6.39) | -0.2 (15.51) | -1.9 (13.67) | -5.1 (15.42)
  AST; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  AST; Week 32; n=52, 53, 55, 45 | -2.7 (5.77) | -1.0 (16.15) | -1.4 (9.19) | -2.8 (17.86)
  AST; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  AST; Week 36; n=52, 52, 55, 45 | 4.6 (38.77) | -2.1 (12.13) | -0.6 (11.86) | -1.9 (17.93)
  AST; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  AST; Week 40; n=52, 53, 55, 44 | 0.1 (13.12) | -2.9 (10.87) | -0.5 (14.40) | -5.1 (14.94)
  AST; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  AST; Week 48; n=51, 53, 54, 44 | -3.3 (7.99) | -3.2 (12.28) | -3.0 (8.28) | -4.4 (16.67)
  AST; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  AST; Week 60; n=48, 47, 53, 44 | -0.9 (9.05) | -2.0 (13.06) | 3.0 (18.70) | -3.2 (17.49)
  AST; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  AST; Week 72; n=47, 47, 52, 42 | -2.7 (6.70) | 3.7 (24.41) | -0.5 (9.75) | -4.6 (15.69)
  AST; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  AST; Week 84; n=46, 48, 52, 42 | -2.2 (7.56) | 2.0 (19.02) | -1.8 (9.46) | 2.3 (40.93)
  AST; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  AST; Week 96; n=45, 48, 52, 40 | -0.8 (22.39) | 20.5 (150.10) | -1.0 (12.58) | -0.3 (25.99)
  AST; Week 108; n=43, 46, 48, 0: number analyzed (Participants) | 43 | 46 | 48 | 0
  AST; Week 108; n=43, 46, 48, 0 | -1.0 (10.89) | -4.0 (11.71) | 0.6 (22.77) |
  AST; Week 120; n=40, 45, 48, 0: number analyzed (Participants) | 40 | 45 | 48 | 0
  AST; Week 120; n=40, 45, 48, 0 | 0.1 (13.16) | -2.5 (13.44) | -2.4 (10.90) |
  AST; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  AST; Week 132; n=40, 46, 49, 0 | -0.2 (11.50) | -3.9 (12.40) | 0.7 (32.61) |
  AST; Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  AST; Week 144; n=37, 45, 47, 0 | -3.4 (8.19) | -4.3 (13.76) | -3.9 (9.45) |
  AST; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  AST; Week 156; n=37, 42, 49, 0 | -3.0 (8.78) | -3.2 (13.94) | -4.1 (13.08) |
  AST; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  AST; Week 168; n=35, 43, 47, 0 | -0.8 (8.95) | -3.4 (12.15) | -3.8 (13.44) |
  AST; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  AST; Week 180; n=36, 41, 47, 0 | -1.9 (7.91) | -4.2 (12.71) | -2.9 (17.09) |
  AST; Week 192; n=36, 39, 47, 0: number analyzed (Participants) | 36 | 39 | 47 | 0
  AST; Week 192; n=36, 39, 47, 0 | -1.5 (8.89) | -5.3 (11.00) | 0.1 (20.52) |
  AST; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  AST; Week 204; n=34, 39, 47, 0 | -1.7 (7.88) | -4.8 (10.98) | -4.5 (12.04) |
  AST; Week 216; n=33, 39, 46, 0: number analyzed (Participants) | 33 | 39 | 46 | 0
  AST; Week 216; n=33, 39, 46, 0 | -2.7 (6.40) | -4.9 (11.54) | -4.3 (13.42) |
  AST; Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  AST; Week 228; n=32, 39, 47, 0 | 13.5 (72.97) | -5.9 (11.78) | -2.8 (10.14) |
  AST; Week 240; n=30, 39, 46, 0: number analyzed (Participants) | 30 | 39 | 46 | 0
  AST; Week 240; n=30, 39, 46, 0 | -1.0 (21.51) | -5.3 (11.70) | -3.4 (11.32) |
  AST; Week 252; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  AST; Week 252; n=31, 38, 46, 0 | -2.2 (10.89) | -2.1 (15.31) | -3.9 (11.09) |
  AST; Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  AST; Week 264; n=32, 38, 47, 0 | -1.6 (10.61) | -4.3 (15.09) | -2.9 (12.87) |
  AST; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  AST; Week 276; n=31, 38, 45, 0 | -1.5 (10.00) | -3.3 (14.38) | -1.4 (12.80) |
  AST; Week 288; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  AST; Week 288; n=31, 38, 45, 0 | -1.4 (11.87) | -3.6 (14.93) | -2.2 (12.98) |
  AST; Week 300; n=30, 37, 44, 0: number analyzed (Participants) | 30 | 37 | 44 | 0
  AST; Week 300; n=30, 37, 44, 0 | -2.0 (9.56) | -5.3 (13.01) | -4.1 (12.07) |
  AST; Week 312; n=31, 34, 43, 0: number analyzed (Participants) | 31 | 34 | 43 | 0
  AST; Week 312; n=31, 34, 43, 0 | 11.7 (82.61) | -2.3 (17.39) | -0.3 (14.27) |
  AST; Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  AST; Week 324; n=3, 4, 3, 0 | 2.7 (12.66) | -5.3 (14.59) | -6.7 (4.16) |
  CK; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  CK; Week 2; n=58, 56, 58, 58 | 40.0 (234.19) | -32.2 (664.29) | 0.4 (183.47) | 159.8 (3217.64)
  CK; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  CK; Week 4; n=58, 57, 59, 57 | -2.3 (125.78) | -82.0 (586.36) | -2.9 (227.73) | -120.3 (1656.37)
  CK; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  CK; Week 8; n=58, 55, 57, 54 | 216.9 (1495.44) | 115.8 (1625.63) | 266.7 (1787.23) | -212.8 (1579.19)
  CK; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  CK; Week 12; n=58, 53, 57, 51 | 120.6 (551.72) | 39.8 (1035.75) | 27.1 (208.15) | -220.1 (1656.33)
  CK; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  CK; Week 16; n=57, 54, 57, 52 | -2.0 (177.01) | 156.3 (1399.82) | 28.6 (218.04) | 269.7 (3855.01)
  CK; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  CK; Week 20; n=56, 54, 55, 49 | 144.2 (969.11) | -68.9 (542.73) | 298.9 (1661.14) | 135.3 (3115.23)
  CK; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  CK; Week 24; n=56, 53, 56, 47 | 27.5 (241.96) | 32.4 (800.50) | 55.9 (252.05) | 103.9 (482.18)
  CK; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  CK; Week 26; n=48, 50, 53, 45 | 133.7 (612.97) | -16.3 (616.41) | 54.4 (316.26) | 21.2 (162.22)
  CK; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  CK; Week 28; n=51, 52, 52, 45 | 9.8 (179.35) | 74.1 (542.07) | 96.8 (475.89) | 4.1 (159.24)
  CK; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  CK; Week 32; n=52, 53, 55, 45 | 3.1 (159.46) | -25.1 (605.67) | 122.1 (364.15) | 110.3 (794.67)
  CK; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  CK; Week 36; n=52, 52, 55, 45 | 325.9 (1995.64) | -33.6 (572.93) | 66.1 (276.38) | 158.7 (625.32)
  CK; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  CK; Week 40; n=52, 53, 55, 44 | 57.1 (350.15) | -48.6 (502.19) | 103.5 (390.10) | 3.8 (128.31)
  CK; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  CK; Week 48; n=51, 53, 54, 44 | -1.3 (173.80) | -54.7 (612.26) | 28.6 (196.37) | 2.8 (124.04)
  CK; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  CK; Week 60; n=48, 47, 53, 44 | 115.4 (743.67) | -80.1 (598.41) | 206.2 (880.62) | 24.5 (158.37)
  CK; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  CK; Week 72; n=47, 47, 52, 42 | -19.8 (152.46) | 53.8 (1031.26) | 67.6 (311.66) | -14.3 (92.49)
  CK; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  CK; Week 84; n=46, 48, 52, 42 | -0.7 (147.67) | 33.6 (900.48) | 14.9 (211.36) | 123.9 (598.22)
  CK; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  CK; Week 96; n=45, 48, 52, 40 | 335.4 (2431.93) | -22.8 (768.54) | 19.6 (249.41) | 143.9 (903.29)
  CK; Week 108; n=43, 46, 48, 0: number analyzed (Participants) | 43 | 46 | 48 | 0
  CK; Week 108; n=43, 46, 48, 0 | 64.2 (339.96) | -88.5 (592.61) | 100.3 (546.46) |
  CK; Week 120; n=40, 45, 48, 0: number analyzed (Participants) | 40 | 45 | 48 | 0
  CK; Week 120; n=40, 45, 48, 0 | 11.5 (229.39) | -48.9 (614.32) | 61.4 (304.98) |
  CK; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  CK; Week 132; n=40, 46, 49, 0 | 30.6 (198.34) | -41.3 (654.65) | 649.6 (3895.73) |
  CK; Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  CK; Week 144; n=37, 45, 47, 0 | 10.6 (143.04) | -72.4 (637.65) | 68.7 (192.20) |
  CK; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  CK; Week 156; n=37, 42, 49, 0 | -5.3 (178.55) | -87.9 (626.53) | 73.3 (396.95) |
  CK; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  CK; Week 168; n=35, 43, 47, 0 | 27.7 (149.18) | -60.7 (648.64) | 74.4 (492.75) |
  CK; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  CK; Week 180; n=36, 41, 47, 0 | 22.4 (120.72) | -16.4 (769.12) | 62.8 (325.34) |
  CK; Week 192; n=36, 39, 47, 0: number analyzed (Participants) | 36 | 39 | 47 | 0
  CK; Week 192; n=36, 39, 47, 0 | 5.2 (123.98) | -98.5 (666.21) | 98.6 (393.41) |
  CK; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  CK; Week 204; n=34, 39, 47, 0 | 79.1 (253.58) | -101.8 (642.05) | 48.3 (148.37) |
  CK; Week 216; n=33, 39, 46, 0: number analyzed (Participants) | 33 | 39 | 46 | 0
  CK; Week 216; n=33, 39, 46, 0 | 43.2 (232.12) | -74.4 (658.64) | 41.9 (177.16) |
  CK; Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  CK; Week 228; n=32, 39, 47, 0 | 64.0 (332.07) | -129.0 (640.89) | 40.4 (133.68) |
  CK; Week 240; n=30, 39, 46, 0: number analyzed (Participants) | 30 | 39 | 46 | 0
  CK; Week 240; n=30, 39, 46, 0 | 1.2 (118.21) | -108.1 (646.43) | 92.0 (285.12) |
  CK; Week 252; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  CK; Week 252; n=31, 38, 46, 0 | 24.6 (96.40) | -110.1 (645.37) | 62.5 (201.59) |
  CK; Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  CK; Week 264; n=32, 38, 47, 0 | 1.9 (135.22) | -31.3 (819.97) | 38.9 (137.90) |
  CK; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  CK; Week 276; n=31, 38, 45, 0 | 39.9 (258.45) | -126.5 (639.63) | 146.4 (350.73) |
  CK; Week 288; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  CK; Week 288; n=31, 38, 45, 0 | 21.6 (139.26) | -98.5 (642.79) | 43.4 (172.08) |
  CK; Week 300; n=30, 37, 44, 0: number analyzed (Participants) | 30 | 37 | 44 | 0
  CK; Week 300; n=30, 37, 44, 0 | 25.3 (129.65) | -100.7 (684.43) | 56.0 (195.62) |
  CK; Week 312; n=31, 34, 43, 0: number analyzed (Participants) | 31 | 34 | 43 | 0
  CK; Week 312; n=31, 34, 43, 0 | 727.5 (4047.61) | -141.3 (681.29) | 209.4 (862.10) |
  CK; Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  CK; Week 324; n=3, 4, 3, 0 | -1.3 (168.42) | -195.0 (417.89) | 102.7 (157.82) |

28. Secondary Outcome: Change From Baseline in Creatinine and Total Bilirubin Over Time by Visit
Description: Blood samples were collected for the analysis of creatinine and total bilirubin. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: as for outcome 7
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Micromoles per liter
  Creatinine; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  Creatinine; Week 2; n=58, 56, 58, 58 | 3.36 (7.519) | 2.58 (7.273) | 4.15 (6.508) | 0.65 (7.483)
  Creatinine; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Creatinine; Week 4; n=58, 57, 59, 57 | 2.24 (6.889) | 2.50 (7.401) | 4.08 (8.072) | -0.32 (5.817)
  Creatinine; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  Creatinine; Week 8; n=58, 55, 57, 54 | 2.38 (8.371) | 2.06 (6.775) | 3.44 (8.717) | -0.92 (9.006)
  Creatinine; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Creatinine; Week 12; n=58, 53, 57, 51 | 3.39 (8.591) | 1.59 (9.300) | 3.79 (8.634) | -1.42 (9.022)
  Creatinine; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Creatinine; Week 16; n=57, 54, 57, 52 | 2.91 (11.874) | 1.10 (6.923) | 2.09 (8.967) | -2.92 (7.744)
  Creatinine; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  Creatinine; Week 20; n=56, 54, 55, 49 | 2.54 (6.384) | 0.85 (7.713) | 5.29 (9.360) | -3.26 (8.085)
  Creatinine; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Creatinine; Week 24; n=56, 53, 56, 47 | 2.52 (7.225) | 2.44 (9.391) | 4.45 (9.743) | -2.03 (15.306)
  Creatinine; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Creatinine; Week 26; n=48, 50, 53, 45 | 2.74 (7.750) | 1.80 (8.796) | 6.03 (8.465) | -2.67 (9.311)
  Creatinine; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  Creatinine; Week 28; n=51, 52, 52, 45 | 2.22 (6.606) | 2.80 (8.908) | 5.01 (9.028) | -3.42 (8.042)
  Creatinine; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  Creatinine; Week 32; n=52, 53, 55, 45 | 3.36 (8.462) | 1.69 (9.226) | 5.00 (8.690) | -3.50 (7.887)
  Creatinine; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  Creatinine; Week 36; n=52, 52, 55, 45 | 3.11 (6.652) | 3.41 (8.115) | 6.00 (8.059) | -3.26 (7.392)
  Creatinine; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  Creatinine; Week 40; n=52, 53, 55, 44 | 2.83 (7.966) | 2.36 (8.318) | 4.76 (7.858) | -2.83 (9.423)
  Creatinine; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Creatinine; Week 48; n=51, 53, 54, 44 | 2.75 (9.061) | 2.18 (8.280) | 4.47 (7.883) | -2.73 (8.533)
  Creatinine; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  Creatinine; Week 60; n=48, 47, 53, 44 | 3.28 (7.507) | 2.30 (7.998) | 4.46 (9.058) | -3.87 (7.866)
  Creatinine; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  Creatinine; Week 72; n=47, 47, 52, 42 | 3.89 (7.917) | 4.71 (7.934) | 6.59 (10.595) | -4.48 (8.461)
  Creatinine; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  Creatinine; Week 84; n=46, 48, 52, 42 | 4.58 (9.834) | 3.80 (8.761) | 6.53 (8.328) | -2.48 (8.697)
  Creatinine; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Creatinine; Week 96; n=45, 48, 52, 40 | 1.90 (11.248) | 5.34 (10.813) | 7.76 (10.318) | -2.28 (10.222)
  Creatinine; Week 108; n=43, 46, 48, 0: number analyzed (Participants) | 43 | 46 | 48 | 0
  Creatinine; Week 108; n=43, 46, 48, 0 | 5.87 (9.133) | 5.18 (7.296) | 7.26 (10.273) |
  Creatinine; Week 120; n=40, 45, 48, 0: number analyzed (Participants) | 40 | 45 | 48 | 0
  Creatinine; Week 120; n=40, 45, 48, 0 | 4.41 (8.648) | 4.15 (7.099) | 6.78 (11.811) |
  Creatinine; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  Creatinine; Week 132; n=40, 46, 49, 0 | 3.76 (8.272) | 4.02 (6.551) | 4.99 (12.168) |
  Creatinine; Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  Creatinine; Week 144; n=37, 45, 47, 0 | 5.99 (11.083) | 5.80 (6.861) | 5.07 (10.449) |
  Creatinine; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  Creatinine; Week 156; n=37, 42, 49, 0 | 5.28 (8.225) | 6.36 (6.819) | 5.16 (9.056) |
  Creatinine; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  Creatinine; Week 168; n=35, 43, 47, 0 | 6.57 (8.702) | 5.62 (8.355) | 6.82 (9.644) |
  Creatinine; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  Creatinine; Week 180; n=36, 41, 47, 0 | 5.89 (6.964) | 5.08 (7.638) | 5.91 (11.737) |
  Creatinine; Week 192; n=36, 39, 47, 0: number analyzed (Participants) | 36 | 39 | 47 | 0
  Creatinine; Week 192; n=36, 39, 47, 0 | 6.90 (9.792) | 7.91 (9.528) | 5.90 (11.316) |
  Creatinine; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  Creatinine; Week 204; n=34, 39, 47, 0 | 6.21 (9.019) | 6.46 (8.491) | 5.16 (10.629) |
  Creatinine; Week 216; n=33, 39, 46, 0: number analyzed (Participants) | 33 | 39 | 46 | 0
  Creatinine; Week 216; n=33, 39, 46, 0 | 8.34 (7.736) | 9.31 (10.863) | 7.42 (8.996) |
  Creatinine; Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Creatinine; Week 228; n=32, 39, 47, 0 | 7.16 (10.365) | 7.19 (7.388) | 6.61 (10.415) |
  Creatinine; Week 240; n=30, 39, 46, 0: number analyzed (Participants) | 30 | 39 | 46 | 0
  Creatinine; Week 240; n=30, 39, 46, 0 | 8.48 (10.016) | 7.33 (9.459) | 7.08 (10.649) |
  Creatinine; Week 252; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  Creatinine; Week 252; n=31, 38, 46, 0 | 6.96 (8.206) | 7.52 (9.245) | 7.64 (11.727) |
  Creatinine; Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  Creatinine; Week 264; n=32, 38, 47, 0 | 5.97 (7.510) | 7.10 (9.486) | 6.99 (12.140) |
  Creatinine; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  Creatinine; Week 276; n=31, 38, 45, 0 | 7.89 (8.309) | 5.84 (10.581) | 6.19 (10.418) |
  Creatinine; Week 288; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  Creatinine; Week 288; n=31, 38, 45, 0 | 8.81 (8.348) | 7.84 (9.546) | 6.20 (12.890) |
  Creatinine; Week 300; n=30, 37, 44, 0: number analyzed (Participants) | 30 | 37 | 44 | 0
  Creatinine; Week 300; n=30, 37, 44, 0 | 10.49 (8.321) | 9.16 (9.580) | 8.19 (12.114) |
  Creatinine; Week 312; n=31, 34, 43, 0: number analyzed (Participants) | 31 | 34 | 43 | 0
  Creatinine; Week 312; n=31, 34, 43, 0 | 7.98 (8.645) | 7.86 (9.096) | 7.10 (12.061) |
  Creatinine; Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  Creatinine; Week 324; n=3, 4, 3, 0 | 15.90 (6.636) | 9.75 (8.155) | 5.03 (4.007) |
  T. Bilirubin; Week 2; n=58, 56, 58, 58: number analyzed (Participants) | 58 | 56 | 58 | 58
  T. Bilirubin; Week 2; n=58, 56, 58, 58 | 0.0 (3.20) | -0.3 (2.71) | -0.4 (4.89) | -3.0 (3.82)
  T. Bilirubin; Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  T. Bilirubin; Week 4; n=58, 57, 59, 57 | 0.1 (3.39) | -0.3 (3.90) | -0.8 (5.90) | -3.4 (4.06)
  T. Bilirubin; Week 8; n=58, 55, 57, 54: number analyzed (Participants) | 58 | 55 | 57 | 54
  T. Bilirubin; Week 8; n=58, 55, 57, 54 | 0.0 (3.99) | -0.5 (3.83) | -0.6 (5.62) | -3.4 (4.24)
  T. Bilirubin; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  T. Bilirubin; Week 12; n=58, 53, 57, 51 | 0.4 (5.43) | -0.9 (3.77) | -0.5 (5.61) | -2.4 (3.75)
  T. Bilirubin; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  T. Bilirubin; Week 16; n=57, 54, 57, 52 | 0.4 (3.96) | -1.2 (3.74) | -0.2 (4.93) | -2.4 (3.79)
  T. Bilirubin; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  T. Bilirubin; Week 20; n=56, 54, 55, 49 | -0.1 (3.96) | -0.7 (3.63) | -0.4 (7.27) | -2.6 (3.83)
  T. Bilirubin; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  T. Bilirubin; Week 24; n=56, 53, 56, 47 | 0.5 (4.26) | 0.2 (4.45) | -0.7 (5.69) | -2.9 (3.86)
  T. Bilirubin; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  T. Bilirubin; Week 26; n=48, 50, 53, 45 | 1.1 (4.97) | 0.5 (3.81) | 1.0 (5.80) | -2.7 (3.44)
  T. Bilirubin; Week 28; n=51, 52, 52, 45: number analyzed (Participants) | 51 | 52 | 52 | 45
  T. Bilirubin; Week 28; n=51, 52, 52, 45 | 1.1 (4.39) | 0.7 (5.19) | 0.5 (5.25) | -2.8 (4.01)
  T. Bilirubin; Week 32; n=52, 53, 55, 45: number analyzed (Participants) | 52 | 53 | 55 | 45
  T. Bilirubin; Week 32; n=52, 53, 55, 45 | 0.7 (3.79) | 0.2 (4.99) | 0.9 (6.82) | -2.6 (3.78)
  T. Bilirubin; Week 36; n=52, 52, 55, 45: number analyzed (Participants) | 52 | 52 | 55 | 45
  T. Bilirubin; Week 36; n=52, 52, 55, 45 | 1.2 (4.94) | 0.6 (4.92) | 1.4 (6.40) | -2.7 (3.62)
  T. Bilirubin; Week 40; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  T. Bilirubin; Week 40; n=52, 53, 55, 44 | 1.6 (5.03) | 1.7 (4.75) | 1.5 (6.30) | -2.9 (3.67)
  T. Bilirubin; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  T. Bilirubin; Week 48; n=51, 53, 54, 44 | 0.9 (4.58) | 0.1 (4.51) | -0.3 (5.37) | -2.6 (3.80)
  T. Bilirubin; Week 60; n=48, 47, 53, 44: number analyzed (Participants) | 48 | 47 | 53 | 44
  T. Bilirubin; Week 60; n=48, 47, 53, 44 | 1.9 (4.31) | 0.0 (4.78) | 0.9 (6.56) | -2.2 (3.86)
  T. Bilirubin; Week 72; n=47, 47, 52, 42: number analyzed (Participants) | 47 | 47 | 52 | 42
  T. Bilirubin; Week 72; n=47, 47, 52, 42 | 1.5 (6.05) | 0.1 (4.59) | 0.6 (6.36) | -2.7 (3.69)
  T. Bilirubin; Week 84; n=46, 48, 52, 42: number analyzed (Participants) | 46 | 48 | 52 | 42
  T. Bilirubin; Week 84; n=46, 48, 52, 42 | 2.3 (5.09) | 0.1 (5.07) | 1.2 (5.49) | -2.6 (4.27)
  T. Bilirubin; Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  T. Bilirubin; Week 96; n=45, 48, 52, 40 | 1.0 (4.15) | 0.0 (5.80) | 1.7 (5.42) | -2.5 (3.92)
  T. Bilirubin; Week 108; n=43, 46, 48, 0: number analyzed (Participants) | 43 | 46 | 48 | 0
  T. Bilirubin; Week 108; n=43, 46, 48, 0 | 0.7 (4.86) | 1.4 (6.34) | 0.8 (5.89) |
  T. Bilirubin; Week 120; n=40, 45, 48, 0: number analyzed (Participants) | 40 | 45 | 48 | 0
  T. Bilirubin; Week 120; n=40, 45, 48, 0 | 0.9 (4.96) | 1.1 (4.72) | 1.3 (7.40) |
  T. Bilirubin; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  T. Bilirubin; Week 132; n=40, 46, 49, 0 | 1.0 (6.16) | 2.0 (8.03) | 1.1 (6.40) |
  T. Bilirubin; Week 144; n=37, 45, 47, 0: number analyzed (Participants) | 37 | 45 | 47 | 0
  T. Bilirubin; Week 144; n=37, 45, 47, 0 | 0.7 (4.70) | 1.1 (7.00) | 0.4 (6.50) |
  T. Bilirubin; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  T. Bilirubin; Week 156; n=37, 42, 49, 0 | 1.6 (5.07) | 1.0 (5.23) | 1.0 (6.93) |
  T. Bilirubin; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  T. Bilirubin; Week 168; n=35, 43, 47, 0 | 1.1 (5.37) | 0.8 (4.19) | 1.4 (5.94) |
  T. Bilirubin; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  T. Bilirubin; Week 180; n=36, 41, 47, 0 | 1.1 (5.54) | 0.0 (4.29) | 1.0 (7.42) |
  T. Bilirubin; Week 192; n=36, 39, 47, 0: number analyzed (Participants) | 36 | 39 | 47 | 0
  T. Bilirubin; Week 192; n=36, 39, 47, 0 | 0.7 (5.88) | 0.3 (4.80) | 0.9 (6.18) |
  T. Bilirubin; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  T. Bilirubin; Week 204; n=34, 39, 47, 0 | 1.1 (5.31) | 0.7 (3.71) | 0.6 (6.61) |
  T. Bilirubin; Week 216; n=33, 39, 46, 0: number analyzed (Participants) | 33 | 39 | 46 | 0
  T. Bilirubin; Week 216; n=33, 39, 46, 0 | 0.5 (5.08) | 0.8 (6.69) | 0.3 (5.91) |
  T. Bilirubin; Week 228; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  T. Bilirubin; Week 228; n=32, 39, 47, 0 | 1.6 (4.61) | 0.5 (3.77) | -0.3 (5.71) |
  T. Bilirubin; Week 240; n=30, 39, 46, 0: number analyzed (Participants) | 30 | 39 | 46 | 0
  T. Bilirubin; Week 240; n=30, 39, 46, 0 | 1.2 (4.92) | 0.9 (4.72) | -0.1 (4.83) |
  T. Bilirubin; Week 252; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  T. Bilirubin; Week 252; n=31, 38, 46, 0 | 1.4 (5.71) | 2.0 (6.03) | 0.2 (6.21) |
  T. Bilirubin; Week 264; n=32, 38, 47, 0: number analyzed (Participants) | 32 | 38 | 47 | 0
  T. Bilirubin; Week 264; n=32, 38, 47, 0 | 0.4 (5.76) | 2.9 (8.95) | -0.1 (6.11) |
  T. Bilirubin; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  T. Bilirubin; Week 276; n=31, 38, 45, 0 | 0.7 (3.52) | 2.8 (10.40) | 0.9 (6.46) |
  T. Bilirubin; Week 288; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  T. Bilirubin; Week 288; n=31, 38, 45, 0 | 0.5 (5.06) | 1.9 (7.87) | 0.0 (6.10) |
  T. Bilirubin; Week 300; n=30, 37, 44, 0: number analyzed (Participants) | 30 | 37 | 44 | 0
  T. Bilirubin; Week 300; n=30, 37, 44, 0 | 1.1 (4.22) | 1.7 (8.78) | 0.9 (5.18) |
  T. Bilirubin; Week 312; n=31, 34, 43, 0: number analyzed (Participants) | 31 | 34 | 43 | 0
  T. Bilirubin; Week 312; n=31, 34, 43, 0 | 1.4 (5.30) | 1.1 (7.12) | 0.8 (5.52) |
  T. Bilirubin; Week 324; n=3, 4, 3, 0: number analyzed (Participants) | 3 | 4 | 3 | 0
  T. Bilirubin; Week 324; n=3, 4, 3, 0 | 5.3 (4.16) | 5.5 (11.47) | 0.7 (4.16) |

29. Secondary Outcome: Change From Baseline in Estimated Creatinine Clearance Over Time by Visit
Description: Blood samples were collected for the analysis of estimated creatinine clearance. Estimated creatinine clearance was calculated using Cockcroft-Gault formula. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 8, 16, 20, 24, 26, 40, 48, 60, 96, 180, 204, 252 and 264
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Milliliters per minute
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Milliliters per minute
  Week 2; n=1, 1, 0, 3: number analyzed (Participants) | 1 | 1 | 0 | 3
  Week 2; n=1, 1, 0, 3 | -3.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  | -0.7 (0.58)
  Week 4; n=58, 57, 59, 57: number analyzed (Participants) | 58 | 57 | 59 | 57
  Week 4; n=58, 57, 59, 57 | -1.4 (12.20) | -3.7 (12.18) | -4.9 (14.83) | -0.1 (10.06)
  Week 8; n=2, 1, 1, 1: number analyzed (Participants) | 2 | 1 | 1 | 1
  Week 8; n=2, 1, 1, 1 | 5.5 (26.16) | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | 7.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  Week 16; n=55, 53, 56, 49: number analyzed (Participants) | 55 | 53 | 56 | 49
  Week 16; n=55, 53, 56, 49 | 2.2 (37.66) | 0.2 (15.60) | -2.7 (13.89) | 3.4 (12.94)
  Week 20; n=2, 0, 0, 1: number analyzed (Participants) | 2 | 0 | 0 | 1
  Week 20; n=2, 0, 0, 1 | 8.0 (7.07) |  |  | 4.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  Week 24; n=52, 53, 55, 46: number analyzed (Participants) | 52 | 53 | 55 | 46
  Week 24; n=52, 53, 55, 46 | -2.7 (22.03) | -6.4 (34.13) | -5.8 (14.77) | 4.8 (15.66)
  Week 26; n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 26; n=0, 1, 0, 0 |  | -7.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |
  Week 40; n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 40; n=0, 1, 0, 0 |  | -95.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |
  Week 48; n=51, 50, 54, 44: number analyzed (Participants) | 51 | 50 | 54 | 44
  Week 48; n=51, 50, 54, 44 | -2.6 (12.72) | -1.1 (16.63) | -4.5 (14.27) | 0.4 (19.04)
  Week 60; n=0, 0, 0, 1: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 60; n=0, 0, 0, 1 |  |  |  | 16.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  Week 96; n=45, 48, 52, 40: number analyzed (Participants) | 45 | 48 | 52 | 40
  Week 96; n=45, 48, 52, 40 | 2.2 (31.70) | -2.4 (20.43) | -9.0 (16.95) | 5.1 (22.48)
  Week 180; n=1, 0, 0, 0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 180; n=1, 0, 0, 0 | 1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |  |
  Week 204; n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 204; n=0, 1, 0, 0 |  | -23.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |
  Week 252; n=0, 1, 0, 0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 252; n=0, 1, 0, 0 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |  |
  Week 264; n=0, 0, 1, 0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Week 264; n=0, 0, 1, 0 |  |  | -143.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point |

30. Secondary Outcome: Change From Baseline in Hemoglobin Level Over Time by Visit
Description: Blood samples were collected for the analysis of hemoglobin level. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: as for outcome 7
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Grams per liter
  Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Week 2; n=57, 56, 59, 59 | 0.1 (6.66) | 0.0 (6.25) | -0.7 (6.61) | 0.7 (6.90)
  Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  Week 4; n=57, 57, 59, 57 | -0.2 (6.41) | 0.5 (5.61) | 0.6 (7.67) | 0.7 (6.40)
  Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  Week 8; n=58, 56, 56, 55 | 2.7 (9.19) | 4.8 (7.23) | 2.0 (8.99) | 2.0 (9.18)
  Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Week 12; n=58, 53, 57, 51 | 2.0 (8.27) | 3.9 (7.84) | 2.6 (9.59) | 2.8 (8.57)
  Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Week 16; n=57, 54, 57, 52 | 1.1 (7.58) | 3.5 (7.55) | 2.3 (9.61) | 1.1 (9.22)
  Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  Week 20; n=56, 54, 55, 49 | 2.1 (8.78) | 3.8 (9.28) | 3.1 (9.66) | 0.8 (9.22)
  Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Week 24; n=56, 53, 56, 47 | 2.6 (9.17) | 4.8 (7.66) | 3.6 (11.04) | 1.9 (8.16)
  Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Week 26; n=48, 50, 53, 45 | 1.8 (7.68) | 3.4 (8.00) | 2.5 (9.17) | 2.2 (8.11)
  Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  Week 28; n=50, 52, 52, 45 | 1.7 (8.51) | 4.0 (7.93) | 1.5 (8.50) | 0.1 (10.50)
  Week 32; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  Week 32; n=51, 53, 55, 45 | 1.6 (8.64) | 3.1 (8.71) | 3.5 (8.49) | 0.6 (8.92)
  Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  Week 36; n=52, 53, 55, 44 | 0.3 (10.21) | 2.9 (9.69) | 2.7 (11.59) | -0.8 (9.79)
  Week 40; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  Week 40; n=51, 53, 55, 45 | 0.5 (11.44) | 2.2 (8.56) | 2.1 (9.46) | -0.2 (7.67)
  Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  Week 48; n=51, 53, 54, 44 | 1.2 (9.84) | 2.7 (8.40) | -0.5 (12.03) | 0.0 (9.52)
  Week 60; n=48, 47, 52, 44: number analyzed (Participants) | 48 | 47 | 52 | 44
  Week 60; n=48, 47, 52, 44 | 2.6 (11.23) | 4.7 (8.73) | 2.2 (11.45) | 2.3 (9.18)
  Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Week 72; n=47, 48, 52, 42 | 1.8 (11.28) | 4.5 (7.39) | 2.4 (10.08) | 2.4 (9.15)
  Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  Week 84; n=46, 48, 51, 42 | 3.3 (11.53) | 4.0 (8.37) | 3.0 (11.34) | 1.7 (9.65)
  Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  Week 96; n=46, 46, 52, 41 | 2.7 (13.41) | 3.3 (6.94) | 3.6 (10.11) | 1.9 (10.06)
  Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  Week 108; n=43, 46, 49, 0 | 4.0 (11.77) | 3.4 (9.42) | 3.0 (10.98) |
  Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  Week 120; n=41, 46, 49, 0 | 4.2 (11.11) | 4.7 (8.72) | 2.1 (11.39) |
  Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  Week 132; n=40, 46, 49, 0 | 3.5 (10.89) | 3.0 (9.90) | 2.5 (12.41) |
  Week 144; n=37, 45, 46, 0: number analyzed (Participants) | 37 | 45 | 46 | 0
  Week 144; n=37, 45, 46, 0 | 4.0 (12.08) | 2.6 (10.64) | 2.3 (11.37) |
  Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  Week 156; n=37, 42, 49, 0 | 4.0 (11.55) | 5.1 (9.76) | 2.7 (11.88) |
  Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  Week 168; n=35, 43, 47, 0 | 6.3 (12.60) | 6.0 (10.91) | 4.8 (10.60) |
  Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  Week 180; n=36, 41, 47, 0 | 5.5 (11.79) | 4.0 (9.23) | 2.7 (11.68) |
  Week 192; n=35, 40, 47, 0: number analyzed (Participants) | 35 | 40 | 47 | 0
  Week 192; n=35, 40, 47, 0 | 3.3 (13.07) | 3.5 (9.55) | 3.0 (11.51) |
  Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  Week 204; n=34, 39, 47, 0 | 4.5 (12.73) | 4.7 (9.84) | 3.2 (11.65) |
  Week 216; n=32, 39, 44, 0: number analyzed (Participants) | 32 | 39 | 44 | 0
  Week 216; n=32, 39, 44, 0 | 4.7 (14.10) | 4.1 (9.97) | 3.4 (10.60) |
  Week 228; n=31, 39, 47, 0: number analyzed (Participants) | 31 | 39 | 47 | 0
  Week 228; n=31, 39, 47, 0 | 5.1 (13.32) | 4.8 (10.55) | 3.1 (10.53) |
  Week 240; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Week 240; n=32, 39, 47, 0 | 6.2 (14.38) | 5.8 (10.64) | 2.1 (11.70) |
  Week 252; n=31, 36, 45, 0: number analyzed (Participants) | 31 | 36 | 45 | 0
  Week 252; n=31, 36, 45, 0 | 6.2 (14.98) | 6.4 (11.76) | 5.8 (10.33) |
  Week 264; n=32, 38, 46, 0: number analyzed (Participants) | 32 | 38 | 46 | 0
  Week 264; n=32, 38, 46, 0 | 6.3 (14.69) | 6.0 (9.28) | 5.5 (11.07) |
  Week 276; n=31, 38, 46, 0: number analyzed (Participants) | 31 | 38 | 46 | 0
  Week 276; n=31, 38, 46, 0 | 6.6 (14.67) | 5.5 (11.06) | 5.4 (10.02) |
  Week 288; n=30, 38, 44, 0: number analyzed (Participants) | 30 | 38 | 44 | 0
  Week 288; n=30, 38, 44, 0 | 7.3 (12.51) | 6.8 (11.38) | 6.9 (10.82) |
  Week 300; n=30, 37, 43, 0: number analyzed (Participants) | 30 | 37 | 43 | 0
  Week 300; n=30, 37, 43, 0 | 4.6 (15.39) | 5.1 (10.47) | 5.5 (11.56) |
  Week 312; n=31, 33, 42, 0: number analyzed (Participants) | 31 | 33 | 42 | 0
  Week 312; n=31, 33, 42, 0 | 7.0 (13.56) | 6.1 (9.29) | 8.0 (10.10) |
  Week 324; n=3, 4, 2, 0: number analyzed (Participants) | 3 | 4 | 2 | 0
  Week 324; n=3, 4, 2, 0 | 4.3 (9.07) | 10.0 (14.33) | 20.5 (7.78) |

31. Secondary Outcome: Change From Baseline in Total Neutrophils, Platelet Count and WBC Count Over Time by Visit
Description: Blood samples were collected for the analysis of total neutrophils, platelet count and WBC count. Baseline value is the last pre-treatment value observed. Change from Baseline is calculated as value at indicated time point minus Baseline value.
Time Frame: as for outcome 7
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Giga cells per liter
  T. neutrophils; Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  T. neutrophils; Week 2; n=57, 56, 59, 59 | 0.042 (1.0528) | -0.084 (1.4018) | 0.104 (1.0318) | 0.716 (1.4565)
  T. neutrophils; Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  T. neutrophils; Week 4; n=57, 57, 59, 57 | 0.038 (1.2691) | -0.083 (1.2859) | 0.155 (1.0877) | 0.375 (1.5303)
  T. neutrophils; Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  T. neutrophils; Week 8; n=58, 56, 56, 55 | 0.251 (1.0956) | -0.066 (1.3186) | 0.341 (1.2077) | 0.273 (0.8715)
  T. neutrophils; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  T. neutrophils; Week 12; n=58, 53, 57, 51 | 0.138 (1.2352) | 0.040 (1.4855) | 0.359 (1.3585) | 0.525 (1.5661)
  T. neutrophils; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  T. neutrophils; Week 16; n=57, 54, 57, 52 | 0.388 (1.7066) | -0.156 (1.2694) | 0.203 (1.0459) | 0.367 (1.2022)
  T. neutrophils; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  T. neutrophils; Week 20; n=56, 54, 55, 49 | 0.270 (1.3671) | 0.032 (1.3837) | 0.525 (1.6689) | 0.740 (1.7181)
  T. neutrophils; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  T. neutrophils; Week 24; n=56, 53, 56, 47 | 0.462 (1.1725) | 0.109 (1.7578) | 0.406 (1.0404) | 0.637 (1.5583)
  T. neutrophils; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  T. neutrophils; Week 26; n=48, 50, 53, 45 | 0.120 (0.8908) | 0.052 (1.7443) | 0.375 (1.1565) | 0.449 (1.3271)
  T. neutrophils; Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  T. neutrophils; Week 28; n=50, 52, 52, 45 | 0.496 (1.1330) | 0.213 (1.4523) | 0.502 (1.2817) | 0.446 (1.1851)
  T. neutrophils; Week 32; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  T. neutrophils; Week 32; n=51, 53, 55, 45 | 0.071 (1.3373) | 0.149 (1.5137) | 0.692 (1.4994) | 0.717 (1.5595)
  T. neutrophils; Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  T. neutrophils; Week 36; n=52, 53, 55, 44 | 0.420 (1.4246) | 0.029 (1.7516) | 0.535 (1.0695) | 0.414 (1.3998)
  T. neutrophils; Week 40; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  T. neutrophils; Week 40; n=51, 53, 55, 45 | 0.430 (1.4711) | 0.178 (1.3099) | 0.575 (1.0510) | 0.730 (1.4181)
  T. neutrophils; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  T. neutrophils; Week 48; n=51, 53, 54, 44 | 0.386 (1.3376) | 0.245 (1.5695) | 0.534 (1.3432) | 0.665 (1.6752)
  T. neutrophils; Week 60; n=48, 47, 52, 44: number analyzed (Participants) | 48 | 47 | 52 | 44
  T. neutrophils; Week 60; n=48, 47, 52, 44 | 0.374 (1.4938) | 0.458 (1.6323) | 0.711 (0.9216) | 0.800 (1.4058)
  T. neutrophils; Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  T. neutrophils; Week 72; n=47, 48, 52, 42 | 0.383 (1.6125) | 0.274 (1.5663) | 0.666 (1.2125) | 0.892 (1.9492)
  T. neutrophils; Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  T. neutrophils; Week 84; n=46, 48, 51, 42 | 0.410 (1.6209) | 0.528 (1.6303) | 1.006 (1.4287) | 0.790 (1.7937)
  T. neutrophils; Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  T. neutrophils; Week 96; n=46, 46, 52, 41 | 0.631 (1.3478) | 0.698 (1.8981) | 0.997 (1.3089) | 0.831 (1.4347)
  T. neutrophils; Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  T. neutrophils; Week 108; n=43, 46, 49, 0 | 0.623 (1.7946) | 0.570 (1.5706) | 1.006 (1.6122) |
  T. neutrophils; Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  T. neutrophils; Week 120; n=41, 46, 49, 0 | 0.372 (1.7590) | 0.650 (1.8334) | 0.769 (1.6486) |
  T. neutrophils; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  T. neutrophils; Week 132; n=40, 46, 49, 0 | 0.777 (2.1995) | 0.405 (1.6979) | 0.671 (1.0761) |
  T. neutrophils; Week 144; n=37, 45, 46, 0: number analyzed (Participants) | 37 | 45 | 46 | 0
  T. neutrophils; Week 144; n=37, 45, 46, 0 | 0.672 (1.3974) | 0.468 (1.6210) | 0.831 (1.4397) |
  T. neutrophils; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  T. neutrophils; Week 156; n=37, 42, 49, 0 | 0.762 (1.7331) | 0.418 (1.6395) | 1.095 (1.2219) |
  T. neutrophils; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  T. neutrophils; Week 168; n=35, 43, 47, 0 | 0.588 (1.5738) | 0.534 (1.6710) | 1.011 (1.2304) |
  T. neutrophils; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  T. neutrophils; Week 180; n=36, 41, 47, 0 | 0.769 (1.4717) | 0.405 (1.7183) | 0.840 (1.0957) |
  T. neutrophils; Week 192; n=35, 40, 47, 0: number analyzed (Participants) | 35 | 40 | 47 | 0
  T. neutrophils; Week 192; n=35, 40, 47, 0 | 0.490 (1.3807) | 0.594 (1.7286) | 0.722 (1.2591) |
  T. neutrophils; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  T. neutrophils; Week 204; n=34, 39, 47, 0 | 0.618 (1.7745) | 0.648 (1.7939) | 0.821 (1.4259) |
  T. neutrophils; Week 216; n=32, 39, 43, 0: number analyzed (Participants) | 32 | 39 | 43 | 0
  T. neutrophils; Week 216; n=32, 39, 43, 0 | 0.543 (1.7307) | 0.588 (1.5854) | 0.914 (1.4470) |
  T. neutrophils; Week 228; n=30, 39, 47, 0: number analyzed (Participants) | 30 | 39 | 47 | 0
  T. neutrophils; Week 228; n=30, 39, 47, 0 | 0.780 (1.7170) | 0.789 (1.6779) | 0.819 (1.1182) |
  T. neutrophils; Week 240; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  T. neutrophils; Week 240; n=32, 39, 47, 0 | 0.508 (1.4277) | 0.813 (1.7505) | 1.083 (2.3145) |
  T. neutrophils; Week 252; n=31, 36, 45, 0: number analyzed (Participants) | 31 | 36 | 45 | 0
  T. neutrophils; Week 252; n=31, 36, 45, 0 | 0.268 (1.4164) | 0.761 (1.5531) | 0.812 (1.3345) |
  T. neutrophils; Week 264; n=32, 38, 46, 0: number analyzed (Participants) | 32 | 38 | 46 | 0
  T. neutrophils; Week 264; n=32, 38, 46, 0 | 0.475 (1.7483) | 0.761 (1.7316) | 1.176 (1.6844) |
  T. neutrophils; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  T. neutrophils; Week 276; n=31, 38, 45, 0 | 0.400 (1.6597) | 0.627 (1.8500) | 1.106 (1.3666) |
  T. neutrophils; Week 288; n=30, 38, 44, 0: number analyzed (Participants) | 30 | 38 | 44 | 0
  T. neutrophils; Week 288; n=30, 38, 44, 0 | 0.456 (1.8521) | 0.673 (1.9230) | 0.913 (1.5880) |
  T. neutrophils; Week 300; n=30, 37, 43, 0: number analyzed (Participants) | 30 | 37 | 43 | 0
  T. neutrophils; Week 300; n=30, 37, 43, 0 | 0.139 (1.2243) | 0.455 (1.4957) | 0.699 (1.1030) |
  T. neutrophils; Week 312; n=31, 33, 41, 0: number analyzed (Participants) | 31 | 33 | 41 | 0
  T. neutrophils; Week 312; n=31, 33, 41, 0 | 0.243 (1.3595) | 0.417 (1.7807) | 0.564 (1.1666) |
  T. neutrophils; Week 324; n=3, 4, 2, 0: number analyzed (Participants) | 3 | 4 | 2 | 0
  T. neutrophils; Week 324; n=3, 4, 2, 0 | 0.860 (2.7921) | 0.315 (1.0660) | 0.960 (0.4950) |
  Platelet count; Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  Platelet count; Week 2; n=57, 56, 59, 59 | 11.0 (30.21) | 16.6 (27.48) | 14.3 (22.17) | 17.1 (33.56)
  Platelet count; Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  Platelet count; Week 4; n=57, 57, 59, 57 | 9.9 (27.70) | 20.1 (30.52) | 14.1 (21.35) | 15.6 (38.98)
  Platelet count; Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  Platelet count; Week 8; n=58, 56, 56, 55 | 10.3 (26.33) | 25.9 (33.21) | 18.4 (27.51) | 10.3 (36.86)
  Platelet count; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  Platelet count; Week 12; n=58, 53, 57, 51 | 13.7 (28.85) | 14.6 (35.00) | 17.7 (33.02) | 11.2 (43.26)
  Platelet count; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  Platelet count; Week 16; n=57, 54, 57, 52 | 16.5 (36.43) | 11.3 (30.85) | 17.9 (34.32) | 9.3 (40.36)
  Platelet count; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  Platelet count; Week 20; n=56, 54, 55, 49 | 17.2 (32.75) | 14.5 (29.72) | 13.7 (32.98) | 17.1 (43.06)
  Platelet count; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  Platelet count; Week 24; n=56, 53, 56, 47 | 12.0 (31.51) | 18.4 (34.30) | 19.3 (27.64) | 23.9 (49.14)
  Platelet count; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  Platelet count; Week 26; n=48, 50, 53, 45 | 8.3 (32.59) | 11.2 (36.32) | 10.3 (30.94) | 17.5 (40.38)
  Platelet count; Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  Platelet count; Week 28; n=50, 52, 52, 45 | 6.6 (33.00) | 15.8 (34.97) | 17.8 (27.83) | 17.2 (44.39)
  Platelet count; Week 32; n=51, 52, 55, 45: number analyzed (Participants) | 51 | 52 | 55 | 45
  Platelet count; Week 32; n=51, 52, 55, 45 | 7.7 (41.79) | 11.6 (36.27) | 15.4 (27.19) | 13.8 (38.26)
  Platelet count; Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  Platelet count; Week 36; n=52, 53, 55, 44 | 5.2 (39.32) | 10.8 (39.28) | 11.8 (32.72) | 12.3 (43.83)
  Platelet count; Week 40; n=51, 53, 54, 45: number analyzed (Participants) | 51 | 53 | 54 | 45
  Platelet count; Week 40; n=51, 53, 54, 45 | 11.1 (44.07) | 8.9 (31.95) | 7.8 (31.86) | 18.9 (36.94)
  Platelet count; Week 48; n=51, 52, 53, 44: number analyzed (Participants) | 51 | 52 | 53 | 44
  Platelet count; Week 48; n=51, 52, 53, 44 | 12.5 (41.82) | 20.0 (38.20) | 17.6 (38.70) | 20.6 (42.78)
  Platelet count; Week 60; n=48, 47, 51, 44: number analyzed (Participants) | 48 | 47 | 51 | 44
  Platelet count; Week 60; n=48, 47, 51, 44 | 20.9 (39.25) | 18.7 (34.22) | 26.6 (37.23) | 30.8 (43.09)
  Platelet count; Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  Platelet count; Week 72; n=47, 48, 52, 42 | 23.7 (37.03) | 22.8 (32.35) | 22.7 (35.13) | 28.3 (37.19)
  Platelet count; Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  Platelet count; Week 84; n=46, 48, 51, 42 | 13.6 (42.78) | 17.2 (32.00) | 21.1 (38.36) | 18.9 (44.07)
  Platelet count; Week 96; n=46, 45, 51, 41: number analyzed (Participants) | 46 | 45 | 51 | 41
  Platelet count; Week 96; n=46, 45, 51, 41 | 25.9 (39.73) | 20.8 (39.00) | 21.7 (36.57) | 17.5 (40.11)
  Platelet count; Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  Platelet count; Week 108; n=43, 46, 49, 0 | 24.5 (44.43) | 24.6 (30.23) | 33.1 (46.23) |
  Platelet count; Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  Platelet count; Week 120; n=41, 46, 49, 0 | 23.8 (48.05) | 26.9 (33.58) | 20.4 (31.47) |
  Platelet count; Week 132; n=40, 46, 48, 0: number analyzed (Participants) | 40 | 46 | 48 | 0
  Platelet count; Week 132; n=40, 46, 48, 0 | 16.8 (33.67) | 21.0 (35.98) | 32.2 (35.34) |
  Platelet count; Week 144; n=37, 45, 44, 0: number analyzed (Participants) | 37 | 45 | 44 | 0
  Platelet count; Week 144; n=37, 45, 44, 0 | 27.1 (50.68) | 23.2 (31.97) | 33.5 (54.61) |
  Platelet count; Week 156; n=37, 42, 47, 0: number analyzed (Participants) | 37 | 42 | 47 | 0
  Platelet count; Week 156; n=37, 42, 47, 0 | 26.6 (53.14) | 30.6 (37.65) | 41.2 (47.37) |
  Platelet count; Week 168; n=35, 43, 46, 0: number analyzed (Participants) | 35 | 43 | 46 | 0
  Platelet count; Week 168; n=35, 43, 46, 0 | 34.9 (43.78) | 36.4 (37.72) | 40.0 (50.19) |
  Platelet count; Week 180; n=36, 41, 46, 0: number analyzed (Participants) | 36 | 41 | 46 | 0
  Platelet count; Week 180; n=36, 41, 46, 0 | 28.4 (48.03) | 27.6 (36.53) | 45.4 (54.46) |
  Platelet count; Week 192; n=35, 40, 46, 0: number analyzed (Participants) | 35 | 40 | 46 | 0
  Platelet count; Week 192; n=35, 40, 46, 0 | 34.7 (58.72) | 24.6 (37.42) | 27.9 (45.02) |
  Platelet count; Week 204; n=34, 39, 45, 0: number analyzed (Participants) | 34 | 39 | 45 | 0
  Platelet count; Week 204; n=34, 39, 45, 0 | 33.9 (59.13) | 26.4 (31.26) | 37.6 (45.21) |
  Platelet count; Week 216; n=32, 39, 44, 0: number analyzed (Participants) | 32 | 39 | 44 | 0
  Platelet count; Week 216; n=32, 39, 44, 0 | 28.1 (48.97) | 25.2 (31.60) | 33.5 (44.09) |
  Platelet count; Week 228; n=31, 39, 46, 0: number analyzed (Participants) | 31 | 39 | 46 | 0
  Platelet count; Week 228; n=31, 39, 46, 0 | 28.7 (49.38) | 27.1 (35.77) | 29.1 (41.22) |
  Platelet count; Week 240; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  Platelet count; Week 240; n=32, 39, 47, 0 | 27.2 (52.69) | 26.2 (31.38) | 27.4 (42.22) |
  Platelet count; Week 252; n=31, 36, 44, 0: number analyzed (Participants) | 31 | 36 | 44 | 0
  Platelet count; Week 252; n=31, 36, 44, 0 | 15.9 (48.02) | 15.4 (31.97) | 30.8 (39.37) |
  Platelet count; Week 264; n=32, 38, 45, 0: number analyzed (Participants) | 32 | 38 | 45 | 0
  Platelet count; Week 264; n=32, 38, 45, 0 | 27.9 (48.97) | 23.2 (29.82) | 32.8 (43.26) |
  Platelet count; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  Platelet count; Week 276; n=31, 38, 45, 0 | 48.4 (55.68) | 34.5 (34.41) | 45.8 (41.35) |
  Platelet count; Week 288; n=30, 38, 43, 0: number analyzed (Participants) | 30 | 38 | 43 | 0
  Platelet count; Week 288; n=30, 38, 43, 0 | 44.1 (60.21) | 35.5 (34.89) | 46.7 (43.13) |
  Platelet count; Week 300; n=30, 37, 40, 0: number analyzed (Participants) | 30 | 37 | 40 | 0
  Platelet count; Week 300; n=30, 37, 40, 0 | 28.5 (55.51) | 26.8 (36.02) | 45.4 (39.15) |
  Platelet count; Week 312; n=31, 33, 41, 0: number analyzed (Participants) | 31 | 33 | 41 | 0
  Platelet count; Week 312; n=31, 33, 41, 0 | 27.3 (52.62) | 30.9 (34.28) | 35.3 (37.26) |
  Platelet count; Week 324; n=3, 4, 2, 0: number analyzed (Participants) | 3 | 4 | 2 | 0
  Platelet count; Week 324; n=3, 4, 2, 0 | 31.7 (17.47) | 8.3 (7.46) | 2.0 (9.90) |
  WBC count; Week 2; n=57, 56, 59, 59: number analyzed (Participants) | 57 | 56 | 59 | 59
  WBC count; Week 2; n=57, 56, 59, 59 | 0.19 (1.176) | 0.13 (1.506) | 0.31 (1.314) | 0.69 (1.606)
  WBC count; Week 4; n=57, 57, 59, 57: number analyzed (Participants) | 57 | 57 | 59 | 57
  WBC count; Week 4; n=57, 57, 59, 57 | 0.16 (1.493) | 0.02 (1.435) | 0.30 (1.263) | 0.29 (1.753)
  WBC count; Week 8; n=58, 56, 56, 55: number analyzed (Participants) | 58 | 56 | 56 | 55
  WBC count; Week 8; n=58, 56, 56, 55 | 0.37 (1.298) | 0.15 (1.595) | 0.48 (1.283) | 0.27 (1.123)
  WBC; Week 12; n=58, 53, 57, 51: number analyzed (Participants) | 58 | 53 | 57 | 51
  WBC; Week 12; n=58, 53, 57, 51 | 0.32 (1.427) | 0.28 (1.696) | 0.73 (1.375) | 0.54 (1.734)
  WBC count; Week 16; n=57, 54, 57, 52: number analyzed (Participants) | 57 | 54 | 57 | 52
  WBC count; Week 16; n=57, 54, 57, 52 | 0.45 (1.806) | 0.02 (1.554) | 0.36 (1.080) | 0.36 (1.542)
  WBC count; Week 20; n=56, 54, 55, 49: number analyzed (Participants) | 56 | 54 | 55 | 49
  WBC count; Week 20; n=56, 54, 55, 49 | 0.36 (1.510) | 0.23 (1.523) | 0.77 (1.848) | 0.78 (1.821)
  WBC count; Week 24; n=56, 53, 56, 47: number analyzed (Participants) | 56 | 53 | 56 | 47
  WBC count; Week 24; n=56, 53, 56, 47 | 0.47 (1.245) | 0.34 (2.060) | 0.64 (1.226) | 0.55 (1.822)
  WBC count; Week 26; n=48, 50, 53, 45: number analyzed (Participants) | 48 | 50 | 53 | 45
  WBC count; Week 26; n=48, 50, 53, 45 | 0.19 (1.130) | 0.26 (2.039) | 0.66 (1.257) | 0.35 (1.578)
  WBC count; Week 28; n=50, 52, 52, 45: number analyzed (Participants) | 50 | 52 | 52 | 45
  WBC count; Week 28; n=50, 52, 52, 45 | 0.67 (1.412) | 0.42 (1.685) | 0.69 (1.428) | 0.39 (1.416)
  WBC count; Week 32; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  WBC count; Week 32; n=51, 53, 55, 45 | 0.25 (1.598) | 0.45 (1.767) | 0.93 (1.704) | 0.71 (1.820)
  WBC count; Week 36; n=52, 53, 55, 44: number analyzed (Participants) | 52 | 53 | 55 | 44
  WBC count; Week 36; n=52, 53, 55, 44 | 0.56 (1.532) | 0.30 (2.068) | 0.92 (1.178) | 0.36 (1.547)
  WBC count; Week 40; n=51, 53, 55, 45: number analyzed (Participants) | 51 | 53 | 55 | 45
  WBC count; Week 40; n=51, 53, 55, 45 | 0.57 (1.668) | 0.42 (1.654) | 0.81 (1.205) | 0.75 (1.680)
  WBC count; Week 48; n=51, 53, 54, 44: number analyzed (Participants) | 51 | 53 | 54 | 44
  WBC count; Week 48; n=51, 53, 54, 44 | 0.43 (1.499) | 0.53 (1.912) | 0.78 (1.447) | 0.73 (1.874)
  WBC count; Week 60; n=48, 47, 52, 44: number analyzed (Participants) | 48 | 47 | 52 | 44
  WBC count; Week 60; n=48, 47, 52, 44 | 0.60 (1.774) | 0.76 (1.686) | 1.04 (1.160) | 0.95 (1.735)
  WBC count; Week 72; n=47, 48, 52, 42: number analyzed (Participants) | 47 | 48 | 52 | 42
  WBC count; Week 72; n=47, 48, 52, 42 | 0.63 (1.932) | 0.56 (1.917) | 1.09 (1.378) | 1.02 (2.280)
  WBC count; Week 84; n=46, 48, 51, 42: number analyzed (Participants) | 46 | 48 | 51 | 42
  WBC count; Week 84; n=46, 48, 51, 42 | 0.71 (1.805) | 0.96 (1.914) | 1.43 (1.622) | 0.95 (1.893)
  WBC count; Week 96; n=46, 46, 52, 41: number analyzed (Participants) | 46 | 46 | 52 | 41
  WBC count; Week 96; n=46, 46, 52, 41 | 0.95 (1.687) | 1.01 (2.069) | 1.38 (1.405) | 0.92 (1.624)
  WBC count; Week 108; n=43, 46, 49, 0: number analyzed (Participants) | 43 | 46 | 49 | 0
  WBC count; Week 108; n=43, 46, 49, 0 | 0.89 (2.190) | 0.90 (1.714) | 1.35 (1.749) |
  WBC count; Week 120; n=41, 46, 49, 0: number analyzed (Participants) | 41 | 46 | 49 | 0
  WBC count; Week 120; n=41, 46, 49, 0 | 0.59 (1.931) | 1.01 (1.988) | 1.16 (1.632) |
  WBC count; Week 132; n=40, 46, 49, 0: number analyzed (Participants) | 40 | 46 | 49 | 0
  WBC count; Week 132; n=40, 46, 49, 0 | 0.92 (2.274) | 0.71 (1.958) | 1.02 (1.103) |
  WBC count; Week 144; n=37, 45, 46, 0: number analyzed (Participants) | 37 | 45 | 46 | 0
  WBC count; Week 144; n=37, 45, 46, 0 | 0.91 (1.667) | 0.82 (1.727) | 1.22 (1.785) |
  WBC count; Week 156; n=37, 42, 49, 0: number analyzed (Participants) | 37 | 42 | 49 | 0
  WBC count; Week 156; n=37, 42, 49, 0 | 1.05 (2.056) | 0.75 (1.797) | 1.64 (1.291) |
  WBC count; Week 168; n=35, 43, 47, 0: number analyzed (Participants) | 35 | 43 | 47 | 0
  WBC count; Week 168; n=35, 43, 47, 0 | 0.97 (1.859) | 0.97 (1.748) | 1.58 (1.472) |
  WBC count; Week 180; n=36, 41, 47, 0: number analyzed (Participants) | 36 | 41 | 47 | 0
  WBC count; Week 180; n=36, 41, 47, 0 | 1.07 (1.778) | 0.69 (1.902) | 1.33 (1.485) |
  WBC count; Week 192; n=35, 40, 47, 0: number analyzed (Participants) | 35 | 40 | 47 | 0
  WBC count; Week 192; n=35, 40, 47, 0 | 0.61 (1.645) | 0.89 (1.972) | 1.11 (1.428) |
  WBC count; Week 204; n=34, 39, 47, 0: number analyzed (Participants) | 34 | 39 | 47 | 0
  WBC count; Week 204; n=34, 39, 47, 0 | 0.98 (2.042) | 0.95 (1.823) | 1.24 (1.554) |
  WBC count; Week 216; n=32, 39, 43, 0: number analyzed (Participants) | 32 | 39 | 43 | 0
  WBC count; Week 216; n=32, 39, 43, 0 | 0.88 (2.175) | 1.01 (1.859) | 1.37 (1.656) |
  WBC count; Week 228; n=31, 39, 47, 0: number analyzed (Participants) | 31 | 39 | 47 | 0
  WBC count; Week 228; n=31, 39, 47, 0 | 0.98 (1.970) | 1.13 (1.918) | 1.31 (1.329) |
  WBC count; Week 240; n=32, 39, 47, 0: number analyzed (Participants) | 32 | 39 | 47 | 0
  WBC count; Week 240; n=32, 39, 47, 0 | 0.79 (1.851) | 1.15 (1.942) | 1.53 (2.455) |
  WBC count; Week 252; n=31, 36, 45, 0: number analyzed (Participants) | 31 | 36 | 45 | 0
  WBC count; Week 252; n=31, 36, 45, 0 | 0.66 (1.649) | 1.10 (1.814) | 1.17 (1.531) |
  WBC count; Week 264; n=32, 38, 46, 0: number analyzed (Participants) | 32 | 38 | 46 | 0
  WBC count; Week 264; n=32, 38, 46, 0 | 0.62 (1.798) | 1.21 (1.985) | 1.66 (2.030) |
  WBC count; Week 276; n=31, 38, 45, 0: number analyzed (Participants) | 31 | 38 | 45 | 0
  WBC count; Week 276; n=31, 38, 45, 0 | 0.92 (1.985) | 1.04 (2.056) | 1.57 (1.721) |
  WBC count; Week 288; n=30, 38, 44, 0: number analyzed (Participants) | 30 | 38 | 44 | 0
  WBC count; Week 288; n=30, 38, 44, 0 | 0.92 (2.188) | 1.13 (2.293) | 1.32 (1.908) |
  WBC count; Week 300; n=30, 37, 43, 0: number analyzed (Participants) | 30 | 37 | 43 | 0
  WBC count; Week 300; n=30, 37, 43, 0 | 0.58 (1.762) | 0.77 (1.856) | 1.02 (1.321) |
  WBC count; Week 312; n=31, 33, 41, 0: number analyzed (Participants) | 31 | 33 | 41 | 0
  WBC count; Week 312; n=31, 33, 41, 0 | 0.57 (1.732) | 0.70 (2.051) | 0.95 (1.274) |
  WBC count; Week 324; n=3, 4, 2, 0: number analyzed (Participants) | 3 | 4 | 2 | 0
  WBC count; Week 324; n=3, 4, 2, 0 | 1.97 (3.075) | 0.53 (0.984) | -0.05 (1.626) |

32. Secondary Outcome: Percentage of Participants Who Discontinued Investigational Product Due to Adverse Events
Description: AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The percentage of participants with adverse events leading to withdrawal/permanent discontinuation of investigational product is presented.
Time Frame: Up to Week 324
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants | 7 | 7 | 7 | 15

33. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Twelve lead ECG was performed after the participants had rested in a semi-supine position for at least 5 minutes using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT (QTc) intervals. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for worst case results at any time on-treatment is presented.
Time Frame: Up to Week 324
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants | 25 | 19 | 15 | 10

34. Secondary Outcome: Number of Participants With AEs and SAEs-Induction Phase
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcomes mentioned before; all events of possible drug-induced liver injury with hyperbilirubinemia.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  Any AE | 54 | 54 | 55 | 59
  Any SAE | 2 | 0 | 2 | 2

35. Secondary Outcome: Number of Participants With Maximum Treatment-emergent Clinical Chemistry Toxicity-Induction Phase
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: ALT, albumin, ALP, AST, CO2/bicarbonate, chloride, cholesterol, CK, creatinine, glucose, high density lipoprotein (HDL) cholesterol, LDL cholesterol, lipase, inorganic phosphorus, potassium, sodium, total bilirubin, triglycerides and urea/blood urea nitrogen (BUN). A toxicity was considered treatment emergent if it developed or increased in intensity from Baseline while on-treatment. Laboratory toxicities were graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=Mild, Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  ALT; Grade 1 | 3 | 4 | 13 | 8
  ALT; Grade 2 | 1 | 5 | 0 | 4
  ALT; Grade 3 | 0 | 0 | 0 | 0
  ALT; Grade 4 | 0 | 0 | 2 | 0
  Albumin; Grade 1 | 0 | 0 | 0 | 0
  Albumin; Grade 2 | 0 | 0 | 0 | 0
  Albumin; Grade 3 | 0 | 0 | 0 | 0
  Albumin; Grade 4 | 0 | 0 | 0 | 0
  ALP; Grade 1 | 0 | 1 | 4 | 3
  ALP; Grade 2 | 0 | 1 | 0 | 0
  ALP; Grade 3 | 0 | 0 | 0 | 0
  ALP; Grade 4 | 0 | 0 | 0 | 0
  AST; Grade 1 | 6 | 8 | 7 | 6
  AST; Grade 2 | 2 | 5 | 1 | 1
  AST; Grade 3 | 1 | 0 | 3 | 2
  AST; Grade 4 | 0 | 0 | 0 | 0
  CO2/bicarbonate; Grade 1 | 1 | 5 | 1 | 6
  CO2/bicarbonate; Grade 2 | 0 | 0 | 0 | 0
  CO2/bicarbonate; Grade 3 | 0 | 0 | 0 | 0
  CO2/bicarbonate; Grade 4 | 0 | 0 | 0 | 0
  Chloride; Grade 1 | 0 | 0 | 0 | 0
  Chloride; Grade 2 | 0 | 0 | 0 | 0
  Chloride; Grade 3 | 0 | 0 | 0 | 0
  Chloride; Grade 4 | 0 | 0 | 0 | 0
  Cholesterol; Grade 1 | 7 | 8 | 12 | 4
  Cholesterol; Grade 2 | 3 | 2 | 3 | 9
  Cholesterol; Grade 3 | 0 | 0 | 2 | 6
  Cholesterol; Grade 4 | 0 | 0 | 0 | 0
  CK; Grade 1 | 7 | 5 | 6 | 4
  CK; Grade 2 | 2 | 2 | 3 | 1
  CK; Grade 3 | 3 | 1 | 1 | 2
  CK; Grade 4 | 2 | 4 | 2 | 4
  Creatinine; Grade 1 | 0 | 0 | 0 | 1
  Creatinine; Grade 2 | 1 | 0 | 0 | 1
  Creatinine; Grade 3 | 0 | 0 | 0 | 0
  Creatinine; Grade 4 | 0 | 0 | 0 | 0
  Glucose; Grade 1 | 10 | 8 | 13 | 6
  Glucose; Grade 2 | 5 | 3 | 1 | 5
  Glucose; Grade 3 | 0 | 0 | 2 | 0
  Glucose; Grade 4 | 0 | 0 | 0 | 1
  HDL cholesterol; Grade 1 | 0 | 0 | 0 | 0
  HDL cholesterol; Grade 2 | 0 | 0 | 0 | 0
  HDL cholesterol; Grade 3 | 0 | 0 | 0 | 0
  HDL cholesterol; Grade 4 | 0 | 0 | 0 | 0
  LDL cholesterol; Grade 1 | 5 | 9 | 8 | 4
  LDL cholesterol; Grade 2 | 4 | 1 | 5 | 8
  LDL cholesterol; Grade 3 | 0 | 0 | 3 | 2
  LDL cholesterol; Grade 4 | 0 | 0 | 0 | 0
  Lipase; Grade 1 | 9 | 3 | 5 | 6
  Lipase; Grade 2 | 6 | 1 | 7 | 5
  Lipase; Grade 3 | 2 | 1 | 4 | 1
  Lipase; Grade 4 | 0 | 0 | 1 | 0
  Inorganic phosphorus; Grade 1 | 5 | 2 | 7 | 6
  Inorganic phosphorus; Grade 2 | 6 | 2 | 2 | 8
  Inorganic phosphorus; Grade 3 | 1 | 1 | 2 | 2
  Inorganic phosphorus; Grade 4 | 0 | 0 | 0 | 0
  Potassium; Grade 1 | 7 | 1 | 2 | 2
  Potassium; Grade 2 | 0 | 0 | 0 | 1
  Potassium; Grade 3 | 0 | 0 | 0 | 0
  Potassium; Grade 4 | 0 | 0 | 0 | 0
  Sodium; Grade 1 | 7 | 4 | 7 | 8
  Sodium; Grade 2 | 0 | 0 | 0 | 1
  Sodium; Grade 3 | 0 | 0 | 0 | 0
  Sodium; Grade 4 | 0 | 0 | 0 | 0
  Total bilirubin; Grade 1 | 0 | 1 | 4 | 0
  Total bilirubin; Grade 2 | 2 | 1 | 1 | 0
  Total bilirubin; Grade 3 | 0 | 0 | 0 | 0
  Total bilirubin; Grade 4 | 0 | 0 | 0 | 0
  Triglycerides; Grade 1 | 0 | 0 | 0 | 0
  Triglycerides; Grade 2 | 0 | 1 | 3 | 2
  Triglycerides; Grade 3 | 0 | 0 | 1 | 0
  Triglycerides; Grade 4 | 0 | 0 | 0 | 1
  Urea/BUN; Grade 1 | 0 | 0 | 0 | 0
  Urea/BUN; Grade 2 | 0 | 0 | 0 | 0
  Urea/BUN; Grade 3 | 0 | 0 | 0 | 0
  Urea/BUN; Grade 4 | 0 | 0 | 0 | 0

36. Secondary Outcome: Number of Participants With Maximum Treatment-emergent Hematology Toxicities-Induction Phase
Description: Blood samples were collected for the analysis of following hematology parameters: APTT, basophils, eosinophils, hematocrit, hemoglobin, INR, lymphocytes, mean corpuscle volume (MCV), monocytes, platelet count, PT, red blood cell (RBC) count, total neutrophils and WBC count. A toxicity was considered treatment emergent if it developed or increased in intensity from Baseline while on-treatment. Laboratory toxicities were graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, where Grade 1=Mild, Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening.
Time Frame: Up to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Participants
  APTT; Grade 1 | 1 | 0 | 1 | 3
  APTT; Grade 2 | 0 | 0 | 0 | 0
  APTT; Grade 3 | 0 | 0 | 0 | 0
  APTT; Grade 4 | 0 | 1 | 1 | 0
  Basophils; Grade 1 | 0 | 0 | 0 | 0
  Basophils; Grade 2 | 0 | 0 | 0 | 0
  Basophils; Grade 3 | 0 | 0 | 0 | 0
  Basophils; Grade 4 | 0 | 0 | 0 | 0
  Eosinophils; Grade 1 | 0 | 0 | 0 | 0
  Eosinophils; Grade 2 | 0 | 0 | 0 | 0
  Eosinophils; Grade 3 | 0 | 0 | 0 | 0
  Eosinophils; Grade 4 | 0 | 0 | 0 | 0
  Hematocrit; Grade 1 | 0 | 0 | 0 | 0
  Hematocrit; Grade 2 | 0 | 0 | 0 | 0
  Hematocrit; Grade 3 | 0 | 0 | 0 | 0
  Hematocrit; Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 1 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 2 | 1 | 0 | 0 | 0
  Hemoglobin; Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin; Grade 4 | 0 | 0 | 0 | 0
  INR; Grade 1 | 0 | 2 | 0 | 1
  INR; Grade 2 | 0 | 0 | 0 | 0
  INR; Grade 3 | 0 | 0 | 0 | 0
  INR; Grade 4 | 0 | 1 | 0 | 0
  Lymphocytes; Grade 1 | 0 | 0 | 0 | 0
  Lymphocytes; Grade 2 | 0 | 0 | 0 | 0
  Lymphocytes; Grade 3 | 0 | 0 | 0 | 0
  Lymphocytes; Grade 4 | 0 | 0 | 0 | 0
  MCV; Grade 1 | 0 | 0 | 0 | 0
  MCV; Grade 2 | 0 | 0 | 0 | 0
  MCV; Grade 3 | 0 | 0 | 0 | 0
  MCV; Grade 4 | 0 | 0 | 0 | 0
  Monocytes; Grade 1 | 0 | 0 | 0 | 0
  Monocytes; Grade 2 | 0 | 0 | 0 | 0
  Monocytes; Grade 3 | 0 | 0 | 0 | 0
  Monocytes; Grade 4 | 0 | 0 | 0 | 0
  Platelet count; Grade 1 | 2 | 0 | 2 | 1
  Platelet count; Grade 2 | 0 | 0 | 0 | 0
  Platelet count; Grade 3 | 0 | 0 | 0 | 0
  Platelet count; Grade 4 | 0 | 0 | 0 | 0
  PT; Grade 1 | 0 | 1 | 0 | 1
  PT; Grade 2 | 0 | 0 | 0 | 0
  PT; Grade 3 | 0 | 0 | 0 | 0
  PT; Grade 4 | 0 | 1 | 0 | 0
  RBC; Grade 1 | 0 | 0 | 0 | 0
  RBC; Grade 2 | 0 | 0 | 0 | 0
  RBC; Grade 3 | 0 | 0 | 0 | 0
  RBC; Grade 4 | 0 | 0 | 0 | 0
  Total neutrophils; Grade 1 | 8 | 6 | 8 | 2
  Total neutrophils; Grade 2 | 3 | 2 | 3 | 2
  Total neutrophils; Grade 3 | 0 | 0 | 0 | 1
  Total neutrophils; Grade 4 | 0 | 0 | 1 | 1
  WBC count; Grade 1 | 0 | 2 | 2 | 1
  WBC count; Grade 2 | 0 | 1 | 0 | 0
  WBC count; Grade 3 | 0 | 0 | 0 | 0
  WBC count; Grade 4 | 0 | 0 | 0 | 0

37. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Adverse Events-Induction Phase
Description: as for outcome 32
Time Frame: Up to Week 24
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 60 | 60 | 61 | 62
Percentage of participants | 0 | 2 | 5 | 13

38. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Adverse Events-Maintenance Phase
Description: as for outcome 32
Time Frame: Week 24 to Week 96
Population: Maintenance Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg | Efavirenz 600 mg
Number analyzed (Participants) | 52 | 53 | 55 | 47
Percentage of participants | 2 | 4 | 2 | 2

39. Secondary Outcome: Area Under the Concentration Time Curve Over the Dosing Interval (AUC[0-tau]) for GSK1265744 at Week 2
Description: Blood samples for pharmacokinetic (PK) analysis were collected at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis. The PK Summary Population comprised of all participants who received GSK1265744 or with Rilpivirine, underwent intensive and/or limited/sparse PK sampling during the study, and provided evaluable GSK1265744 and Rilpivirine plasma concentration data
Time Frame: pre-dose, 1, 2, 3, 4, 8 and 24 hours post-dose at Week 2
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg
Number analyzed (Participants) | 14 | 12 | 11
Hours*micrograms per milliliter | 45.69 (32) | 133.74 (32) | 227.58 (57)

40. Secondary Outcome: Maximum Observed Concentration (Cmax) for GSK1265744 at Week 2
Description: Blood samples for PK analysis were collected at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: pre-dose, 1, 2, 3, 4, 8 and 24 hours post-dose at Week 2
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg
Number analyzed (Participants) | 14 | 12 | 11
Micrograms per milliliter | 2.77 (33) | 7.49 (28) | 13.12 (44)

41. Secondary Outcome: Concentration at the End of a Dosing Interval (Ctau) for GSK1265744 at Week 2
Description: as for outcome 40
Time Frame: pre-dose, 1, 2, 3, 4, 8 and 24 hours post dose at Week 2
Population: PK Summary Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg
Number analyzed (Participants) | 14 | 12 | 9
Micrograms per milliliter | 1.45 (37) | 4.34 (38) | 5.83 (61)

42. Secondary Outcome: AUC(0 to Tau) for Rilpivirine
Description: Data was not collected for analysis of rilpivirine PK parameters.
Time Frame: pre-dose and 2 to 4 hours post-dose at Weeks 26 and 36
Population: PK Summary Population. Data were not collected for rilpivirine PK parameters since this drug has been approved already for treatment and the PK of the drug has been well characterized
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg
Number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: Cmax for Rilpivirine
Description: Data was not collected for analysis of rilpivirine PK parameters.
Time Frame: pre-dose and 2 to 4 hours post-dose at Weeks 26 and 36
Population: as for outcome 42
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg
Number analyzed (Participants) | 0 | 0 | 0

44. Secondary Outcome: Ctau for Rilpivirine
Description: Data was not collected for analysis of rilpivirine PK parameters.
Time Frame: pre-dose and 2 to 4 hours post-dose at Weeks 26 and 36
Population: as for outcome 42
Arm/Group | GSK1265744 10 mg | GSK1265744 30 mg | GSK1265744 60 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from start of study treatment (Day 1) to Week 24 for induction phase; Week 24 to Week 96 for Maintenance Phase and from Week 96 to Week 324 for Open-label phase.
Description: Non-SAEs and SAEs were collected in the Safety Population (Induction and Open-label phase) and Maintenance Safety Population (Maintenance Phase). Participants randomized to Efavirenz 600 mg arm were considered to have completed their participation in the study after Week 96; hence were no longer followed as part of this study.
Groups:
- GSK1265744 10 mg (Induction Phase): Participants were administered one tablet of GSK1265744 10 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or 300 mg/200 mg TDF/FTC) from Day 1 to Week 24 during the double-blind induction phase. All doses were administered orally with meal.
- GSK1265744 30 mg (Induction Phase): Participants were administered one tablet of GSK1265744 30 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. All doses were administered orally with meal.
- GSK1265744 60 mg (Induction Phase): Participants were administered two tablets of GSK1265744 30 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. All doses were administered orally with meal.
- Efavirenz 600 mg (Induction Phase): Participants were administered one tablet of efavirenz 600 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. All doses were administered orally with meal.
- GSK1265744 10 mg (Maintenance Phase): Participants were administered one tablet of GSK1265744 10 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or 300 mg/200 mg TDF/FTC) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received one tablet of GSK1265744 10 mg and one tablet of placebo in combination with one tablet of RPV 25 mg once daily from Week 24 to 96. All doses were administered orally with meal.
- GSK1265744 30 mg (Maintenance Phase): Participants were administered one tablet of GSK1265744 30 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received one tablet of GSK1265744 30 mg and one tablet of placebo in combination with one tablet of RPV 25 mg once daily from Week 24 to 96. All doses were administered orally with meal.
- GSK1265744 60 mg (Maintenance Phase): Participants were administered two tablets of GSK1265744 30 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received two tablets of GSK1265744 30 mg in combination with one tablet of RPV 25 mg once daily from Week 24 to 96. All doses were administered orally with meal.
- Efavirenz 600 mg (Maintenance Phase): Participants were administered one tablet of efavirenz 600 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants continued to receive one tablet of efavirenz 600 mg in combination with ABC/3TC or TDF/FTC once daily.
- GSK1265744 10 mg (Open-label Phase): Participants were administered one tablet of GSK1265744 10 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or 300 mg/200 mg TDF/FTC) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received one tablet of GSK1265744 10 mg and one tablet of placebo in combination with one tablet of RPV once daily. Participants continuing in the open-label phase of the study received one tablet of GSK1265744 30 mg along with RPV 25 mg once daily. All doses were administered orally with meal.
- GSK1265744 30 mg (Open-label Phase): Participants were administered one tablet of GSK1265744 30 mg and one tablet of placebo once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received one tablet of GSK1265744 30 mg and one tablet of placebo in combination with one tablet of RPV 25 mg once daily. Participants continuing in the open-label phase of the study received one tablet of GSK1265744 30 mg along with RPV 25 mg once daily. All doses were administered orally with meal.
- GSK1265744 60 mg (Open-label Phase): Participants were administered two tablets of GSK1265744 30 mg once daily along with investigator selected, fixed dose dual NRTI therapy (either ABC/3TC 600 mg/300 mg or TDF/FTC 300 mg/200 mg) from Day 1 to Week 24 during the double-blind induction phase. In the Maintenance Phase (double-blind), eligible participants received two tablets of GSK1265744 30 mg in combination with one tablet of RPV 25 mg once daily. Participants continuing in the open-label phase of the study received one tablet of GSK1265744 30 mg along with RPV 25 mg once daily. All doses were administered orally with meal.
- Efavirenz 600mg (Open-label Phase): Participants in this arm did not enter open-label phase and were considered to have completed the study after Week 96.
Arm/Group | GSK1265744 10 mg (Induction Phase) | GSK1265744 30 mg (Induction Phase) | GSK1265744 60 mg (Induction Phase) | Efavirenz 600 mg (Induction Phase) | GSK1265744 10 mg (Maintenance Phase) | GSK1265744 30 mg (Maintenance Phase) | GSK1265744 60 mg (Maintenance Phase) | Efavirenz 600 mg (Maintenance Phase) | GSK1265744 10 mg (Open-label Phase) | GSK1265744 30 mg (Open-label Phase) | GSK1265744 60 mg (Open-label Phase) | Efavirenz 600mg (Open-label Phase)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/61 | 0/62 | 0/52 | 0/53 | 0/55 | 0/47 | 0/46 | 1/47 | 1/51 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/60 | 0/60 | 2/61 | 2/62 | 5/52 | 5/53 | 5/55 | 2/47 | 7/46 | 8/47 | 5/51 | 0/0
Other Adverse Events (participants affected / at risk) | 46/60 | 47/60 | 50/61 | 54/62 | 35/52 | 44/53 | 47/55 | 33/47 | 32/46 | 38/47 | 40/51 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1265744 10 mg (Induction Phase) (N=60) | GSK1265744 30 mg (Induction Phase) (N=60) | GSK1265744 60 mg (Induction Phase) (N=61) | Efavirenz 600 mg (Induction Phase) (N=62) | GSK1265744 10 mg (Maintenance Phase) (N=52) | GSK1265744 30 mg (Maintenance Phase) (N=53) | GSK1265744 60 mg (Maintenance Phase) (N=55) | Efavirenz 600 mg (Maintenance Phase) (N=47) | GSK1265744 10 mg (Open-label Phase) (N=46) | GSK1265744 30 mg (Open-label Phase) (N=47) | GSK1265744 60 mg (Open-label Phase) (N=51) | Efavirenz 600mg (Open-label Phase) (N=0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1265744 10 mg (Induction Phase) (N=60) | GSK1265744 30 mg (Induction Phase) (N=60) | GSK1265744 60 mg (Induction Phase) (N=61) | Efavirenz 600 mg (Induction Phase) (N=62) | GSK1265744 10 mg (Maintenance Phase) (N=52) | GSK1265744 30 mg (Maintenance Phase) (N=53) | GSK1265744 60 mg (Maintenance Phase) (N=55) | Efavirenz 600 mg (Maintenance Phase) (N=47) | GSK1265744 10 mg (Open-label Phase) (N=46) | GSK1265744 30 mg (Open-label Phase) (N=47) | GSK1265744 60 mg (Open-label Phase) (N=51) | Efavirenz 600mg (Open-label Phase) (N=0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (4) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 7 (7) | 11 (13) | 8 (8) | 5 (7) | 7 (9) | 5 (6) | 5 (5) | 6 (7) | 5 (6) | 5 (5) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (15) | 11 (14) | 11 (13) | 13 (13) | 0 (0) | 3 (3) | 8 (8) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (7) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (7) | 5 (8) | 7 (8) | 10 (10) | 4 (4) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 3 (3) | 0 (0)
Feeling drunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 1 (1) | 4 (4) | 3 (5) | 4 (7) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5) | 3 (4) | 3 (3) | 4 (4) | 3 (4) | 6 (6) | 3 (4) | 2 (3) | 3 (3) | 4 (5) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gonorrhoea (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (7) | 4 (4) | 3 (3) | 1 (1) | 4 (5) | 4 (4) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (9) | 2 (2) | 8 (12) | 3 (5) | 2 (2) | 4 (5) | 2 (2) | 5 (5) | 5 (10) | 5 (5) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 3 (3) | 2 (5) | 3 (3) | 1 (1) | 3 (5) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 2 (3) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 6 (6) | 6 (10) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syphilis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 5 (6) | 4 (4) | 2 (3) | 3 (3) | 4 (4) | 3 (3) | 4 (6) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 8 (8) | 9 (10) | 9 (11) | 9 (11) | 14 (16) | 12 (14) | 5 (7) | 3 (3) | 15 (28) | 14 (18) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urethritis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 4 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 2 (2) | 2 (2) | 3 (4) | 2 (3) | 4 (6) | 4 (4) | 3 (3) | 6 (10) | 3 (4) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (4) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 4 (4) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 5 (5) | 2 (2) | 18 (19) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 13 (17) | 13 (14) | 7 (8) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 4 (4) | 3 (4) | 2 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 5 (5) | 3 (3) | 15 (15) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 5 (6) | 2 (2) | 4 (4) | 4 (4) | 2 (3) | 3 (3) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 6 (6) | 7 (7) | 14 (15) | 3 (3) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (5) | 4 (4) | 6 (6) | 3 (4) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 5 (7) | 4 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (4) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 2 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 3 (3) | 8 (8) | 1 (1) | 6 (7) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.